# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for DMID Protocol: 16-0034

**Study Title:** 

Phase I, Randomized, Double-blinded, Placebo-Controlled Dose De-escalation Study to Evaluate the Safety and Immunogenicity of Alum Adjuvanted Zika Virus Purified Inactivated Vaccine (ZPIV) Administered by the Intramuscular Route in Adult Subjects who Reside in a Flavivirus Endemic Area

NCT03008122

Version 1.0

**DATE: 07DEC2022** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

# Phase I, Randomized, Double-blinded, Placebo-Controlled Dose De-escalation Study to Evaluate the Safety and Immunogenicity of Alum Adjuvanted Zika Virus Purified Inactivated Vaccine (ZPIV) Administered by the Intramuscular Route in Adult Subjects who Reside in a Flavivirus Endemic Area

| Protocol Number Code: | DMID Protocol: 16-0034 |
|---|---|
| <b>Development Phase:</b> | Phase I |
| Products: | Adjuvanted Zika Virus Purified Inactivated Vaccine and Normal Saline, 0.9% Sodium Chloride, USP |
| Form/Route: | Intramuscular injection |
| Indication Studied: | Zika |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | March 21, 2017 |
| Clinical Trial Completion Date: | August 10, 2021 |
| Date of the Analysis Plan: | 07DEC2022 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| <b>TABLE</b> | OF CONTENTS | III |
|---|---|---|
| LIST OF | ABBREVIATIONS | VII |
| 1. | PREFACE | 1 |
| 2. | INTRODUCTION | 2 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 3 |
| 3.1. | Study Objectives | 3 |
| 3.2. | Endpoints | 3 |
| 3.3. | Study Definitions and Derived Variables | 5 |
| 4. | INVESTIGATIONAL PLAN | 7 |
| 4.1. | Overall Study Design and Plan | 7 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 8 |
| 4.3. | Selection of Study Population | 8 |
| 4.3.1. | Subject Inclusion Criteria | 8 |
| 4.3.2. | Subject Exclusion Criteria | 10 |
| 4.4. | Treatments | 12 |
| 4.4.1. | Treatments Administered. | 12 |
| 4.4.2. | Identity of Investigational Product(s) | 12 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 12 |
| 4.4.4. | Selection of Doses in the Study | 12 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 13 |
| 4.4.6. | Blinding | 13 |
| 4.4.7. | Prior and Concomitant Therapy | 13 |
| 4.4.8. | Treatment Compliance | 13 |
| 4.5. | Immunogenicity and Safety Variables | 13 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 15 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 16 |
| 6.1. | General Principles | 16 |
| 6.2. | Timing of Analyses. | 16 |
| 6.3. | Analysis Populations | 16 |
| 6.3.1. | Safety Population | 17 |

# **Table of Contents** (continued)

| 6.3.2. | Immunogenicity (IMM) Population | 17 |
|---|---|---|
| 6.3.3. | Per-Protocol (PP) Population. | 17 |
| 6.4. | Covariates and Subgroups | 17 |
| 6.5. | Missing Data | 18 |
| 6.6. | Interim Analyses and Data Monitoring | 18 |
| 6.7. | Multicenter Studies | 18 |
| 6.8. | Multiple Comparisons/Multiplicity | 18 |
| 7. | STUDY SUBJECTS | 19 |
| 7.1. | Disposition of Subjects | 19 |
| 7.2. | Protocol Deviations | 19 |
| 8. | IMMUNOGENICITY EVALUATION | 20 |
| 8.1. | Primary Immunogenicity Analysis | 20 |
| 8.2. | Secondary Immunogenicity Analyses | 20 |
| 8.2.1. | ZIKV Microneutralization Antibodies (MN50) | 20 |
| 8.2.2. | ZIKV ELISA Antibodies | 20 |
| 8.3. | Exploratory Immunogenicity Analyses | 21 |
| 9. | SAFETY EVALUATION | 22 |
| 9.1. | Demographic and Other Baseline Characteristics | 22 |
| 9.1.1. | Pre-Existing Medical Conditions | 22 |
| 9.1.2. | Prior and Concomitant Medications | 22 |
| 9.2. | Measurements of Treatment Compliance | 22 |
| 9.3. | Adverse Events | 22 |
| 9.3.1. | Solicited Events and Symptoms | 22 |
| 9.3.2. | Unsolicited Adverse Events | |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 24 |
| 9.5. | Pregnancies | 25 |
| 9.6. | Clinical Laboratory Evaluations | 25 |
| 9.7. | Vital Signs and Physical Evaluations | 27 |
| 9.8. | Concomitant Medications | |
| 9.9. | Other Safety Measures | 27 |
| 10. | PHARMACOKINETICS | 29 |

### **Table of Contents** (continued) 11. 12. 13. 14. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR 15. PLANNED ANALYSES 34 16. 17. APPENDIX 1. TABLE MOCK-UPS......38 14.1.1 14.1.2 14.1.3 14.2 14.3 Safety Data......86 14.3.1 Displays of Adverse Events......86 Solicited Adverse Events 89 14.3.1.1 14.3.1.2 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events......140 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events.......143 14.3.4 14.3.5 Chemistry Results 146 14.3.5.1 14.3.5.2 14.3.5.3 14.3.6 14.4 APPENDIX 2. FIGURE MOCK-UPS.......164 10.1 14.2.2 Immunogenicity Response Figures by Measure, Treatment Group, and Time 14.3.1.1 Solicited Adverse Events 179

### **Table of Contents** (continued) 14.3.1.2 14.3.5 14.3.5.1 14.3.5.2 14.3.5.3 14.3.5 16.2 16.2.1 16.2.2 Protocol Deviations 198 16.2.3 Subjects Excluded from the Immunogenicity Analysis......200 16.2.4 16.2.6 16.2.7 Adverse Events 204 16.2.7.1 Solicited Events 204 16.2.7.2 Unsolicited Events 206 16.2.8 16.2.9 16.2.8.6 Pregnancy Reports 218

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|---------|--------------------------------------------------------------------|
| AESI | Adverse Event of Special Interest |
| AFI | Acute Febrile Illness |
| ALT | Alanine Aminotransferase |
| ARI | Acute Rash Illness |
| AST | Aspartate Aminotransferase |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| BUN | Blood Urea Nitrogen |
| С | Centigrade |
| CAIMED | Centro Ambulatorio de Investigaciones Medicas |
| CDC | Centers for Disease Control and Prevention |
| CFR | Code of Federal Regulations |
| CHIKV | Chikungunya virus |
| CI | Confidence Interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CONSORT | Consolidated Standards of Reporting Trials |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| DCC | Data Coordinating Center |
| DENV | Dengue Virus |
| DHHS | Department of Health and Human Services |
| DMID | Division of Microbiology and Infectious Diseases, NIAID, NIH, DHHS |
| DoD | Department of Defense |
| DRM | Data Review Meeting |
| EDC | Electronic Data Capture |
| ELISA | Enzyme-linked Immunosorbent Assay |
| ER | Emergency Room |
| F | Fahrenheit |
| FDA | Food and Drug Administration |

# **List of Abbreviations** (continued)

| FWA | Federal Wide Assurance |
|---------|-----------------------------------------------------|
| GCP | Good Clinical Practice |
| GGT | Gamma Glutamyl Transferase |
| GMFR | Geometric Mean Fold Rise |
| GMT | Geometric Mean Titer |
| НСТ | Hematocrit |
| HD | High Dose |
| HGB | Hemoglobin |
| HIPAA | Health Insurance Portability and Accountability Act |
| HLA | Human Leukocyte Antigen |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| ICMJE | International Committee of Medical Journal Editors |
| IDE | Investigational Device Exemption |
| IEC | Independent or Institutional Ethics Committee |
| IM | Intramuscular |
| IND | Investigational New Drug Application |
| IRB | Institutional Review Board |
| ISM | Independent Safety Monitor |
| ITT | Intention to Treat |
| JAMA | Journal of the American Medical Association |
| JEV | Japanese Encephalitis Virus |
| L | Liter |
| LD | Low Dose |
| LLN | Lower Limit of Normal |
| MAR | Missing at Random |
| MCAR | Missing Completely at Random |
| mcg | Microgram |
| MD | Medium Dose |
| MedDRA® | Medical Dictionary for Regulatory Activities |

# **List of Abbreviations** (continued)

| mEq | Milliequivalent |
|---------|------------------------------------------------------------------|
| mg | Milligram |
| mITT | Modified Intention to Treat |
| mL | Milliliter |
| mmHg | Millimeters of Mercury |
| MNAR | Missing Not at Random |
| MOP | Manual of Procedure |
| N | Number (typically refers to subjects) |
| NCI | National Cancer Institute, NIH, DHHS |
| NDA | New Drug Application |
| NEJM | New England Journal of Medicine |
| NIAID | National Institute of Allergy and Infectious Diseases, NIH, DHHS |
| NIH | National Institutes of Health |
| OCRA | Office of Clinical Research Affairs, DMID, NIAID, NIH, DHHS |
| OHRP | Office for Human Research Protections |
| OHSR | Office for Human Subjects Research |
| ORA | Office of Regulatory Affairs, DMID, NIAID, NIH, DHHS |
| PBMCs | Peripheral Blood Mononuclear Cells |
| PFU | Plaque Forming Units |
| PHI | Protected Health Information |
| PI | Principal Investigator |
| PP | Per Protocol |
| PREP | Public Readiness and Emergency Preparedness |
| PT | Preferred Term |
| QA | Quality Assurance |
| QC | Quality Control |
| RBC | Red Blood Cell |
| RCD | Reverse Cumulative Distribution |
| RNA | Ribonucleic Acid |
| <u></u> | Serious Adverse Event |
| SAE | Serious Adverse Event |

# **List of Abbreviations** (continued)

| SDCC | Statistical and Data Coordinating Center |
|-------|------------------------------------------|
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TBEV | Tick-borne Encephalitis Virus |
| U | Units |
| ULN | Upper Limit of Normal |
| US | United States |
| VTEU | Vaccine and Treatment Evaluation Unit |
| WBC | White Blood Cells |
| WHO | World Health Organization |
| WNV | West Nile Virus |
| WRAIR | Walter Reed Army Institute of Research |
| YFV | Yellow Fever Virus |
| ZIKV | Zika Virus |
| ZPIV | Zika Virus Purified Inactivated Vaccine |

### 1. PREFACE

This Statistical Analysis Plan (SAP) for DMID Protocol 16-0034, "Phase I, Randomized, Double-blinded, Placebo-Controlled Dose De-escalation Study to Evaluate the Safety and Immunogenicity of Alum Adjuvanted Zika Virus Purified Inactivated Vaccine (ZPIV) Administered by the Intramuscular Route in adult Subjects Who Reside in a Flavivirus Endemic Area" describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity and safety outcomes, and (4) shells of proposed tables and data listings and mock figures. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

### 2. INTRODUCTION

Zika virus (ZIKV) disease (also known as Zika) is an emerging mosquito-borne disease caused by an RNA virus from the family *Flaviviridae*, genus *Flavivirus*. As a Flavivirus, ZIKV is related to the four dengue viruses (DENV 1-4), West Nile virus (WNV), Japanese encephalitis virus (JEV), yellow fever virus (YFV), and tick-borne encephalitic virus (TBEV). The majority of human ZIKV infections result in an asymptomatic infection or a benign, self-limited acute febrile illness. ZIKV infections are characterized primarily by the presence of rash, fever, conjunctivitis, and/or arthralgia, which have been found in the majority of cases seeking care or detected by public health surveillance [8]. In February 2016, the World Health Organization (WHO) declared the emerging ZIKV epidemic a "Public Health Emergency of International Concern." Active mosquito-borne transmission of ZIKV has now been reported in more than 35 countries in South America, Central America, and the Caribbean including Puerto Rico (PAHO 2016).

There is no specific treatment or vaccine currently available to treat or prevent ZIKV infections, other than mosquito control measures. Development of a preventive vaccine against ZIKV infections is a high global public health priority. The ZIKV vaccine used in this trial is a purified inactivated virus vaccine that was produced by the Walter Reed Army Institute of Research (WRAIR). ZPIV is intended to be used in flavivirus endemic areas and among US military members and travelers who may have already received another flavivirus vaccine. Therefore, evaluating the safety and immune response in both flavivirus-naïve and flavivirus-immune subjects is important. This clinical trial was conducted in Puerto Rico, whose population has been exposed to at least the flaviviruses, DENV 1-4 and ZIKV, with potential exposure to WNV in visits to the mainland U.S. and YFV through vaccination. This study setting provides the opportunity to evaluate ZPIV among a largely flavivirus-immune population residing in an area with active ZIKV and DENV transmission.

### 3. STUDY OBJECTIVES AND ENDPOINTS

### 3.1. Study Objectives

### **Primary Objectives:**

- 1. Assess the safety and reactogenicity of a homologous prime boost regimen of ZPIV given at two different dose levels in a dose de-escalation format in healthy adult subjects who live in Puerto Rico, a flavivirus endemic area.
- 2. Compare the safety and reactogenicity profile of ZPIV after each vaccination, between dosage groups, and by pre-vaccination flavivirus immune status.

### **Secondary Objectives:**

- 1. Assess the humoral immune response to a homologous prime-boost regimen of ZPIV after each dose of vaccine as determined by kinetics of the immune responses, seroconversion rates, and Geometric Mean Titers (GMT) overall, and compare results between dosage groups and by prevaccination flavivirus immune status.
- 2. Assess the durability of the humoral immune response to ZPIV at 6, 12, 18, and 24 months after the second vaccine administration overall, and compare results between dosage groups and by pre-vaccination flavivirus immune status.

### **Exploratory Objectives**

1. Estimate the incidence of ZIKV and DENV infections between Visit 00 and the subject's last visit and describe the clinical presentation including disease severity overall, by dosage group, product received, and pre-vaccination flavivirus immune status.

# 3.2. Endpoints

### **Primary Endpoints:**

- 1. Frequency and severity of solicited injection site and systemic reactogenicity from time of study vaccine administration through Day 8 after each administration of study vaccine overall and by dosage group and pre-vaccination flavivirus immune status.
- 2. Frequency and severity of unsolicited vaccine-related adverse events (AE), including vaccine-related laboratory AE, from first administration of study vaccine until 28 days after the last vaccination overall and by dosage group and pre-vaccination flavivirus immune status.
- 3. Frequency, type, and duration of serious adverse events (SAE) and adverse events of special interest (AESI) considered related to study vaccine from the first administration of study vaccine until the end of the study overall, and by dosage group and pre-vaccination flavivirus immune status.
- 4. Frequency of new onset chronic medical conditions reported at any time from the first administration of study vaccine until the end of the study overall, and by dosage group and prevaccination flavivirus immune status.
- 5. Comparison of the frequency, type and duration of vaccine-related Grade 3 local, systemic, or laboratory AE, and Grade 2 or greater local or systemic reactogenicity through Day 8 after each

study vaccine administration between dosage groups and by pre-vaccination flavivirus immune status.

6. Comparison of study withdrawals and discontinuation of study vaccination due to any reason between dosage groups and by pre-vaccination flavivirus immune status.

### **Secondary Endpoints:**

- 1. Frequency of seroconversion to ZIKV at each post-vaccination visit measured by ZIKV ELISA and neutralization assay in comparison with baseline samples (collected at Visit 00) overall, and by dosage group and pre-vaccination flavivirus immune status.
- 2. Per Visit GMT as measured by ZIKV ELISA and neutralization assay after each study vaccine administration and for each post-vaccination visit overall, and by dosage group and prevaccination flavivirus immune status.
- 3. Peak GMT as measured by ZIKV ELISA and neutralization assay after each vaccination and overall, and by dosage group and pre-vaccination flavivirus immune status.
- 4. Proportion of subjects with at least a 4-fold rise in ZIKV GMT as measured by ZIKV ELISA and neutralization assay at 4 weeks after each vaccination compared with baseline overall, and by dosage group and pre-vaccination flavivirus immune status.

### **Exploratory Endpoints:**

- 1. Number and proportion of subjects who develop an acute febrile illness (AFI) or an acute rash illness (ARI) who have evidence of acute ZIKV or DENV infection detected within 14 days of symptom onset. This endpoint will be analyzed for all subjects overall, and by dosage group, product received, and pre-vaccination flavivirus immune status.
- 2. Number and severity of laboratory confirmed ZIKV and DENV infections during the study, overall, by treatment group, and pre-vaccination immune status, where severity is described by:
  - Duration of symptoms
  - Grade of symptoms (mild, moderate, severe)
  - Use of concomitant medications
  - Need for hospitalization or other medical care

Laboratory confirmation will be made by AFI or ARI with either: 1) evidence of acute ZIKV and DENV infection within 14 days of symptom onset or 2) a 4-fold rise in DENV or ZIKV neutralization titers between samples collected at the last visit prior to and at the first visit following the AFI/ARI, where available.

# 3.3. Study Definitions and Derived Variables

### **Baseline Values**

Unless otherwise specified, baseline values will be defined as the last values obtained prior to the first investigational vaccination. Vital signs (pulse and blood pressure) assessed at screening will be considered as baseline. Any medical condition that is present at the time that the subject is screened will be considered as baseline and not reported as an adverse event.

### **Adverse Events of Special Interest**

For this study, Neurologic and Neuroinflammatory Disorders will be considered as adverse events of special interest (AESI). These include Acute Disseminated Encephalomyelitis (ADEM, including site specific variants), Cranial Nerve Disorders (including paralyses/paresis), Guillain-Barre Syndrome (GBS, including Miller Fisher Syndrome and other variants), Immune-mediated Peripheral Neuropathies and Plexopathies, Optic Neuritis, Multiple Sclerosis, Narcolepsy, Transverse Myelitis, meningitis, or meningoencephalitis.

### **Baseline Flavivirus Immune Status**

Subjects enrolled in the study will have blood drawn during the screening visit (Visit 00) or prevaccination at the first visit (Visit 01) to determine baseline flavivirus immune status. Serum will be tested via serology for antibodies to ZIKV and DENV. Baseline flavivirus immune status will be treated as a categorical variable and will be used to stratify tables and figures throughout the analyses specified in this SAP. The goal of determining the baseline flavivirus status is to see if there is an effect of baseline flavivirus seropositivity on response to ZPIV. With this in mind, subjects are categorized initially at ZIKV seropositive (based on a positive IgM or IgG assay pre-vaccination) or ZIKV seronegative (based on negative IgM and IgG tests pre-vaccination). Subjects are then subcategorized as DENV seropositive or seronegative, within each ZIKV category.

Baseline flavivirus immune status will be defined primarily as follows:

- ZIKV Seropositive: any subject with detectable ZIKV antibodies pre-vaccination
- ZIKV Seronegative: any subject without detectable ZIKV antibodies pre-vaccination

Baseline flavivirus immune status will then be further classified into the following groups:

- ZIKV Seropositive and DENV Seropositive
- ZIKV Seropositive and DENV Seronegative
- ZIKV Seronegative and DENV Seropositive
- ZIKV Seronegative and DENV Seronegative

Baseline DENV and ZIKV serostatus will be determined via IgM antibody and IgG ELISA assays, with subject results reported as either 'positive' or 'negative'. If a subject has a positive ZIKV result from either the IgM or IgG ELISA assays, they will be considered ZIKV seropositive at baseline. If a subject has inconclusive results for their baseline flavivirus immune status, they will not be included in analyses stratified by baseline flavivirus immune status but will be included in analyses of all subjects.

### **Post-Baseline Seropositivity**

Seropositivity post-baseline is defined as a titer  $\geq$ 10 and  $\geq$ 100 for ZIKV MN50 and a titer  $\geq$ 200 and  $\geq$ 600 for ZIKV ELISA.

### **Seroconversion**

Seroconversion for ZIKV MN50 titers and ZIKV ELISA titers is defined as ≥4-fold rise from baseline.

### **Acute Febrile Illness and Acute Rash Illness**

Acute febrile illness (AFI) is defined as grade 1 or higher fever on at least 2 consecutive days accompanied by any of the following: new rash not limited to vaccination site, arthralgia, or nonpurulent conjunctivitis. Acute rash illness (ARI) is defined as any new rash not limited to vaccination site.

### **Laboratory Confirmation of ZIKV or DENV Infection Among Those with AFI or ARI**

Among subjects with AFI or ARI, laboratory confirmation of ZIKV or DENV infection will be made by either 1) evidence of acute ZIKV and DENV infection within 14 days of symptom onset (confirmed via PCR) or 2) a 4-fold rise in DENV or ZIKV neutralization titers between samples collected at the last visit prior to and at the first visit following the AFI/ARI illness visit, where available.

### **Consideration of ZIKV Microneutralization Assay Results in Analysis**

The lower limit of quantitation (LLOQ) for ZIKV microneutralization assay results is 10. Any values less than the LLOQ will be assigned a value of 5 by the lab. This imputed value will be used for the purpose of calculating summary statistics such GMT and will be displayed in listings of immunogenicity data. If a subject has a baseline titer below the LLOQ (reported as 5), then they will be considered seroconverted if the post-baseline titer is at least 20 (at least a 4-fold rise). Similarly, a subject with a baseline ZIKV MN50 below the LLOQ will be considered seropositive if the post-baseline titer is at least 10 or 100, as applicable.

### 4. INVESTIGATIONAL PLAN

### 4.1. Overall Study Design and Plan

This study is a single-center, double-blinded, placebo-controlled, Phase 1, dose de-escalation study to evaluate the safety, reactogenicity, and immunogenicity of a purified inactivated, alum-adjuvanted ZIKV vaccine (ZPIV) administered in a homologous prime-boost regimen to healthy male and non-pregnant female adult subjects living in a flavivirus-endemic area. Two dose levels will be evaluated. Each subject will receive either placebo or 5 mcg (Group 1), or 2.5 mcg (Group 2) of ZPIV administered by IM injection. The study will consist of a screening period of up to 28 days, a vaccination period in which subjects will receive a prime dose of vaccine on Day 1 followed by a homologous boost on Day 29, and a follow-up period of 24 months post boost vaccination. See Table 1 of Appendix 1.

As this is a phase I study, the study will begin with enrollment of two sentinel subjects in Group 1 who will receive 5 mcg ZPIV open label. One sentinel subject will be vaccinated, followed for one day for safety and reactogenicity, and if no halting rules are met per determination of the PI and co-PI, then the second sentinel subject will receive 5 mcg ZPIV open-label. Both sentinels will be followed for safety through Day 8 and if no predefined halting rules are met and no safety concerns are identified, then enrollment of the Group 1 non-sentinel subjects will proceed in double-blind fashion. The same procedure will be used for administration of the boost vaccination to the Group 1 sentinels: 1 sentinel will receive 5 mcg ZPIV open-label, be followed for 1 day for safety and reactogenicity, and if no halting rules are met, then the second sentinel will receive the boost vaccine. Both sentinels will be followed until Day 8 after second vaccination for safety and reactogenicity and if no halting rules are then boost vaccination of the non-sentinel Group 1 subjects can proceed. Enrollment of the 2.5 mcg ZPIV group (Group 2) can begin after or at the same time non-sentinel subjects in Group 1 receive the 1st dose of vaccine.

Solicited local and systemic reactogenicity will be recorded through Day 8 after the prime and boost administration of study vaccine by the subject in a memory aid, and will be reviewed with the clinic staff during clinic visits on Days 2 and 8, and during a telephone visit on Day 4. Safety laboratories will be collected on Days 8 and 15 after administration of the prime and boost dose. Unsolicited AEs will be recorded and evaluated by medical history and targeted physical examinations as needed until 28 days after the second vaccination. SAEs, AESIs, and history of new medical conditions with onset after the first vaccination will be collected for the duration of the study.

Blood will be drawn to evaluate humoral immunity to ZIKV and DENV pre- and at multiple visits post-each vaccination, including baseline serology testing on Visit 00 to determine pre-vaccination flavivirus immune status. CPT tubes will be collected and peripheral blood mononuclear (PBMCs) cells will be harvested and stored for future assessment of immunity including cellular and humoral immunity and systems biology.

Subjects who develop an AFI (grade 1 or higher fever on at least 2 consecutive days accompanied by any of the following: new rash not limited to vaccination site, arthralgia, or nonpurulent conjunctivitis) or ARI (new rash not limited to vaccination site) at any time after signing the ICF until the end of study will be asked to contact the clinic within 3 days of symptom onset and return as soon as possible and at least within 14 days for blood and urine collection to evaluate for acute ZIKV and DENV infection. Subjects will also be asked about any history of AFI and ARI at each clinic visit and phone call after Visit 00. Subjects presenting for evaluation of AFI/ARI will have a medical history including travel

history collected, all symptoms recorded, physical exam if indicated, and concomitant medications and AEs collected, regardless of when the visit occurs.

The schedule of study procedures is displayed in Table 2.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

The strategy for the initial development of this vaccine is to conduct a series of phase I studies to assess the safety and immunogenicity in flavivirus-naïve and flavivirus-experienced subjects. Because it is not known how previous exposure to flaviviruses will affect the safety and immunogenicity profile of this vaccine, this strategy will address a critical gap necessary to complete an early and rapid assessment of the viability of this ZIKV vaccine candidate. All trials will initiate with a 5 mcg dose. The first two clinical trials will explore the safety and immune response to the vaccine in flavivirus naïve subjects and in subjects that have been previously vaccinated with JEV or YFV vaccines. This trial will be conducted in Puerto Rico, whose population has been exposed to DENV 1-4, ZIKV and potentially YFV and/or WNV. A fourth clinical trial will be conducted by Beth Israel Deaconess Medical Center to evaluate the safety and immunogenicity of an accelerated vaccination schedule with the Zika vaccine candidate in healthy adults. The initial doses and regimens that will be utilized in these initial trials was selected based on experience with other inactivated flavivirus vaccines and recent data from mouse and NHP studies. Experience with licensed flavivirus vaccines suggests a 5 mcg dose should be safe and immunogenic; the 5 mcg dose was safe and protective in a NHP model [1]. Therefore, for these trials, subjects will be enrolled initially in the 5 mcg group. To determine if lower doses of ZPIV are equally or comparably immunogenic to the 5 mcg dose, subjects in this trial will then be enrolled in the 2.5 mcg group, or in a 1.25 mcg group in other trials. ZPIV is intended to be used in flavivirus endemic areas and among US military members and travelers who may have already received another flavivirus vaccine. Therefore, evaluating the safety and immune response in both flavivirus-naïve and flavivirus-immune subjects is important. This study provides the opportunity to evaluate ZPIV among a largely flavivirusimmune population who resides in an area with active ZIKV and DENV transmission.

# **4.3.** Selection of Study Population

Approximately ninety subjects, males and non-pregnant, non-breastfeeding females, 21-49 years of age, inclusive, who are in good health (based on physical examination, medical history and clinical judgment) and meet all eligibility criteria, will be enrolled. The study population's racial and ethnic make-up should reflect the demographics of the larger community at the clinical trial site.

### 4.3.1. Subject Inclusion Criteria

Subjects eligible to participate in this study must meet all of the following inclusion criteria:

- 1. Must be a male or non-pregnant, non-breastfeeding female between the age of 21 and 49 years, inclusive at the time of screening and enrollment.
- 2. Must be willing and able to read, sign and date the informed consent document before study related procedures are performed.
- 3. Must be willing and able to comply with study requirements and available for follow-up visits for the entire study.
- 4. Must have a means to be contacted by telephone.

- 5. Must have a body mass index (BMI)  $\geq$ 18.1 and  $\leq$ 35.0 kg/m<sup>2</sup>.
- 6. Must have acceptable\* screening laboratory findings within 28 days before enrollment.
  - \*Acceptable clinical laboratory parameters include:
    - -Hemoglobin: women:  $\geq 11.5 \text{ g/dL}$ ; men  $\geq 13.5 \text{ g/dL}$
    - -Hematocrit: women:  $\geq 34.5\%$ ; men  $\geq 40.5\%$
    - -White blood cell count:  $\geq 3.500 \text{ cells/mm}^3 \text{ but } \leq 10.800 \text{ cells/mm}^3$
    - -*Platelets*:  $\geq 150,000 \text{ but } \leq 450,000 \text{ per mm}^3$
    - *-Urine dipstick (clean urine sample): protein* < 1+, *glucose negative*
    - -Serum creatinine  $\leq l x$  institutional upper limit of normal (ULN)
    - -Blood urea nitrogen (BUN) <25
    - -Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)  $\leq$  1.25 x institutional ULN
    - -Total bilirubin < 1.25 x institutional ULN
  - \*Note: If laboratory screening tests are out of acceptable range, repeat of screening tests is permitted once, provided there is an alternative explanation for the out of range value.
- 7. Must be in good health based on the investigator's clinical judgment when considering findings from past medical history, medication use, vital signs, and an abbreviated physical examination.
  - Note 1: Good health is defined by the absence of any medical condition described in the exclusion criteria in a subject with a normal abbreviated physical exam and vital signs. If the subject has a preexisting condition not listed in exclusion criteria, it cannot meet any of the following criteria: 1.) first diagnosed in last 3 months; 2.) worsening in terms of clinical outcome in last 6 months; or 3.) involves need for medication that may pose a risk to subject's safety or impede assessment of adverse events or immunogenicity if they participate in study.
  - Note 2: An abbreviated physical exam differs from a complete exam in that it does not include a genitourinary and rectal exam.
  - Note 3: Vital signs must be normal by protocol toxicity grading scale or determined to be normal-variant by investigator. In the event of an abnormal heart rate or blood pressure due to physiological variation or activity, the subject may rest for 10 minutes in a quiet room, and then blood pressure and/or heart rate may be re-measured. Repeated vital signs may be used to determine eligibility.
- 8. Women of childbearing potential\* must have a negative serum pregnancy test at screening and a negative urine pregnancy test immediately prior to each vaccination.
  - Note: All female subjects are considered of childbearing potential unless postmenopausal or surgically sterilized and  $\geq 3$  months have passed since sterilization procedure. Postmenopausal is defined as amenorrhea for  $\geq 12$  months without an alternative medical cause. Permanent female sterilization procedures include tubal ligation, bilateral salpingectomy, hysterectomy, bilateral oophorectomy, or successful Essure placement.
- 9. Women of childbearing potential must use an acceptable method of contraception\* from one month (30 days) prior to the first vaccination until the end of the study.
  - \*Acceptable methods of contraception include the following:

- -Use highly effective contraceptive methods, defined by <1% failure rate per year independent of user adherence, including long-acting reversible contraception (LARC): progestin-releasing subdermal implants and intrauterine devices (IUD), OR -Use effective contraceptive methods, defined by 5-9% failure rate with typical use and <1% failure rate with consistent and correct use, including: prescription oral contraceptives, contraceptive injections, combined pill, progestin-only pill, hormone-releasing transdermal patch or vaginal ring, and depot medroxyprogesterone acetate injection (Depo-Provera), OR -Male sex partners must have had a vasectomy  $\geq$ 3 months prior to first vaccination, OR -Practice abstinence defined as refraining from heterosexual intercourse from 30 days before first vaccination until the end of the study.
- 10. Female subjects must agree to not donate eggs (ova, oocytes) from the start of screening period until the end of the study.
- 11. Subjects must provide concurrent consent at the time of enrollment and 1<sup>st</sup> vaccination to future use of stored blood samples to measure immunity to ZIKV.

### 4.3.2. Subject Exclusion Criteria

Subjects eligible to participate in this study must not meet any of the following exclusion criteria:

- 1. Has plans to become pregnant during the course of the study or is currently pregnant or breastfeeding.
- 2. Plans to receive a licensed flavivirus vaccine or participate in another flavivirus vaccine trial during the study.
- 3. Has positive serology for HIV 1/2, Hepatitis C virus, or Hepatitis B surface antigen.
- 4. Has known or suspected congenital or acquired immunodeficiency, or recent history or current use of immunosuppressive therapy\*
  - \*Anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (at least 2 weeks within the previous 3 months) systemic corticosteroids therapy (at a dose of at least 0.5 mg/kg/day). Intranasal or topical prednisone (or equivalent) is allowed.
- 5. Had organ and/or stem cell transplantation whether or not on chronic immunosuppressive therapy.
- 6. Has history of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure\*.
  - \*Subjects with a history of skin cancer must not be vaccinated at the previous tumor site.
- 7. Has history of chronic or acute severe neurologic condition\*.
  - \*Including history of Guillain-Barre syndrome, seizure disorder or epilepsy, Bell's palsy, meningitis, or disease with any focal neurologic deficits.
- 8. Has diabetes mellitus type 1 or type 2, including cases controlled with diet alone.
  - \*Note: history of isolated gestational diabetes is not an exclusion criterion.
- 9. Has history of thyroidectomy, or thyroid disease requiring medication during the last 12 months.

- 10. Has major psychiatric illness during last 12 months that in the investigator's opinion would preclude participation.
- 11. Has history of other chronic disease or condition\*.
  - \*Includes the conditions and diagnoses defined as AESI in Section 9, as well as autoimmune disease, hypercholesterolemia, chronic hepatitis or cirrhosis, chronic pulmonary disease, chronic renal disease, and chronic cardiac disease including hypertension even if medically controlled
  - Vital signs must be normal by protocol toxicity grading scale or determined to be normal-variant by investigator. In the event of an abnormal heart rate or blood pressure due to physiological variation or activity, the subject may rest for 10 minutes in a quiet room, and then blood pressure and/or heart rate may be re-measured. Repeated vital signs may be used to determine eligibility.
- 12. Has current or past history of substance abuse that in the investigator's opinion would preclude participation.
- 13. Has tattoos, scars, or other marks on both deltoid areas that would, in the opinion of the investigator, interfere with assessment of the vaccination site.
- 14. Has a history of chronic urticaria (recurrent hives).
- 15. Has known allergy or history of anaphylaxis or other serious reaction to a vaccine or vaccine component\*.
  - \*Including aluminum hydroxide (alum) or aminoglycosides (e.g., neomycin and streptomycin).
- 16. Had major surgery (per the investigator's judgment) in the month prior to screening or plans to have major surgery during the study.
- 17. Received blood products or immunoglobulin in the 3 months prior to screening or planned use during the course of the study.
- 18. Donated a unit of blood within 8 weeks before Day 1 or plans to donate blood during the course of the study.
- 19. Received live attenuated vaccine from 30 days before Day 1 or plans to receive a live attenuated vaccine from Day 1 until 30 days after the last vaccination.
- 20. Received killed or inactivated vaccine from 14 days before Day 1 or plans to receive a killed or inactivated vaccine from Day 1 until 14 days after the last vaccination.
- 21. Received experimental therapeutic agents within 3 months prior to the first study vaccination or plans to receive any experimental therapeutic agents during the course of the study.
- 22. Is currently participating or plans to participate in another clinical study involving an investigational product, blood drawing, or an invasive procedure listed below.
  - \*An invasive procedure requiring administration of anesthetics or intravenous dyes or removal of tissue would be excluded. This includes endoscopy, bronchoscopy, or administration of IV contrast.
- 23. Has an acute illness or temperature ≥38.0°C on Day 1 or Day 29\* or within 2 days prior to vaccination.

- \*Subjects with fever or an acute illness on the day of vaccination or in the 2 days prior to vaccination may be re-assessed and enrolled if healthy or only minor residual symptoms remain within 2 days of Day 1 or Day 29.
- 24. Is a study site employee\* or staff paid entirely or partially by the OCRR contract or subcontract for the trial, or staff who are supervised by the PI or Sub-Investigators.
  - \*Including the Principal Investigator, sub-Investigators listed in Form FDA 1572 or Investigator of Record Form
- 25. In the investigator's opinion, the subject cannot communicate reliably, is unlikely to adhere to the study requirements, or has a condition that would limit their ability to complete the study.

### 4.4. Treatments

### 4.4.1. Treatments Administered

All subjects were to receive two doses of either 5 mcg ZPIV, 2.5 mcg ZPIV, or placebo administered intramuscularly 28 days apart.

### 4.4.2. Identity of Investigational Product(s)

ZPIV (Puerto Rico PRVABC59 strain), a formalin-inactivated whole virus vaccine produced by WRAIR, was administered in two intramuscular (IM) injections 28 days apart. Aluminum Hydroxide Adjuvant Alhydrogel® (aluminum hydroxide [or alum]) was used to adjuvant the ZPIV vaccine and to further dilute the adjuvanted vaccine for the 2.5 mcg dose. Use of alum as an adjuvant is well established and generally well tolerated.

### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Enrollment/randomization was performed through the enrollment module of AdvantageEDC, the electronic data capture system maintained by the SDCC. The list of randomized treatment assignments was prepared by statisticians at the SDCC and included in the enrollment module for this trial. The electronic data capture system assigned each subject a treatment code after the demographic and eligibility data have been entered into the system. A designated individual at each site was provided with a treatment key, which links the treatment code to the actual treatment assignment, to be kept in a secure place.

At the time of consent and upon entry of demographic data and confirmation of eligibility for this trial, the subject is enrolled. In group 1 (5 mcg ZPIV, N=45; placebo, N=5), two sentinel subjects were enrolled first and received ZPIV in an open-label fashion. All other subjects were randomized in a double-blind fashion. Upon completion of enrollment in Group 1, Group 2 subjects (2.5 mcg ZPIV, N=35; placebo, N=5) were randomized. Subjects received the same study product at their first and second investigational vaccinations.

### 4.4.4. Selection of Doses in the Study

Experience with licensed flavivirus vaccines suggests a 5 mcg dose should be safe and immunogenic; the 5 mcg dose was safe and protective in a NHP model [1]. Therefore, for this trial, subjects were enrolled initially in the 5 mcg group. To determine if lower doses of ZPIV are equally or comparably immunogenic to the 5 mcg dose, subjects were then enrolled in the 2.5 mcg group.

### 4.4.5. Selection and Timing of Dose for Each Subject

All subjects were scheduled to receive the assigned vaccination on Day 1 and Day 29  $(\pm 3)$ .

### 4.4.6. Blinding

This is a double-blinded study with the exception of the two sentinel subjects in Group 1. Non-sentinel subjects in Group 1, all subjects in Group 2, investigators, study personnel performing any study-related assessments following study vaccine administration, and laboratory personnel performing assays are blinded to study treatment within a group. The two sentinel subjects received open-label 5.0 mcg ZPIV (i.e., sentinels, investigators and study personnel were not blinded to sentinel study treatment). Laboratory testing personnel remain blinded to the identity and timepoint of individual samples.

The unblinded study vaccine administrator(s) is a study clinician credentialed to administer vaccines but is not involved in study-related assessments or have subject contact for data collection following study vaccine administration.

### 4.4.7. Prior and Concomitant Therapy

Assessment of study eligibility included a review of all permitted and prohibited medications per the subject inclusion and exclusion criteria. Prescription and over-the-counter drugs and vaccines were recorded, as well as herbals, vitamins, and supplements. Pre-study and concomitant use of any medications, therapies, or vaccines were reported. Medications included all current medications and non-study vaccinations taken within 30 days prior to signing the ICF through approximately Day 29 after the last study vaccination. Subjects who do not receive all study vaccinations would have concomitant medications collected through approximately Day 29 after the last study vaccination, or early termination, whichever occurs first. Subjects presenting with a history of AFI or ARI would have all concomitant medications taken since start of illness recorded.

Medications that might interfere with the evaluation of the investigational vaccine should not be used during the study period unless necessary. Medications in this category include the prohibited medications per the subject exclusion criteria. In addition, the site principal investigator or appropriate sub-investigator may identify other medications that should not be used due to a risk to subject safety or assessment of reactogenicity and immunogenicity. Use of medications as prophylaxis prior to study vaccination was prohibited.

### 4.4.8. Treatment Compliance

All subjects were to receive a prime dose of vaccine on Day 1 followed by a homologous boost on Day 29. All doses of vaccine were administered in the clinic by a vaccine administrator(s) credentialed to administer vaccines.

# 4.5. Immunogenicity and Safety Variables

In general, multiple observations within a specific visit period were accepted. In the case of multiple observations within a specific window, the assessment value closest to the scheduled visit date will be used in the analyses for the post-baseline records. If observations have the same distance to the scheduled assessment, the latest one will be used. Unless otherwise specified, the last assessment value recorded prior to the prime dose will be used as baseline. All the recorded data will be listed. Samples from days on which a subject was vaccinated were collected prior to vaccination.

All subjects were to have venous blood samples for assessment of humoral immunity collected on Days 1, 15, 29, 43, 57, 209, 388, and 569. Assay results are reported as the ZIKV titers giving 50% reduction in viral infection (MN50) and IgG ELISA titers. DENV neutralization titers were also to be recorded in subjects reporting ARI or AFI. Samples from the immunogenicity visits immediately before and after the illness visit were used to measure DENV titers, which will be used to aid laboratory confirmation of ZIKV/DENV infection.

Solicited adverse events were collected from the time of study vaccine administration through Day 8 after each dose. Subjects received a memory aid to record any solicited AEs on each day. The following injection site reactogenicity events were measured and grading according to the scale in Table 3 and Table 4: pain, tenderness, pruritis, ecchymosis, erythema, and induration. The following systemic solicited events were measured and graded according to the scale in Table 4 and Table 5: feverishness, fatigue, malaise, myalgia, arthralgia, headache, nausea, vomiting, diarrhea, abdominal pain, rash, and fever.

Vital signs of heart rate and blood pressure were measured in subjects at Days 1, 2, 8, 15, 29, 30, 36, 43, and 57. The measurements were assessed for adverse events of bradycardia/tachycardia and systolic and diastolic hypotension/hypertension according to the scale in Table 6.

Venous blood and urine were collected from subjects on Day 8 and Day 15 following each vaccination for safety clinical laboratory tests. The tests include WBC, hemoglobin, hematocrit, and platelets, ALT, AST, total bilirubin, BUN, creatinine, and urine dipstick for protein and glucose. Laboratory values were assessed for adverse events according to the grading scale in Table 7. Unsolicited adverse events were collected from all subjects through Day 57 (28 days after the 2<sup>nd</sup> vaccination). These events were assessed for severity and relatedness to study product. Serious adverse events (SAE), adverse events of special interest (AESI), and new onset chronic medical conditions (NOCMC) were collected for the duration of each subject's follow-up. Adverse events of special interest (AESI) for this study are neurologic and neuroinflammatory disorders collected through the duration of the subject's follow-up period.

Subjects were observed for development of an AFI/AFI and all related adverse events from the time of signing the informed consent form through follow-up. Subjects who reported an ARI/AFI were assessed for the following symptoms which are graded on a scale from 1 (least severe) to 3 (most severe): fever, feverishness, lethargy, restlessness, rash not at injection site, nonpurulent conjunctivitis, headache, shortness of breath, retino-orbital pain, myalgia, arthralgia, arthritis, nausea, abdominal pain, vomiting (evaluated for presence only), and bleeding (evaluated for presence only).

### 5. SAMPLE SIZE CONSIDERATIONS

The sample size for this study was selected to obtain preliminary estimates of vaccine safety and immunogenicity in a time sensitive manner. This study was not designed to test a specific null hypothesis. As this is a phase I study of ZPIV, it is primarily designed to collect initial information about safety and immune responses of two different doses of the vaccine.

The sample size in each dose cohort is small, thus the precision of estimates for AEs is limited. Rare AEs associated with dose are not demonstrable in a clinical study of this size; however, the probabilities of observing one or more AEs within a dose group at the minimum dose sample size of 35 and among the approximately 80 subjects receiving ZPIV are presented in Table 8. The minimum detectable event rates to achieve various levels of power are also displayed in Table 9.

If there are AEs associated with a particular dose of ZPIV, this study will have at least 80% power to observe at least one such event in a dose cohort if the true rate is 4.5%. If there are AEs associated with ZPIV overall, independent of dose, this study will have approximately 80% power to observe at least one such event in all ZIKV vaccine subjects if the true rate is 2.0%.

The study enrollment plan was modified in protocol amendment 5.0 (18 December 2018) to address the loss of evaluable subjects in Group 1 and delay of enrollment due to Hurricane Maria. The original study design planned to enroll 40 ZPIV recipients and 5 placebo recipients in each Group. Due to Hurricane Maria, 11 subjects enrolled in Group 1 had loss of samples at key timepoints. To rebalance the number of evaluable subjects between Groups, Group 1 enrollment was increased by 5 subjects and Group 2 enrollment was decreased by 5 subjects, for a total enrollment of 50 subjects in Group 1 and 40 in Group 2. Treatment assignments for both groups are assigned according to the originally planned 8:1 ratio of ZPIV:placebo.

### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, minimum and maximum, unless otherwise specified. The frequency and percentage of observed levels will be reported for all categorical measures; denominators for percentages will be defined for each analysis.

Listings will be provided for all data. Sort order will be specified on each listing shell in Appendix 3.

Summary tables will be structured with a column for each treatment group (2.5 mcg ZPIV, 5 mcg ZPIV, Placebo) and for all subjects for safety summaries.

All tables will be annotated with the total population size relevant to that table/group, including any missing observations.

# **6.2.** Timing of Analyses

This study has 3 planned interim analyses, all of which were to be performed on cleaned, monitored and locked datasets. The first two interim analyses were to consider safety, reactogenicity, and immunogenicity data and to take place at the following time points:

- The first interim analysis would take place after the last subject in Group 1 had been followed through 28 days post-second ZPIV administration (Day 57) and the first interim database had been locked.
- The second interim analysis would take place after the last subject in Group 2 had been followed through 28 days post-second ZPIV administration (Day 57) and the second interim database had been locked.
- The third interim analysis would describe the incidence and severity of AFI/ARI after all subjects had completed one-year follow-up after the 2<sup>nd</sup> vaccination.

The second and third interim analyses were performed at the same time, thus two separate interim analyses occurred prior to the CSR, dated 12DEC2018 and 22DEC2020. The analyses performed for the interim analyses were described in a separate Statistical Analysis Plan, "Interim Statistical Analysis Plan for DMID Protocol: 16-0034 v1.0" dated 01OCT2018.

The final analysis will be presented in the Clinical Study Report which will occur after all safety and protocol-specified humoral immunogenicity results, including all primary and secondary endpoint data, collected through Day 750 are available and the database has been locked. Given the urgency to obtain data in a timely manner, additional humoral and cellular immunogenicity assessments could be summarized in one or more addenda to the main CSR.

# **6.3.** Analysis Populations

Three analysis populations are defined: safety, immunogenicity, and per-protocol. In the case of misrandomization or treatment administration error, subjects in all analysis populations will be analyzed according to the study vaccine received.

### **6.3.1.** Safety Population

The Safety population will include all subjects who receive at least one study vaccination.

### 6.3.2. Immunogenicity (IMM) Population

The immunogenicity population will include all subjects who receive at least one study vaccination and contribute both pre- and at least one post-study vaccination sample for immunogenicity testing for which valid results are reported. Subjects with a loss of samples at pre-vaccination timepoints due to the natural disaster (i.e., Hurricane Maria) will be excluded from the GMFR and seroconversion analysis but will be included in post-baseline immunogenicity analyses where available. This population will be used for analysis of all immunogenicity data.

### 6.3.3. Per-Protocol (PP) Population

The Per Protocol (PP) population includes all subjects in the immunogenicity population with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent to major protocol deviations, such as:
  - Second vaccination not received,
  - Second vaccination received out of window,
  - Receipt of non-study licensed live vaccine within 30 days prior to or after each study vaccination,
  - Receipt of non-study licensed inactivated vaccine within 14 days prior to or after each study vaccination,
  - Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days prior to or after each study vaccination.
- Data from any visit that occurs substantially out of window.

The Per Protocol population may differ across post-vaccination visits and denominators will be the number of samples tested and included in the analysis at each visit.

# 6.4. Covariates and Subgroups

As well as treatment group, subjects will additionally be classified by baseline flavivirus immune status, defined primarily as follows:

- ZIKV Seropositive: any subject with detectable ZIKV antibodies pre-vaccination
- ZIKV Seronegative: any subject without detectable ZIKV antibodies pre-vaccination

Baseline flavivirus immune status will then be further classified into the following groups:

- ZIKV Seropositive and DENV Seropositive
- ZIKV Seropositive and DENV Seronegative
- ZIKV Seronegative and DENV Seropositive
- ZIKV Seronegative and DENV Seronegative

If a subject has inconclusive results for baseline flavivirus immune status, they will not be summarized with either subgroup defined above but will be included in summaries of all subjects pooled.

Subgroups based on baseline flavivirus immune status will be used in analysis of the secondary and exploratory endpoints only. For all tables and figures presenting group-aggregate analyses by subgroup—or any columns, rows, or panels within them—a single stratum must include at least two subjects in order to be generated.

### 6.5. Missing Data

No imputation will be performed for missing values. Missing data are assumed to be missing completely at random.

# 6.6. Interim Analyses and Data Monitoring

This study has 3 planned interim analyses as described in Section 6.2. Summaries described for the second and third interim reports were combined into a single report thus a total of 2 interim analyses were actually performed. The analyses performed for the interim analyses were described in "Interim Statistical Analysis Plan for DMID Protocol: 16-0034 v0.1." No unblinding of any individual subject treatment will be released in any interim analysis. Interim analyses will not include any formal hypothesis testing. They will, however, be made available to the study team and may impact the course of this study, be published, or be used in the planning of future studies.

### 6.7. Multicenter Studies

Not applicable.

# **6.8.** Multiple Comparisons/Multiplicity

No adjustments for multiple comparisons/multiplicity were planned.

### 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

A flowchart showing the disposition of study subjects, adapted from the CONSORT Statement will be included in Figure 1. This figure will present the number of subjects assesses for eligibility, randomized, terminated early, and included in the safety, immunogenicity, and per protocol populations. The CONSORT diagram will be presented by treatment group.

The disposition of subjects in the study will be tabulated by treatment group (Table 11). The table will include the number of subjects screened, enrolled/randomized, vaccinated, discontinued dosing, terminated early, completed follow-up and completed the study per-protocol. Listing 2 includes subjects who terminated early or discontinued from the study.

Between-group comparisons of the numbers of subjects overall and by baseline flavivirus status who withdrew early and the numbers who discontinued treatment (i.e., did not receive the second dose) will be presented in Table 12 using Fisher's exact 2-tailed test.

The number and percent of subjects excluded from each analysis population will be presented in Table 13 by treatment group and reason for exclusion. The number of subjects included in each immunogenicity summary will be presented in Table 14 by analysis population, treatment group, and immunogenicity time point. A listing of subjects excluded from analysis populations is available in Listing 5.

Dates of first treatment administration will be listed by treatment group in Table 15 and reasons for screen failure will be summarized in Table 16.

### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and treatment group for all subjects (Table 10). All subject-specific protocol deviations and non-subject-specific protocol deviations will be included as data listings (Listing 3 and Listing 4).

### 8. IMMUNOGENICITY EVALUATION

### 8.1. Primary Immunogenicity Analysis

Not applicable.

# 8.2. Secondary Immunogenicity Analyses

### 8.2.1. ZIKV Microneutralization Antibodies (MN50)

Seropositivity rates will be calculated based on ZIKV MN50 titers  $\geq$ 10 and  $\geq$ 100. Seroconversion rates will be calculated based on the number of subjects experiencing at least a 4-fold rise in ZIKV MN50 titers from baseline.

Geometric mean titer (GMT) and 95% CI for ZIKV MN50 results at each visit and for peak titer results will be summarized by treatment group overall and by baseline flavivirus immune status for the immunogenicity (IMM) population in Table 20 and per protocol (PP) population in Table 21.

Geometric mean fold rise from baseline (GMFR) and 95% CI results at each post-baseline visit and for each subject's peak ZIKV MN50 titer results will be summarized by treatment group overall and by baseline flavivirus immune status for the IMM population in Table 22 and PP population in Table 23.

Seropositivity rates and 95% CIs at each visit and for peak ZIKV MN50 titer results will be summarized by treatment group overall and by baseline flavivirus immune status for the IMM population in Table 24 and PP population in Table 25.

Seroconversion rates and 95% CI at each post-baseline visit and using peak titer results will be presented by treatment group overall and by baseline flavivirus immune status for the IMM population in Table 26 and PP population in Table 27. Denominators for percentages will be the number of subjects with non-missing data at the applicable time point and 95% CI will be calculated using Clopper-Pearson methodology from a binomial distribution.

Graphical presentations of immune response by treatment group and baseline flavivirus immune status will include reverse cumulative distribution curves (Figure 2 through Figure 11 and longitudinal presentation of GMTs (Figure 16 and Figure 17), seropositivity at a threshold of  $\geq$ 10 (Figure 18 and Figure 19), seropositivity at a threshold of  $\geq$ 100 (Figure 20 and Figure 21), and percent seroconversion (Figure 22 and Figure 23).

A listing of ZIKV MN50 titers by subject, treatment group, baseline flavivirus immune status, planned time point, and actual study day is presented in Listing 8.

### 8.2.2. ZIKV ELISA Antibodies

Seropositivity rates will be calculated based on ZIKV IgG ELISA titers ≥200 and ≥600. Seroconversion rates will be calculated based on the number of subjects experiencing at least a 4-fold rise in ZIKV IgG ELISA titers from baseline.

The analyses described in Section 8.2.1 will be repeated for ZIKV ELISA titers: GMT and 95% CI results are presented in Table 28 (IMM) and Table 29 (PP), GMFR and 95% CI results are presented in Table 30 (IMM) and Table 31 (PP), seropositivity rates and 95% CIs are presented in Table 32 (IMM) and Table 33 (PP), and seroconversion results and 95% CIs are presented in Table 34 (IMM) and Table 35 (PP). Denominators for percentages will be the number of subjects with non-missing data at

the applicable time point and 95% CI will be calculated using Clopper-Pearson methodology from a binomial distribution.

Graphical presentations of immune response by treatment group and baseline flavivirus immune status will include reverse cumulative distribution curves (Figure 24 through Figure 35) and longitudinal presentation of GMTs (Figure 38 and Figure 39), seropositivity at a threshold of  $\geq$ 200 (Figure 40 and Figure 41), seropositivity at a threshold of  $\geq$ 600 (Figure 42 and Figure 43), and percent seroconversion (Figure 44 and Figure 45).

A listing of ZIKV ELISA titers by subject, treatment group, baseline flavivirus immune status, planned time point, and actual study day is presented in Listing 8.

# 8.3. Exploratory Immunogenicity Analyses

Not applicable.

### 9. SAFETY EVALUATION

# 9.1. Demographic and Other Baseline Characteristics

Summaries of sex, ethnicity, race, baseline flavivirus immune status, age, and BMI will be presented by treatment group and overall (Table 17 and Table 18). In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the eCRF as "No" to each racial option.

### 9.1.1. Pre-Existing Medical Conditions

Pre-existing medical conditions will be summarized by MedDRA System Organ Class, treatment group and overall (Table 19). Individual subject listings will be presented for all demographics in Listing 6.

### 9.1.2. Prior and Concomitant Medications

Prior and concomitant medications will be summarized by WHO Drug Level 1 and Level 2 Codes, treatment group, and overall (Table 237). Individual subject listings will be presented for all concomitant medications (Listing 22).

# 9.2. Measurements of Treatment Compliance

All subjects were to receive 2 doses of investigational product administered in the clinic. The number of doses of investigational product administered to subjects will be presented by enrollment group as part of the subject disposition table (Table 11).

A listing of subjects who discontinued dosing and the reason will be included in Listing 2.

### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once per AE using the event with maximum severity and any repetitions of adverse events within a subject will be ignored; the denominator will be the total treatment group size or the corresponding number of subjects receiving the second dose, as appropriate. All unsolicited adverse events reported will be included in Listing 11.

An overall summary of adverse events from first administration of study vaccine to the end of the study is presented in Table 36, Table 37, and Table 38 for all subjects, baseline flavivirus positive subjects and baseline flavivirus negative subjects, respectively.

### 9.3.1. Solicited Events and Symptoms

Statistical comparisons of the frequency and duration of vaccine related Grade 3 local, systemic, or laboratory AE, and Grade 2 or greater local or systemic reactogenicity are presented post dose 1, post dose 2, and post any dose in Table 43, overall and by pre-vaccination flavivirus immune status. Frequencies of each adverse event are compared between dosage groups using Fisher's Exact test. The distribution of the duration of adverse events (excluding laboratory AEs) will be compared between all dosage groups using the 2-samples Wilcoxon rank sum test.

The frequency and proportion of subjects experiencing any local or systemic solicited event over the 8-day post-vaccination reporting period will be summarized by dose number, pre-vaccination flavivirus immune status, severity and treatment group in Table 44 (post dose 1, post dose 2, and post any dose).

The number, percentage, and exact 95% CI of subjects experiencing each solicited event over the 8-day post-vaccination reporting period, collected in-clinic pre-vaccination, post-vaccination and via memory aid, will be summarized by pre-vaccination flavivirus immune status, dose number and symptom in Table 45 (all subjects), Table 46 (baseline ZIKV seropositive subjects), Table 47 (baseline ZIKV seropositive subjects), Table 48 (baseline ZIKV seropositive and DENV seropositive subjects), Table 49 (baseline ZIKV seropositive and DENV seronegative subjects), Table 50 (baseline ZIKV seronegative and DENV seronegative subjects).

The frequency and proportion of subjects experiencing any mild, moderate, or severe solicited local or systemic reaction will be summarized by pre-vaccination flavivirus immune status, treatment group, dose number and reaction in Table 52 (local; all subjects), Table 53, (local; baseline ZIKV seropositive), Table 54 (local; baseline ZIKV seronegative), Table 55 (local; baseline ZIKV seropositive and DENV seropositive), Table 56 (local; baseline ZIKV seronegative), Table 57 (local; baseline ZIKV seronegative and DENV seropositive), Table 58 (local; baseline ZIKV seronegative and DENV seropositive), Table 60, (systemic; baseline ZIKV seropositive), Table 61 (systemic; baseline ZIKV seronegative), Table 62 (systemic; baseline ZIKV seropositive and DENV seropositive), Table 63 (systemic; baseline ZIKV seropositive), Table 64 (systemic; baseline ZIKV seronegative and DENV seropositive), and Table 65 (systemic; baseline ZIKV seronegative) DENV seronegative DENV seronegative DENV seronegative).

The frequency and proportion of subjects experiencing a mild, moderate, or severe **local or systemic solicited reaction** will be summarized by baseline flavivirus immune status, treatment group, dose number, reaction, pre-dose, and by post-vaccination day in the following tables:

Table A: Severity of Solicited Local or Systemic Reactogenicity Events, by Post-Vaccination Day:

| Baseline Flavivirus<br>Immune Status | 2.5 mcg ZIPV | | 5 mcg ZIPV | | | Placebo | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Post-Dose | Post-Dose 2 | Post Any<br>Dose | Post-Dose | Post-Dose 2 | Post Any<br>Dose | Post-Dose | Post-Dose 2 | Post Any<br>Dose |
| All Subjects | Table 66 | Table 67 | Table 68 | Table 69 | Table 70 | Table 71 | Table 72 | Table 73 | Table 74 |
| Baseline ZIKV<br>Seropositive | Table 75 | Table 76 | Table 77 | Table 78 | Table 79 | Table 80 | Table 81 | Table 82 | Table 83 |
| Baseline ZIKV<br>Seronegative | Table 84 | Table 85 | Table 86 | Table 87 | Table 88 | Table 89 | Table 90 | Table 91 | Table 92 |
| Baseline ZIKV<br>Seropositive and<br>DENV Seropositive | Table 93 | Table 94 | Table 95 | Table 96 | Table 97 | Table 98 | Table 99 | Table 100 | Table 101 |
| Baseline ZIKV<br>Seropositive and<br>DENV Seronegative | Table 102 | Table 103 | Table 104 | Table 105 | Table 106 | Table 107 | Table 108 | Table 109 | Table 110 |

| Baseline ZIKV<br>Seronegative and<br>DENV Seropositive | Table 111 | Table 112 | Table 113 | Table 114 | Table 115 | Table 116 | Table 117 | Table 118 | Table 119 |
|---|---|---|---|---|---|---|---|---|---|
| Baseline ZIKV<br>Seronegative and<br>DENV Seronegative | Table 120 | Table 121 | Table 122 | Table 123 | Table 124 | Table 125 | Table 126 | Table 127 | Table 128 |

Figure 46, Figure 47, and Figure 48 will summarize the solicited local adverse event data overall and by treatment group and display the maximum severity experience by each subject for each solicited event following any dose, post dose 1, and post dose 2, respectively. Similar summaries for solicited systemic events are presented in Figure 49, Figure 50, and Figure 51.

Figure 52, Figure 53, and Figure 54 will summarize the solicited local event data overall and by treatment group and display the maximum severity experienced by each subject pre-dose and each day post-dose, post any dose, post dose 1, and post dose 2, respectively. Figure 55, Figure 56, and Figure 57 are similar summaries for solicited systemic event data.

A listing of systemic and local solicited events is provided in Listing 9 and Listing 10, respectively.

### 9.3.2. Unsolicited Adverse Events

The frequency of all unsolicited AEs reported per subject from first administration of study vaccine to 28 days after the last vaccination are presented by MedDRA SOC, PT, severity, relationship to study treatment, and baseline flavivirus status in Table 129 (2.5 mcg ZPIV), Table 130 (5 mcg ZPIV), and Table 131 (placebo).

The frequency of all unsolicited AEs reported per subject from first administration of study vaccine to 28 days after the last vaccination are presented in the following tables by MedDRA SOC, PT, severity, dose, and baseline flavivirus status in Table 132 (2.5 mcg ZPIV), Table 133 (5 mcg ZPIV), and Table 134 (placebo).

Figure 58, Figure 59, and Figure 60 are graphical representations of the number and severity of all unsolicited adverse events overall and by treatment group and MedDRA SOC following any dose, post dose 1, and post dose 2, respectively. Similar presentations for adverse events determined to be related to study product are available in Figure 61, Figure 62, and Figure 63.

Refer to Listing 11 for a detailed listing of all unsolicited adverse events. Table 189 includes a listing of all serious adverse events and Table 190 includes a listing of all non-serious unsolicited moderate or severe adverse events.

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

Serious adverse events including deaths will be listed in Table 189. A listing of AESIs and NOCMCs will be presented in Table 191.

The number and percentage of subjects reporting new onset chronic medical conditions is summarized by MedDRA SOC and PT by treatment group and baseline flavivirus immune status in Table 135. Similar summaries for the number and percentage of subjects reporting AESIs related to study treatment are presented in Table 136. The duration in days of AESIs is summarized in Table 137.

Summaries of the number of subjects reporting serious adverse events related to study treatment are available in Table 138. The duration in days of the related SAEs is summarized in Table 139.

### 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt was made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. A listing of pregnancies and outcomes will be presented (Listing 20, Listing 24, Listing 25, Listing 26, and Listing 27).

### 9.6. Clinical Laboratory Evaluations

Safety laboratory tests include WBC, hemoglobin, hematocrit and platelets for hematology; ALT, AST, total bilirubin, BUN, and creatinine for chemistry; and urine dipstick for protein and glucose for urinalysis. Table 192 (chemistry), Table 193 (hematology) and Table 194 (urinalysis) are listings of all abnormal laboratory results.

The severity of clinical lab results by frequency and proportion of subjects for chemistry, hematology, and urinalysis clinical laboratory parameters conducted at screening (baseline) and Days 8, 15, 36, 43, and by maximum severity post-baseline are presented overall and by pre-vaccination flavivirus immune status and parameter as listed in Table B below.

The frequency and proportion of subjects with abnormal hematology, chemistry and urinalysis clinical laboratory parameters related to study treatment at each timepoint and by maximum severity post-baseline are presented by pre-vaccination flavivirus immune status and parameter as listed in Table C below.

Descriptive statistics of each hematology and chemistry clinical laboratory parameter at each scheduled time point, including change from baseline statistics, are presented by parameter as listed in Table D below.

Labs may also be performed as necessary at unscheduled visits for follow-up of an adverse event. Figure 64, Figure 65, and Figure 66 display abnormal results by laboratory parameter, severity, and treatment group and includes all values reported after treatment administration (scheduled and supplemental) for chemistry, hematology, and urinalysis labs, respectively. Mean changes from baseline at each scheduled time point for each chemistry and hematology lab are presented by treatment group in Figure 67 through Figure 75. Listing 17, Listing 18, and Listing 19 include listings of chemistry, hematology, and urinalysis results at any time post-treatment administration, respectively.

**Table B: Severity of Clinical Lab Results:** 

| Any Chemistry Parameter | Table 195 |
|--------------------------|-----------|
| ALT | Table 196 |
| AST | Table 197 |
| Total Bilirubin | Table 198 |
| BUN | Table 199 |
| Creatinine | Table 200 |
| Any Hematology Parameter | Table 212 |

| WBC | Table 213 |
|--------------------------|-----------|
| Hemoglobin | Table 214 |
| Hematocrit | Table 215 |
| Platelet Count | Table 216 |
| Any Urinalysis Parameter | Table 226 |
| Protein | Table 227 |
| Glucose | Table 228 |

Table C: Severity of Abnormal Clinical Lab Results Related to Study Treatment

| Any Chemistry Parameter | Table 201 |
|--------------------------|-----------|
| ALT | Table 202 |
| AST | Table 203 |
| Total Bilirubin | Table 204 |
| BUN | Table 205 |
| Creatinine | Table 206 |
| Any Hematology Parameter | Table 217 |
| WBC | Table 218 |
| Hemoglobin | Table 219 |
| Hematocrit | Table 220 |
| Platelet Count | Table 221 |
| Any Urinalysis Parameter | Table 229 |
| Protein | Table 230 |
| Glucose | Table 231 |

Table D: Descriptive Statistics of Chemistry and Hematology Clinical Lab Results

| | All Subjects |
|-----------------------------|--------------|
| <b>Chemistry Parameters</b> | |
| ALT | Table 207 |
| AST | Table 208 |
| Total Bilirubin | Table 209 |
| BUN | Table 210 |
| Creatinine | Table 211 |
| Hematology Parameters | |
| WBC | Table 222 |
|----------------|-----------|
| Hemoglobin | Table 223 |
| Hematocrit | Table 224 |
| Platelet Count | Table 225 |

## 9.7. Vital Signs and Physical Evaluations

Vital sign measurements included systolic blood pressure, diastolic blood pressure, pulse, and oral temperature. The frequency and proportion of subjects with abnormal vital signs results is presented by study visit, treatment group and severity in Table 232 (any assessment), Table 233 (oral temperature), Table 234 (pulse), Table 235 (systolic blood pressure) and Table 236 (diastolic blood pressure). Listing 20 includes a listing of vital signs at any time post-treatment administration; physical exam findings are presented in Listing 21.

### 9.8. Concomitant Medications

Concomitant medications will be summarized in Table 237 by WHO ATC Code Levels 1 and 2 and by treatment group. A listing of concomitant medications is presented in Listing 22.

### 9.9. Other Safety Measures

Summary tables of acute febrile illness (AFI) and acute rash illness (ARI) events will be presented. The percentage of subjects who develop ARI or AFI will be summarized by treatment group and baseline flavivirus status. Additionally, summary tables for AFI/ARI events will be presented by baseline flavivirus status.

Summaries of subjects reporting any events, any medically treated events, and any events requiring concomitant medication, including the total number of events and the number, percentage and exact 95% Clopper-Pearson CI of subjects reporting an event, will be presented for all subjects and by baseline flavivirus immune status in Table 140, Table 141, Table 142, Table 143, and Table 144. Similar summaries presented by infection confirmation method are presented in Table 147, Table 148, Table 149, Table 150 and Table 151.

Summaries of laboratory confirmed ZIKV and DENV infections are also presented. ZIKV and DENV infection is presented via two methods: subjects presenting with ARI/AFI and positive Arbovirus PCR result within 14 days of symptom onset or subjects presenting with ARI/AFI and a 4-fold rise in ZIKV or DENV titers following the onset of illness compared to prior to illness. The total number of laboratory confirmed ZIKV or DENV infections are summarized by treatment group, baseline flavivirus status, and confirmation method in Table 154, Table 155, Table 156, Table 157, and Table 158.

The distribution of the maximum severity of symptoms of each ARI/AFI event by baseline flavivirus status and treatment group will be presented in Table 161, Table 162, Table 163, Table 164, and Table 165, as well as by infection confirmation status in Table 168, Table 169, Table 170, Table 171, and Table 172. For subjects reporting at least one AFI/ARI the duration of reported symptoms will be described in Table 175, Table 176, Table 177, Table 178, Table 179, and by infection confirmation status in Table 182, Table 183, Table 184, Table 185, and Table 186.

Individual subject listings of AFI/ARI data will be included in Listing 12 (subject information), Listing 13 (medical treatment sought for ARI/AFI), Listing 14 (ARI/AFI symptoms), Listing 15 (vital signs), and Listing 16 (laboratory results).

# 10. PHARMACOKINETICS

Not applicable.

## 11. IMMUNOGENICITY

See Section 8.

# 12. OTHER ANALYSES

Not applicable.

### 13. REPORTING CONVENTIONS

P-values ≥0.001 and ≤0.999 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001" The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but <1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

# 14. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

The study enrollment plan was modified in protocol amendment 5.0 (18 December 2018) to address the loss of evaluable subjects in Group 1 and delay of enrollment due to Hurricane Maria. The original study design planned to enroll 40 ZPIV recipients and 5 placebo recipients in each Group. Due to Hurricane Maria, 11 subjects enrolled in Group 1 had loss of samples at key timepoints. To rebalance the number of evaluable subjects between Groups, Group 1 enrollment was increased by 5 subjects and Group 2 enrollment was decreased by 5 subjects, for a total enrollment of 50 subjects in Group 1 and 40 in Group 2. Treatment assignments for both groups are assigned according to the originally planned 8:1 ratio of ZPIV:placebo.

The data summaries described for the second and third interim analyses were combined into a single interim analysis. Therefore, only two interim analyses were actually performed prior to final database lock and the clinical study report.

Baseline flavivirus screening was expanded from testing for ZIKV and DENV antibodies to testing for antibodies to 4 flaviviruses: ZIKV, DENV, YFV, and WNV. Results of baseline YFV and WNV testing will not be used in analysis for the CSR.

The second exploratory endpoint was modified in protocol version 6.0 (06 December 2021) to clarify how ZIKV and DENV infection would be confirmed in subjects reporting AFI/ARI. The timepoints were adjusted to run ZIKV and DENV MN50 on samples immediately before and immediately following the illness visit(s) wherever possible.

#### 16. REFERENCES

- 1. Abbink, P et al (2016). Protective Efficacy of Multiple Vaccine Platforms Against Zika Virus Challenge in Rhesus Macaques. *Science*, Epub ahead of print
- 2. Atkinson B, H. P. (2016 May). Detection of Zika virus in semen (letter). *Emerging Infectious Diseases Vol 22*.
- 3. Broutet N, K. F. (2016). Zika Virus as a Cause of Neurologic Disorders. NEJM 374, 1506-1509.
- 4. Calvetg, a. R. (2016). Detection and sequencing of ZIKA virus from amniotic fluid of fetuses with microcephaly in Brazil: a case study. *Lancet Infectious Disease*, Epub ahead of print.
- 5. Cao-Lormeau, V.-M. e. (2016). Guillain-Barré Syndrome outbreak associated with Zika virus infection in French Polynesia: a case-control study. *The Lancet Vol 387*, 1051-1052.6. Carteaux, G, et al (2016). Zika Virus Associated with Meningoencephalitis. *NEJM*, 374, 1595.
- 6. D'Ortenzio E, M. S. (2016). Evidence of sexual Transmission of Zika virus. NEJM, epub.
- 7. Duffy, M. C. (2016). Zika Virus Outbreak on Yap Island, Federated States of Micronesia. *NEJM*, 2536-2543.
- 8. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.
- 9. Dupont-Rouzeyrol, M. e. (2016). Infectious Zika viral particles in breastmilk. *The Lancet* 387,1051.
- 10. Larocca, RA (2016). Vaccine Protection against Zika virus from Brazil. *Nature* doi:10.1038/nature18952.
- 11. Martinez LJ, L. L. (2015). Safety and Immunogenicity of a Dengue Virus Serotype-1 Purified Inactivated Vaccine: Results of a Phase 1 Clinical Trial. *Am. J. Trop. Med Hyg 93*:, 454-460.
- 12. Rasmussen SA, J. D. (2016). Zika Virus and Birth Defects- Reviewing the Evidence for Causality. *NEJM*, sr1604338.
- 13. Valnera Austria GmBH. (2015, August). IXIARO Prescribing Information

## 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

### **APPENDICES**

## APPENDIX 1. TABLE MOCK-UPS

## LIST OF TABLES

| Table 1: | Schematic of Study Design |
|---|---|
| Table 2: | Schedule of Study Procedures |
| Table 3: | Local (Injection Site) Reactogenicity and Measurement |
| Table 4: | Subjective Systemic Reactogenicity Grading60 |
| Table 5: | Quantitative Systemic Reactogenicity Grading61 |
| Table 6: | Vital Sign Adverse Event Grading Scale |
| Table 7: | Laboratory Adverse Event Grading Scale |
| Table 8: | Probability of Observing at Least One Adverse Event Given Various True Event Rates |
| | 64 |
| Table 9: | Minimum Detectable Event Rates given various levels of Power65 |
| Table 10: | Distribution of Protocol Deviations by Category, Type, and Treatment Group, All Enrolled Subjects |
| Table 11: | Subject Disposition by Treatment Group68 |
| Table 12: | Early Withdrawals and Treatment Discontinuations by Treatment Group – All Enrolled and Randomized Subjects |
| Table 13: | Analysis Populations by Treatment Group70 |
| Table 14: | Number of Subjects in Immunogenicity and Per Protocol Populations with Data Available by Analysis Type, Time Point, and Treatment Group73 |
| Table 15: | Date of First Treatment by Treatment Group74 |
| Table 16: | Ineligibility Summary of Screen Failures |
| Table 17: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group |
| Table 18: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group – Safety Population |
| Table 19: | Summary of Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group |
| Table 20: | ZIKV Microneutralization Antibody (MN50) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population |
| Table 21: | ZIKV Microneutralization Antibody (MN50) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population |
| Table 22: | ZIKV Microneutralization Antibody (MN50) Geometric Mean Fold Rise (GMFR) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population80 |

| Table 23: | ZIKV Microneutralization Antibody (MN50) Geometric Mean Fold Rise (GMFR) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population80 |
|---|---|
| Table 24: | ZIKV Microneutralization Antibody (MN50) Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population |
| Table 25: | ZIKV Microneutralization Antibody (MN50) Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population |
| Table 26: | ZIKV Microneutralization Antibody (MN50) Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population |
| Table 27: | ZIKV Microneutralization Antibody (MN50) Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population |
| Table 28: | ZIKV ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population |
| Table 29: | ZIKV ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population |
| Table 30: | ZIKV ELISA Geometric Mean Fold Rise (GMFR) Results with 95% Confidence<br>Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status –<br>Immunogenicity Population |
| Table 31: | ZIKV ELISA Geometric Mean Fold Rise (GMFR) Results with 95% Confidence<br>Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per<br>Protocol Population |
| Table 32: | ZIKV ELISA Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population |
| Table 33: | ZIKV ELISA Seropositivity Results with 95% Confidence Intervals by Time Point,<br>Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population85 |
| Table 34: | ZIKV ELISA Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population |
| Table 35: | ZIKV ELISA Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population85 |
| Table 36: | Overall Summary of Adverse Events – All Subjects |
| Table 37: | Overall Summary of Adverse Events – Baseline ZIKV Seropositive Subjects88 |
| Table 38: | Overall Summary of Adverse Events – Baseline ZIKV Seronegative Subjects88 |

| Table 39: | Overall Summary of Adverse Events – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
|---|---|
| Table 40: | Overall Summary of Adverse Events – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 41: | Overall Summary of Adverse Events – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 42: | Overall Summary of Adverse Events – Baseline ZIKV Seronegative and DENV Seronegative Subjects |
| Table 43: | Comparison of the Frequency, Type and Duration of Vaccine-Related Grade 3 Local, Systemic or Laboratory AEs and Grade 2 or Greater Local or Systemic Reactogenicity Through Day 8 Post Vaccination |
| Table 44: | Number and Percentage of Subjects Experiencing Any Local or Systemic Solicited Events through Day 8 Post Vaccination by Dose, Baseline Flavivirus Immune Status, Severity and Treatment Group |
| Table 45: | Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – All Subjects |
| Table 46: | Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seropositive Subjects |
| Table 47: | Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seronegative Subjects |
| Table 48: | Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects96 |
| Table 49: | Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative |
| Table 50: | Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive |
| Table 51: | Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative |
| Table 52: | Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity and Treatment Group – All Subjects97 |
| Table 53: | Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive Subjects98 |

| Table 54: | Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative Subjects98 |
|---|---|
| Table 55: | Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
| Table 56: | Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 57: | Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 58: | Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects |
| Table 59: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – All Subjects |
| Table 60: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive Subjects 100 |
| Table 61: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative Subjects 100 |
| Table 62: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
| Table 63: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 64: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 65: | Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects |
| Table 66: | Number and Percentage of Subjects Experiencing Solicited Local or Systemic Events by Symptom, Severity, and Day Post Dosing – 2.5 mcg ZPIV – Post Dose 1101 |
| Table 67: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 2.5 mcg ZPIV – Post Dose 2 |
| Table 68: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 2.5 mcg ZPIV – Post Any Dose |
| Table 69: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 5 mcg ZPIV – Post Dose 1 |

| Table 70: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 5 mcg ZPIV – Post Dose 2 |
|---|---|
| Table 71: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 5 mcg ZPIV – Post Any Dose103 |
| Table 72: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Placebo – Post Dose 1 |
| Table 73: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Placebo – Post Dose 2 |
| Table 74: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Placebo – Post Any Dose |
| Table 75: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 2.5 mcg ZPIV –<br>Post Dose 1 |
| Table 76: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 2.5 mcg ZPIV –<br>Post Dose 2 |
| Table 77: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 2.5 mcg ZPIV –<br>Post Any Dose |
| Table 78: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 5 mcg ZPIV –<br>Post Dose 1 |
| Table 79: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 5 mcg ZPIV –<br>Post Dose 2 |
| Table 80: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 5 mcg ZPIV –<br>Post Any Dose |
| Table 81: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – Placebo – Post<br>Dose 1 |
| Table 82: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – Placebo – Post<br>Dose 2 |
| Table 83: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – Placebo – Post<br>Any Dose |
| Table 84: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 2.5 mcg ZPIV –<br>Post Dose 1 |

| Table 85: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 2.5 mcg ZPIV<br>Post Dose 2 |
|---|---|
| Table 86: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 2.5 mcg ZPIV Post Any Dose |
| Table 87: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 5 mcg ZPIV – Post Dose 1 |
| Table 88: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 5 mcg ZPIV – Post Dose 2 |
| Table 89: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 5 mcg ZPIV – Post Any Dose |
| Table 90: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – Placebo – Post<br>Dose 1 |
| Table 91: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – Placebo – Post<br>Dose 2 |
| Table 92: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – Placebo – Post<br>Any Dose |
| Table 93: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 1 |
| Table 94: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 2 |
| Table 95: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Any Dose |
| Table 96: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 1 |
| Table 97: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 2 |

| Table 98: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 5 mcg ZPIV – Post Any Dose |
|---|---|
| Table 99: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Placebo – Post Dose 1 |
| Table 100: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Placebo – Post Dose 2 |
| Table 101: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Placebo – Post Any Dose |
| Table 102: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 1 |
| Table 103: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 2 |
| Table 104: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Any Dose |
| Table 105: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 5 mcg ZPIV – Post Dose 1 |
| Table 106: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 5 mcg ZPIV – Post Dose 2 |
| Table 107: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 5 mcg ZPIV – Post Any Dose |
| Table 108: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – Placebo – Post Dose 1 |
| Table 109: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – Placebo – Post Dose 2 |
| Table 110: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – Placebo – Post Any Dose |

| Table 111: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 1 |
|---|---|
| Table 112: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 2 |
| Table 113: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Any Dose |
| Table 114: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 1 |
| Table 115: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 2 |
| Table 116: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 5 mcg ZPIV – Post Any Dose |
| Table 117: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – Placebo – Post Dose 1 |
| Table 118: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – Placebo – Post Dose 2 |
| Table 119: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – Placebo – Post Any Dose |
| Table 120: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 1 |
| Table 121: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 2 |
| Table 122: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Any Dose |
| Table 123: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 5 mcg ZPIV – Post Dose 1 |

| Table 124: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative<br>Subjects – 5 mcg ZPIV – Post Dose 2 |
|---|---|
| Table 125: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative<br>Subjects – 5 mcg ZPIV – Post Any Dose |
| Table 126: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative<br>Subjects – Placebo – Post Dose 1 |
| Table 127: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative<br>Subjects – Placebo – Post Dose 2 |
| Table 128: | Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,<br>Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative<br>Subjects – Placebo – Post Any Dose |
| Table 129: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship to Study Treatment, and Baseline Flavivirus Immune Status – 2.5 mcg ZPIV116 |
| Table 130: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship to Study Treatment, and Baseline Flavivirus Immune Status – 5 mcg ZPIV117 |
| Table 131: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship to Study Treatment, and Baseline Flavivirus Immune Status – Placebo |
| Table 132: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class, Preferred Term, Severity, Dose, and Baseline Flavivirus Immune Status – 2.5 mcg ZPIV |
| Table 133: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class, Preferred Term, Severity, Dose, and Baseline Flavivirus Immune Status – 5 mcg ZPIV |
| Table 134: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class, Preferred Term, Severity, Dose, and Baseline Flavivirus Immune Status – Placebo |
| Table 135: | Number and Percentage of Subjects Reporting NOCMCs by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status.121 |
| Table 136: | Number and Percentage of Subjects Reporting AESIs Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status |
| Table 137: | Duration (Days) of AESIs Related to Study Treatment by MedDRA System Organ Class<br>Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status123 |

| Table 138: | Number and Percentage of Subjects Reporting Serious Adverse Events Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status |
|---|---|
| Table 139: | Duration (Days) of Serious Adverse Events Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status |
| Table 140: | Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – All Subjects |
| Table 141: | Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seropositive Subjects |
| Table 142: | Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative Subjects |
| Table 143: | Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects125 |
| Table 144: | Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects125 |
| Table 145: | Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects125 |
| Table 146: | Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects126 |
| Table 147: | Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – All Subjects |
| Table 148: | Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – Baseline ZIKV Seropositive Subjects |
| Table 149: | Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – Baseline ZIKV Seronegative Subjects |
| Table 150: | Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
| Table 151: | Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 152: | Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 153: | Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – Baseline ZIKV Seronegative and DENV Seronegative Subjects |

| Table 154: | Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – All Subjects129 |
|---|---|
| Table 155: | Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – Baseline ZIKV Seropositive Subjects |
| Table 156: | Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – Baseline ZIKV Seronegative Subjects |
| Table 157: | Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
| Table 158: | Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 159: | Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 160: | Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – Baseline ZIKV Seronegative and DENV Seronegative Subjects |
| Table 161: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – All Subjects |
| Table 162: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seropositive Subjects132 |
| Table 163: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative Subjects132 |
| Table 164: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
| Table 165: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 166: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 167: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects |

| Table 168: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – All Subjects |
|---|---|
| Table 169: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – Baseline ZIKV Seropositive Subjects |
| Table 170: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – Baseline ZIKV Seronegative Subjects |
| Table 171: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
| Table 172: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 173: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 174: | Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects134 |
| Table 175: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post<br>Final Vaccination by Treatment Group – All Subjects |
| Table 176: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post<br>Final Vaccination by Treatment Group – Baseline ZIKV Seropositive Subjects136 |
| Table 177: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative Subjects136 |
| Table 178: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post<br>Final Vaccination by Treatment Group – Baseline ZIKV Seropositive and DENV<br>Seropositive Subjects |
| Table 179: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post<br>Final Vaccination by Treatment Group – Baseline ZIKV Seropositive and DENV<br>Seronegative Subjects |
| Table 180: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 181: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects |

| Table 182: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post<br>Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation<br>Status – All Subjects |
|---|---|
| Table 183: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post<br>Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation<br>Status – Baseline ZIKV Seropositive Subjects |
| Table 184: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post<br>Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation<br>Status – Baseline ZIKV Seronegative Subjects |
| Table 185: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status – Baseline ZIKV Seropositive and DENV Seropositive Subjects |
| Table 186: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status – Baseline ZIKV Seropositive and DENV Seronegative Subjects |
| Table 187: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status – Baseline ZIKV Seronegative and DENV Seropositive Subjects |
| Table 188: | Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status – Baseline ZIKV Seronegative and DENV Seronegative Subjects |
| Table 189: | Listing of Serious Adverse Events |
| Table 190: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events141 |
| Table 191: | Listing of AESIs and NOCMCs |
| Table 192: | Listing of Abnormal Laboratory Results – Chemistry |
| Table 193: | Listing of Abnormal Laboratory Results – Hematology145 |
| Table 194: | Listing of Abnormal Laboratory Results – Urinalysis |
| Table 195: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Chemistry Parameter |
| Table 196: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – ALT |
| Table 197: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – AST |
| Table 198: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Total Bilirubin |
| Table 199: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – BUN |
| Table 200: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline |

| Table 201: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Chemistry Parameter |
|---|---|
| Table 202: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – ALT149 |
| Table 203: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – AST149 |
| Table 204: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Total Bilirubin149 |
| Table 205: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – BUN149 |
| Table 206: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Creatinine149 |
| Table 207: | Laboratory Summary Statistics by Time Point and Treatment Group – ALT150 |
| Table 208: | Laboratory Summary Statistics by Time Point and Treatment Group – AST151 |
| Table 209: | Laboratory Summary Statistics by Time Point and Treatment Group – Total Bilirubin |
| Table 210: | Laboratory Summary Statistics by Time Point and Treatment Group – BUN151 |
| Table 211: | Laboratory Summary Statistics by Time Point and Treatment Group – Creatinine.151 |
| Table 212: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Hematology Parameter |
| Table 213: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – WBC |
| Table 214: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status– Hemoglobin |
| Table 215: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status– Hematocrit |
| Table 216: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status– Platelet Count |
| Table 217: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Hematology Parameter |
| Table 218: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status—WBC156 |
| Table 219: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Hemoglobin157 |
| Table 220: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Hematocrit157 |

| Table 221: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Platelet Count.157 |
|---|---|
| Table 222: | Laboratory Summary Statistics by Time Point and Treatment Group – WBC158 |
| Table 223: | Laboratory Summary Statistics by Time Point and Treatment Group – Hemoglobin158 |
| Table 224: | Laboratory Summary Statistics by Time Point and Treatment Group – Hematocrit158 |
| Table 225: | Laboratory Summary Statistics by Time Point and Treatment Group – Platelet Count158 |
| Table 226: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Urinalysis Parameter |
| Table 227: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Urine Protein |
| Table 228: | Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status– Urine Glucose |
| Table 229: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Urinalysis Parameter |
| Table 230: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Urine Protein160 |
| Table 231: | Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Urine Glucose 160 |
| Table 232: | Vital Signs by Maximum Severity, Time Point and Treatment Group – Any Assessment |
| Table 233: | Vital Signs by Maximum Severity, Time Point and Treatment Group – Oral Temperature |
| Table 234: | Vital Signs by Maximum Severity, Time Point and Treatment Group – Pulse162 |
| Table 235: | Vital Signs by Maximum Severity, Time Point and Treatment Group – Systolic Blood Pressure |
| Table 236: | Vital Signs by Maximum Severity, Time Point and Treatment Group – Diastolic Blood<br>Pressure |
| Table 237: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group |

Table 1: Schematic of Study Design

| Dosage Group | Approximate # of<br>Subjects<br>(8:1 ratio) | Treatment at Days 1 and 29 |
|---|---|---|
| Group 1 Sentinels | 2 | 5 mcg ZPIV |
| Group 1 Non-Sentinels | 43 | 5 mcg ZPIV |
| | 5 | Placebo |
| Group 2 | 35 | 2.5 mcg ZPIV |
| | 5 | Placebo |

**Table 2:** Schedule of Study Procedures

| Study Visit | V00 | V0<br>1 | V02 | V03 | V0<br>4 | V05 | V06 | V07 | V08 | V09 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 | Fever/<br>Rash | Early<br>Term | Unsch<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Overall Study Day | Screen<br>D-28 to1 | D1 Vaccination | D2 | D4 +1<br>Phone call | D8 ±1 | D15±1 | D29 ±3 | D30 | D32 +1<br>Phone call | D36±1 | D43±2 | D57±3 | D107 ± 14<br>Phone call | D157±14 Phone call | D209 ±14 | D268 ±14 Phone<br>Call | D328 ±14<br>Phone call | D388 ±14 | | | |
| Study Day after Second<br>Vaccination | | | | | | | D1 Vaccination 2 | D2 | D4+1<br>Phone call | D8 ±1 | D15 ±2 | D29 ±3 | D79±14 Phone call | D129±14 Phone call | D181 ±14 | D240 <u>+</u> 14 Phone call | D300 ±14 Phone call | D360 ±14 | | | |
| Informed Consent <sup>1</sup> | X | | | | | | | | | | | | | | | | | | | | |
| Review Eligibility | X | X | | | | | X | | | | | | | | | | | | | | |
| Medical History <sup>3</sup> | X | $X^2$ | X | X | X | X | $X^2$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital Signs (T,P,& BP) <sup>5</sup> | X | X | X | | X | X | X | X | | X | X | X | | | | | | | X | $X^{15}$ | $X^{15}$ |
| Height & Weight | X | | | | | | | | | | | | | | | | | | | | |
| Abbreviated Physical Exam <sup>6</sup> | X | | | | | | | | | | | | | | | | | | | | |
| Serology (HIV-1/2, HBV, HCV) | X | | | | | | | | | | | | | | | | | | | | |
| Serology (ZIKV, DENV) | X | | | | | | | | | | | | | | | | | | X <sup>19</sup> | | |
| Randomization/<br>Enrollment | | X | | | | | | | | | | | | | | | | | | | |
| Evaluate Pre-<br>administration<br>reactogenicity | | X | | | | | X | | | | | | | | | | | | | | |
| Study Product<br>Administration and<br>observation for 30 minutes | | X | | | | | X | | | | | | | | | | | | | | |

**Table 2: Schedule of Study Procedures (***continued***)** 

| Study Visit | V00 | V0<br>1 | V02 | V03 | V0<br>4 | V05 | V06 | V07 | V08 | V09 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 | Fever/<br>Rash | Early<br>Term | Unsch<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Give Memory Aid <sup>9</sup> | | X | | | | | X | | | | | | | | | | | | | | |
| Evaluate vaccine site <sup>11</sup> | | X | X | | X | X | X | X | | X | X | X | | | | | | | | $X^{13}$ | $X^{13}$ |
| Targeted Physical Exam <sup>6</sup> | | X | X | | X | X | X | X | | X | X | X | | | X | | | X | X | X | X |
| Serum or Urine Pregnancy<br>Test <sup>7</sup> | X | X | | | | | X | | | | | X | | | | | | | | X <sup>13</sup> | X <sup>13</sup> |
| Safety Lab Evaluations <sup>8</sup> | X | | | | X | X | | | | X | X | | | | | | | | | X <sup>14</sup> | X <sup>14</sup> |
| Urine for protein and glucose | X | | | | X | X | | | | X | X | | | | | | | | | X <sup>14</sup> | X <sup>14</sup> |
| Concomitant Medications | X | X | X | X | X | X | $X^2$ | X | X | X | X | X | | | | | | | X | X | X |
| Review Memory Aid | | | X | X | X | | | X | X | X | | | | | | | | | | $X^{12}$ | $X^{12}$ |
| AE Collection | | X | X | X | X | X | X | X | X | X | X | X | | | | | | | X | $X^{15}$ | X <sup>15</sup> |
| AFI/ARI/ SAE/AESI/new medical conditions <sup>22, 20</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum for Humoral<br>Immunity | | X <sup>1</sup> 6 | | | | X | X <sup>16</sup> | | | | X | X | | | X | | | X | | X <sup>17</sup> | X <sup>17</sup> |
| CPT tubes for future immunity/systems biology <sup>21</sup> | | X <sup>1</sup> 6,1 8, | X <sup>18</sup> | | X <sup>1</sup> <sub>8</sub> | X <sup>18</sup> | X <sup>16</sup> | X <sup>18</sup> | | X <sup>18</sup> | X <sup>18</sup> | X | | | X | | | X | | X <sup>17</sup> | X <sup>17</sup> |
| Paxgene tubes for future systems biology | | $X^1$ | X | | X | X | X <sup>16</sup> | X | | X | X | | | | | | | | | X <sup>17</sup> | X <sup>17</sup> |
| AFI/ARI /SAE/AESI/new medical conditions <sup>22, 20</sup> | X | X | X | X | X | X | | | | | | | | | | | | | | | |
| Medical History <sup>3</sup> | X | X | X | X | X | X | | | | | | | | | | | | | | | |

### **Table 2: Schedule of Study Procedures (***continued***)**

| Study Visit | V00 | V0<br>1 | V02 | V03 | V0<br>4 | V05 | V06 | V07 | V08 | V09 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 | Fever/<br>Rash | Early<br>Term | Unsch<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Serum for Humoral<br>Immunity | | | X | | | X | | | | | | | | | | | | | | | |
| CPT tubes for future immunity/systems biology | | | X | | | X | | | | | | | | | | | | | | | |
| Targeted Physical exam <sup>6</sup> | | | X | | | X | | | | | | | | | | | | | | | |

### Table 2: Schedule of Study Procedures (continued)

| Study Visit | V00 | V0<br>1 | V02 | V03 | V0<br>4 | V05 | V06 | V07 | V08 | V09 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 | Fever/<br>Rash | Early<br>Term | Unsch<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

Definitions: AE = adverse event; BP = blood pressure; DENV = dengue virus; HBV = hepatitis B virus; HCV = hepatitis C virus; HIV 1/2 = human immunodeficiency virus types 1 and 2; HR = heart rate; T = body temperature; SAE = serious adverse event; AESI = Adverse event of Special Interest; ZIKV = Zika virus.

<sup>&</sup>lt;sup>1</sup> Must describe study, administer informed consent, and have informed consent form (ICF) signed prior to initiation of any study-related procedures.

<sup>&</sup>lt;sup>2</sup> Subjects must meet eligibility criteria; these criteria should be reviewed prior to administration of prime and boost dose of study vaccine or placebo.

<sup>&</sup>lt;sup>3</sup> Obtain complete medical history from subject at first screening visit and update it at Day 1 prior to vaccination; interim medical history obtained at follow-up visits.

<sup>&</sup>lt;sup>5</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature. Repeat of vital signs allowed once if found to be abnormal on Day 1 and Day 29.

<sup>&</sup>lt;sup>6</sup> Abbreviated physical examination is a complete exam with no genitourinary and rectal exam performed. Targeted physical exams are done at scheduled clinic visits if indicated based on review of medical history.

<sup>&</sup>lt;sup>7</sup> Females of childbearing potential will have serum pregnancy test done at screening and urine pregnancy test done in the 24 hours prior to each study vaccination; Results must be negative to enroll subject and negative prior to each study vaccination. Urine pregnancy test may be done if subject withdrawals from study early or has an unscheduled visit.

<sup>&</sup>lt;sup>8</sup> Screening laboratory tests, including WBC, hemoglobin, hematocrit, platelet count, ALT, AST, bilirubin, BUN, and creatinine, may be repeated once on a second screening visit If test is out of acceptable range, provided there is an alternative explanation for the out of range value; All screening tests need to be done within 28 days of Day 1, otherwise all tests, except for serology for HIV 1/2, Hepatitis C virus, or Hepatitis B surface antigen, will need to be repeated within the screening period. Safety laboratories include WBC, hemoglobin, hematocrit, platelet count, ALT, AST, bilirubin, BUN, and creatinine.

<sup>&</sup>lt;sup>9</sup> Distribute memory aid to subjects and give them study materials.

<sup>&</sup>lt;sup>11</sup> Assess vaccination site.

<sup>&</sup>lt;sup>12</sup> If visit occurs <8 days after 1<sup>st</sup> of 2<sup>nd</sup> vaccination. Includes local and systemic reactogenicity assessment

<sup>&</sup>lt;sup>13</sup> If prior to <28 days after the last study vaccination.

<sup>&</sup>lt;sup>14</sup> If visit occurs <15 days after 1<sup>st</sup> or 2<sup>nd</sup> vaccination.

<sup>&</sup>lt;sup>15</sup> If visit occurs on or prior to Day 57.

<sup>&</sup>lt;sup>16</sup> Obtained prior to vaccination.

<sup>&</sup>lt;sup>17</sup> If visit occurs within window of a study Day when these labs would be collected.

<sup>&</sup>lt;sup>18</sup> Part of the plasma from the CPT tubes will be saved for systems biology.

<sup>&</sup>lt;sup>19</sup> Baseline serology will include testing for DENV and ZIKV. AFI/ARI assessment will include testing for DENV, ZIKV, and CHIKV.

Table 3: Local (Injection Site) Reactogenicity and Measurement

| Reactogenicity | Mild | Moderate | Severe |
|---|---|---|---|
| | (Grade 1) | (Grade 2) | (Grade 3) |
| Local reactions | | | |
| Pain | Does not interfere with activity <b>and</b> no pain medication is taken | Repeated use of non-narcotic pain reliever >24 hours <b>or</b> interferes with activity | Any use of narcotic pain reliever <b>or</b> prevents daily activity |
| Tenderness | Discomfort only to touch | Discomfort with movement and it interferes with daily activity | Significant discomfort at rest <b>and</b> it prevents daily activity |
| Pruritis (itching) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Ecchymosis (bruising) <sup>a</sup> | 25-50 mm | 51-100 mm | >100 mm |
| Erythema (redness) <sup>a</sup> | 25-50 mm | 51-100 mm | >100 mm |
| Induration (hardness)/swelling <sup>b</sup> | 25-50 mm and does not interfere with activity | 51-100 mm <b>or</b> interferes with activity | >100 mm or prevents daily activity |

<sup>&</sup>lt;sup>a</sup> In addition to grading the measured local reaction at the greatest single diameter, the measurement should be recorded as a continuous variable. The size of erythema, ecchymosis, and induration/swelling by itself will not be used as halting criteria.

<sup>&</sup>lt;sup>b</sup> Induration/swelling should be evaluated and graded using the functional scale as well as the actual measurement.

 Table 4:
 Subjective Systemic Reactogenicity Grading

| Some interference with daily activity Some interference with daily activity Some interference with daily activity or it requires > 24 hours of use of non-narcotic Significant interference, prevents daily activity or it requires any use of narcotic |
|---|
| activity or it requires > 24 prevents daily activity or it requires any use of narcotic |
| pain medication pain medication |
| Some interference with daily Significant interference, |
| activity prevents daily activity |

**Table 5:** Quantitative Systemic Reactogenicity Grading

| Systemic (Quantitative) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Fever# - oral† | 38.0°C – 38.4°C | 38.5°C – 38.9°C | >38.9°C |
| | $100.4^{\circ}F - 101.1^{\circ}F$ | $101.2^{\circ}F - 102.0^{\circ}F$ | >102.0°F |

Oral temperature assessed on Day 1 prior to the first study vaccination will be considered as baseline.

<sup>&</sup>lt;sup>#</sup> A fever can be considered not related to the study vaccine if an alternative etiology can be documented.

<sup>†</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature

 Table 6:
 Vital Sign Adverse Event Grading Scale

| Physiologic Parameter | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Bradycardia - beats per minute | 50 – 54 | 45 – 49 | <45 |
| | (or $45 - 49$ if baseline $< 60$ ) | (or 40 – 44 if baseline < 60) | (or <40 if baseline < 60) |
| Tachycardia - beats per minute | 101 – 115 | 116 – 130 | >130 (or ventricular<br>dysrhythmias) |
| Hypotension (systolic) mm Hg | 85 – 89 | 80 – 84 | <80 |
| Hypotension (diastolic) mm Hg | 50 – 54 | 45 – 49 | <45 |
| Hypertension (systolic) mm Hg | 141 – 150 | 151 – 160 | >160 |
| Hypertension (diastolic) mm Hg | 91 – 95 | 96 – 100 | >100 |
| #Pulse and blood pressure assessed at s | screening will be considered as baseling | e. | |
**Table 7:** Laboratory Adverse Event Grading Scale

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| Hematology | | | |
| WBC 10 <sup>3</sup> /UL (Decrease) | 2.5 – 3.4 | 1.5 – 2.4 | <1.5 |
| WBC 10 <sup>3</sup> /UL (Increase) | 10.9–15.0 | 15.1 – 20.0 | >20.0 |
| HgB g/dL<br>Female | 10.5-11.4 | 8.5-10.4 | <8.5 |
| HgB g/dL<br>Male | 12.0-13.4 | 10.0-11.9 | <10.0 |
| HCT % decrease<br>Female | 31.5-34.2 | 25.5-31.4 | <25.5 |
| HCT % decrease<br>Male | 36.0-40.2 | 30-35.9 | <30 |
| HCT % increase | 1.01-1.1 X ULN | 1.11-1.2 X ULN | >1.2 X ULN |
| Platelets cell/10³/UL (Decrease) | 100-149 | 99-75 | <75 |
| Chemistry | | | |
| ALT | 1.25 – 3.0 x ULN | >3.0 – 5.0 x ULN | >5.0 x ULN |
| AST | 1.25 – 3.0 x ULN | >3.0 – 5.0 x ULN | > 5.0 x ULN |
| Bilirubin– when ALT ≥3 x ULN | 1.25 – 1.5 x ULN | >1.5 – 2.0 x ULN | >2.0 x ULN |
| Bilirubin | 1.25 – 2.0 x ULN | >2.0 – 2.5 x ULN | >2.5 x ULN |
| BUN mg/dL | 26-30 | 31-35 | > 35 |
| Creatinine mg/dL | 1.1 – 1.7 | 1.8 – 2.0 | >2.0 |
| Urine Dipstick | | | |
| Protein | 1+ | 2+ | >2+ |
| Glucose | 1+ | 2+ | >2+ |

**Table 8:** Probability of Observing at Least One Adverse Event Given Various True Event Rates

| Sample Size | "True"<br>Unknown Event<br>Rate | Probability of<br>Observing an<br>Event (%) | Sample Size | "True"<br>Unknown Event<br>Rate | Probability of<br>Observing an<br>Event (%) |
|---|---|---|---|---|---|
| 35 | 0.1% | 3.4 | 80 | 0.1% | 7.7 |
| | 0.5% | 16.1 | | 0.5% | 33.0 |
| | 1.0% | 29.7 | | 1.0% | 55.2 |
| | 2.0% | 50.7 | 1 | 2.0% | 80.1 |
| | 3.0% | 65.6 | 1 | 3.0% | 91.3 |
| | 4.0% | 76 | 1 | 4.0% | 96.2 |
| | 5.0% | 83.4 | 1 | 5.0% | 98.3 |
| | 10.0% | 97.5 | 1 | 10.0% | >99.9 |
| | 20.0% | >99.9 | | 20.0% | >99.9 |

**Table 9:** Minimum Detectable Event Rates given various levels of Power

| Sample Size | Desired Power<br>Level | Detectable<br>Event Rate | Sample Size | Desired Power<br>Level | Detectable<br>Event Rate |
|---|---|---|---|---|---|
| 35 | 0.80 | 4.5% | 80 | 0.80 | 2.0% |
| | 0.90 | 6.4% | | 0.90 | 2.8% |
| | 0.95 | 8.2% | | 0.95 | 3.7% |
| | 0.99 | 12.3% | | 0.99 | 5.6% |

# Table 10: Distribution of Protocol Deviations by Category, Type, and Treatment Group, All Enrolled Subjects

[Implementation note: the table will only include the deviation categories and types that occurred.]

| Category | Deviation Type | | g ZPIV<br>=X) | 5 mcg<br>(N= | ZPIV<br>=X) | Plac<br>(N= | cebo<br>=X) | | ibjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | No. of Subj. | No. of Dev. | No. of Subj. | No. of Dev. | No. of Subj. | No. of Dev. | No. of Subj. | No. of Dev. |
| Any category | Any type | X | X | X | X | X | X | X | X |
| Eligibility/ enrollment | Any type | X | X | X | X | X | X | X | X |
| | Did not meet inclusion criterion | X | X | X | X | X | X | X | X |
| | Met exclusion criterion | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | |
| | Other | | | | | | | | |
| Treatment administration | Any type | | | | | | | | |
| schedule | Out of window visit | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | |
| | Missed treatment administration | | | | | | | | |
| | Delayed treatment administration | | | | | | | | |
| | Other | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | |
| | Out of window visit | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | |
| | Other | | | | | | | | |
| Protocol procedure/ | Any type | | | | | | | | |
| assessment | Incorrect version of ICF signed | | | | | | | | |
| | Blood not collected | | | | | | | | |
| | Other specimen not collected | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | |
| | Specimen result not obtained | | | | | | | | |

Table 10: Distribution of Protocol Deviations by Category, Type, and Treatment Group, All Enrolled Subjects (continued)

| Category | Deviation Type | | g ZPIV<br>=X) | | ZPIV<br>=X) | | cebo<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | No. of Subj. | No. of Dev. | No. of Subj. | No. of Dev. | No. of Subj. | No. of Dev. | No. of Subj. | No. of Dev. |
| | Required procedure not conducted | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | |
| | Study product temperature excursion | | | | | | | | |
| | Specimen temperature excursion | | | | | | | | |
| | Other | | | | | | | | |
| Treatment administration | Any type | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | |
| | Study product temperature excursion | | | | | | | | |
| | Other | | | | | | | | |
| Blinding policy/ procedure | Any type | | | | | | | | |
| | Treatment unblinded | | | | | | | | |
| | Other | | | | | | | | |
| N=Number of subjects enrolled | 1 | | | | | | | | |

# 14.1.1 Disposition of Subjects

**Table 11:** Subject Disposition by Treatment Group

| <b>Subject Disposition</b> | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo | All Subjects |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) |
| Screened | N/A | N/A | N/A | xxx |
| Enrolled/Randomized | xx | xx | XX | XX |
| Received Vaccination 1 | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Received Vaccination 2 | | | | |
| Received All Scheduled Treatments <sup>a</sup> | | | | |
| Discontinued Dosing <sup>b</sup> | | | | |
| Terminated from Study Follow-Up <sup>b</sup> | | | | |
| Completed Follow-Up b | | | | |
| Completed Study Per Protocol b, c | | | | |

Denominators for percentages are the numbers of subjects enrolled/randomized unless otherwise specified.

<sup>&</sup>lt;sup>a</sup> Refer to Appendix 16.2.1 for reasons subjects discontinued treatment or terminated early.

<sup>&</sup>lt;sup>b</sup> Out of all randomized and vaccinated subjects.

<sup>&</sup>lt;sup>c</sup> Refer to Appendix 16.2.3 for reasons subjects were excluded from the Per Protocol population.

Table 12: Early Withdrawals and Treatment Discontinuations by Treatment Group – All Enrolled and Randomized Subjects

| 2.5 mcg ZPIV (N=X) | 5 mcg ZPIV (N=X) | Placebo (N=X) | p-value <sup>a</sup> |
|---|---|---|---|
| n (%) | n (%) | n (%) | |
| X | X | х | N/A |
| x (xx) | x (xx) | x (xx) | X.XXX |
| x (xx) | x (xx) | x (xx) | X.XXX |
| | | - | |
| | x<br>x (xx) | x X X x (xx) | x X x x x x x (xx) x (xx) |

### **Baseline ZIKV Seronegative**

**Baseline ZIKV Seropositive and DENV Seropositive** 

**Baseline ZIKV Seropositive and DENV Seronegative** 

**Baseline ZIKV Seronegative and DENV Seropositive** 

### **Baseline ZIKV Seronegative and DENV Seronegative**

N = Number of subjects enrolled

<sup>&</sup>lt;sup>a</sup> Fisher's exact 2-tailed test of the homogeneity and independence of withdrawals or discontinuations between the 3 treatment groups.

<sup>&</sup>lt;sup>b</sup>Used as denominator for percentages.

# **Table 13:** Analysis Populations by Treatment Group

[Implementation note: For visit-specific PP population exclusions, include only the reasons for which at least one subject is excluded.]

| | | | cg ZPIV<br>=X) | | g ZPIV<br>=X) | | cebo<br>=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Subjects Excluded | n | % | n | % | n | % | n | % |
| Safety Population | Did not receive at least one study vaccination | | | | | | | | |
| Immunogenicity Population | Does not have pre- and at least one post-study vaccination samples for immunogenicity testing for which valid results were reported. | | | | | | | | |
| | Loss of samples at pre-vaccination timepoints due to natural disaster <sup>a</sup> | | | | | | | | |
| | Any Time Point | | | | | | | | |
| | Any Reason | | | | | | | | |
| | Found to be ineligible at baseline | | | | | | | | |
| | Second vaccination not received <sup>b</sup> | | | | | | | | |
| | Second vaccination received out of window <sup>b</sup> | | | | | | | | |
| | Receipt of non-study licensed live vaccine within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | Receipt of non-study licensed inactivated vaccine within 14 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| Per Protocol Population | Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | The visit occurred substantially out of window | | | | | | | | |
| | Other major protocol deviation deemed exclusionary by study team | | | | | | | | |
| | Prior to or at Day 1 visit (Visit 01): | | | | | | | | |
| | Any Reason | | | | | | | | |
| | Receipt of non-study licensed live vaccine within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | Receipt of non-study licensed inactivated vaccine within 14 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |

**Table 13: Analysis Populations by Treatment Group (continued)** 

| | | | eg ZPIV<br>=X) | | g ZPIV<br>=X) | | cebo<br>=X) | All Su<br>(N= | |
|---|---|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Subjects Excluded | n | % | n | % | n | % | n | % |
| | Other major protocol deviation deemed exclusionary by study team | | | | | | | | |
| | Prior to or at Day 15 visit (Visit 05): | | | | | | | | |
| | Any Reason | | | | | | | | |
| | Receipt of non-study licensed live vaccine within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | Receipt of non-study licensed inactivated vaccine within 14 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | The visit occurred substantially out of window | | | | | | | | |
| | Other major protocol deviation deemed exclusionary by study team | | | | | | | | |
| | Prior to or at Day 29 visit (Visit 06): | | | | | | | | |
| | Any Reason | | | | | | | | |
| | Second vaccination not received <sup>b</sup> | | | | | | | | |
| | Second vaccination received out of window <sup>b</sup> | | | | | | | | |
| | Receipt of non-study licensed live vaccine within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | Receipt of non-study licensed inactivated vaccine within 14 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days prior to or after study vaccination <sup>b</sup> | | | | | | | | |
| | The visit occurred substantially out of window | | | | | | | | |
| | Other major protocol deviation deemed exclusionary by study team | | | | | | | | |
| | Repeat Day 29 for: | | | | | | | | |
| | Prior to or at Day 43 visit (Visit 10): | | | | | | | | |
| | Prior to or at Day 57 visit (Visit 11): | | | | | | | | |

Table 13: Analysis Populations by Treatment Group (continued)

| | | | g ZPIV<br>=X) | ٠ - | g ZPIV<br>=X) | | cebo<br>=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Subjects Excluded | n | % | n | % | n | % | n | % |
| | Prior to or at Day 290 visit (Visit 14): | | | | | | | | |
| | Prior to or at Day 388 visit (Visit 17): | | | | | | | | |
| | Prior to or at Day 569 visit (Visit 20): | | | | | | | | |
| | Prior to or at Day 750 visit (Visit 23): | | | | | | | | |

N=Total number of subjects enrolled.

Subjects may be excluded from an analysis population for multiple reasons.

<sup>&</sup>lt;sup>a</sup> Subjects are excluded only from immunogenicity analyses which use pre-vaccination titers, e.g., GMFR

b Subjects are excluded from per protocol analyses at all timepoints subsequent to the occurrence of this protocol deviation. All instances of exclusion are summarized in this table. Subject data collected up to the time the exclusionary criterion is met is eligible for analysis.

Table 14: Number of Subjects in Immunogenicity and Per Protocol Populations with Data Available by Analysis Type, Time Point, and Treatment Group

| Analysis<br>Population | Treatment<br>Group | Basel | ine | Da | y 15 | | 9 (Pre-<br>se 2) | Day 43<br>Post-l | (14 Days<br>Dose 2) | Day 57 (<br>Post-I | (28 Days<br>Dose 2) | Days Po | Day 209 (180<br>Days Post-Dose<br>2) | | 88 (359<br>ost-Dose<br>2) | Days Po | 69 (540<br>ost-Dose<br>2) | Days P | 50 (721<br>ost-Dose<br>2) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | " | | l | | ' | 1 | Geome | tric Mean | Titer & S | eropositiv | vity | | | | " | | • | | • |
| Immunogenicity | 2.5 mcg | | | | | | | | | | | | | | | | | | |
| | 5 mcg | | | | | | | | | | | | | | | | | | |
| | Placebo | | | | | | | | | | )<br> | | | | | | | | |
| Per Protocol | 2.5 mcg | | | | | | | | | | | | | | | | | | |
| | 5 mcg | | | | | | | | | | )<br> | | | | | | | | |
| | Placebo | | | | | | | | | | I | | | | | | | | |
| | | | 1. | | | Ge | ometric l | Mean Fold | Rise <sup>a</sup> and | Serocon | versiona | · · | | | | II. | ı | I. | |
| Immunogenicity | 2.5 mcg | | | | | | | | | | | | | | | | | | |
| | 5 mcg | | | | | | | | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | | | | | | | | |
| Per Protocol | 2.5 mcg | | | | | | | | | | | | | | | | | | |
| | 5 mcg | | | | | | | | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | | | | | | | | |

<sup>a</sup> For time points following baseline, the subject must also have baseline measurements to be counted in this table.

# **Table 15:** Date of First Treatment by Treatment Group

[Implementation Note: dates could be grouped by calendar month, bi-weekly or weekly, depending on the distribution.]

| Date of Dosing | 2.5 mcg ZPIV<br>(N=X) | 5 mcg ZPIV<br>(N=X) | Placebo<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|
| [date 1] | X | X | X | X |
| [date 2] | | | | |
| [date 3] | | | | |
| [date 4] | | | | |
| [Etc.] | | | | |

# **Table 16:** Ineligibility Summary of Screen Failures

[Implementation note: final table will only include criteria where n > 0]

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % <sup>b</sup> |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | | 100 |
| | Any inclusion criterion | | |
| | [Criterion 1] | | |
| Inclusion | [Criterion 2] | | |
| | [Criterion 3] | | |
| | [Etc.] | | |
| | Any exclusion criterion | | |
| г. 1. ' | [Criterion 1] | | |
| Exclusion | [Criterion 2] | | |
| | [Etc.] | 1 | |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup> Denominator for percentages is the total number of screen failures.

# 14.1.2 Demographic Data by Study Group

Table 17: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group

| Variable | Characteristic | | eg ZPIV<br>=X) | | g ZPIV<br>=X) | | cebo<br>=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % |
| Sex | Male | х | XX | х | xx | х | xx | х | xx |
| | Female | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | Х | xx | Х | xx | Х | XX | X | XX |
| | Hispanic or Latino | | | | | | | | |
| | Not Reported | | | | | | | | |
| | Unknown | | | | | | | | |
| Race | American Indian or Alaska Native | X | xx | X | xx | Х | XX | X | xx |
| | Asian | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | |
| | Black or African American | | | | | | | | |
| | White | | | | | | | | |
| | Multi-Racial | | | | | | | | |
| | Unknown | | | | | | | | |
| Baseline | Baseline ZIKV Seropositive | X | xx | X | xx | Х | xx | X | XX |
| Flavivirus<br>Immune Status | Baseline ZIKV Seronegative | | | | | | | | |
| | Baseline ZIKV Seropositive and DENV Seropositive | | | | | | | | |
| | Baseline ZIKV Seropositive and DENV Seronegative | | | | | | | | |
| | Baseline ZIKV Seronegative and DENV Seropositive | | | | | | | | |
| | Baseline ZIKV Seronegative and DENV Seronegative | | | | | | | | |

Table 18: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group
- Safety Population

| Variable | Statistic | 2.5 mcg ZPIV<br>(N=X) | 5 mcg ZPIV<br>(N=X) | Placebo<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | Mean | XX | | | |
| | Standard Deviation | xx.x | | | |
| Age (years) | Median | xx.x | | | |
| | Minimum | xx | | | |
| | Maximum | xx | | | |
| | Mean | xx | | | |
| | Standard Deviation | xx.x | | | |
| BMI (kg/m²) <sup>a</sup> | Median | xx.x | | | |
| | Minimum | xx | | | |
| | Maximum | XX | | | _ |

N=Number of subjects in the Safety population

<sup>&</sup>lt;sup>a</sup> at screening

### 14.1.3 Prior and Concurrent Medical Conditions

Table 19: Summary of Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| | | eg ZPIV<br>=X) | | zPIV<br>=X) | | cebo<br>=X) | | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | n | % | n | % | n | % | N<br>X | % |
| Any SOC | Х | xx | х | xx | х | xx | X | XX |
| [SOC 1] | | | | | | | | |
| [SOC 2] | | | | | | | | |
| [SOC 3] | | | | | | | | |
| [Etc.] | | | | | | | | |

# 14.2 Immunogenicity Data

### ZIKV Microneutralization Titers

Table 20: ZIKV Microneutralization Antibody (MN50) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population

[Implementation note: If a baseline flavivirus subgroup includes fewer than 2 subjects, the GMT and 95% CI fields will be populated with 'N/A'.]

| Baseline Flavivirus Immune Status | | 2.5 mcg ZPI | $\mathbf{v}$ | | 5 mcg ZPIV | 7 | | Placebo | |
|---|---|---|---|---|---|---|---|---|---|
| | n | GMT | 95% CI | n | GMT | 95% CI | n | GMT | 95% CI |
| All Subjects | х | xx | xx.x, xx.x | х | xx | xx.x, xx.x | X | XX | xx.x, xx.x |
| Baseline ZIKV Seropositive | | | | | | | | | |
| Baseline ZIKV Seronegative | | | | | | | | | |
| Baseline ZIKV Seropositive and DENV<br>Seropositive | | | | | | | | | |
| Baseline ZIKV Seropositive and DENV<br>Seronegative | | | | | | | | | |
| Baseline ZIKV Seronegative and DENV<br>Seropositive | | | | | | | | | |
| Baseline ZIKV Seronegative and DENV Seronegative | | | | | | | | | |
| | | | | | - | | | | • |
| | All Subjects Baseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive | All Subjects Baseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive | All Subjects X XX Baseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seronegative | n GMT 95% CI All Subjects x xx xx.x, xx.x Baseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seronegative and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive | All Subjects x xx xxx.xx.xx x Baseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seronegative and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive | All Subjects X XX XXX, XX.X, XX.X XX Saseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seronegative and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seronegative | n GMT 95% CI n GMT 95% CI All Subjects x xx xx.x.x.x x xx xx.x.x.x x Baseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seronegative and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seronegative | n GMT 95% CI n GMT 95% CI n All Subjects x xx xx.x, xx.x x xx xx.x, xx.x x Baseline ZIKV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seropositive Baseline ZIKV Seropositive and DENV Seronegative Baseline ZIKV Seronegative and DENV Seronegative Baseline ZIKV Seronegative and DENV Seropositive Baseline ZIKV Seronegative and DENV Seropositive | n GMT 95% CI n GMT 95% CI n GMT All Subjects |

n = Number of subjects in the immunogenicity population with non-missing immunogenicity data at the specified time point.

<sup>95%</sup> CI = 95% confidence interval based on Student's t-distribution.

- Table 21: ZIKV Microneutralization Antibody (MN50) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status Per Protocol Population
- Table 22: ZIKV Microneutralization Antibody (MN50) Geometric Mean Fold Rise (GMFR) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status Immunogenicity Population

[Implementation note: baseline results are not included in this table.]

Table 23: ZIKV Microneutralization Antibody (MN50) Geometric Mean Fold Rise (GMFR) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population

[Implementation note: baseline results are not included in this table.]

Table 24: ZIKV Microneutralization Antibody (MN50) Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population

[Implementation note: If a baseline flavivirus subgroup includes fewer than 2 subjects, the % and 95% CI fields will be populated with 'N/A'.]

| Time Point | Outcome | Baseline Flavivirus Immune<br>Status | | 2.5 mc | g ZPIV | | | 5 mc | eg ZPIV | | | Pla | cebo | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | N* | n | % | 95% CI | N* | n | % | 95% CI | N* | n | % | 95% CI |
| Baseline | Titer ≥10 | All Subjects | | | | | | | | | | | | |
| | | Baseline ZIKV Seropositive | | | | | | | | | | | | |
| | | Baseline ZIKV Seronegative | | | | | | | | | | | | |
| | | Baseline ZIKV Seropositive and DENV Seropositive | | | | | | | | | | | | |
| | | Baseline ZIKV Seropositive and DENV Seronegative | | | | | | | | | | | | |
| | | Baseline ZIKV Seronegative and DENV Seropositive | | | | | | | | | | | | |
| | | Baseline ZIKV Seronegative and DENV Seronegative | | | | | | | | | | | | |
| | Titer | All Subjects | | | | | | | | | | | | |
| | ≥100 | Baseline ZIKV Seropositive | | | | | | | | | | | | |
| | | Baseline ZIKV Seronegative | | | | | | | | | | | | |
| | | Baseline ZIKV Seropositive and DENV Seropositive | | | | | | | | | | | | |
| | | Baseline ZIKV Seropositive and DENV Seronegative | | | | | | | | | | | | |
| | | Baseline ZIKV Seronegative and DENV Seropositive | | | | | | | | | | | | |
| | | Baseline ZIKV Seronegative and DENV Seronegative | | | | | | | | | | | | |
| Repeat Baselin | e for: | <u> </u> | | • | | • | | • | • | - | • | | | |
| Day 29 (Pre-<br>Dose 2) | | | | | | | | | | | | | | |

Table 24: ZIKV Microneutralization Antibody (MN50) Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status -- Immunogenicity Population (continued)

| Day 57 (28<br>Days Post-<br>Dose 2) |
|---------------------------------------|
| Day 209 (180<br>Days Post-<br>Dose 2) |
| Day 750 (721<br>Days Post-<br>Dose 2) |
| Peak Post-<br>Baseline |

 $N^* =$  Number of subjects with results available at the specified time point

Table with similar format:

Table 25: ZIKV Microneutralization Antibody (MN50) Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population

n = number of subjects seropositive at the specified time point

<sup>95%</sup> CI = Exact 95% Clopper-Pearson confidence interval.

Table 26: ZIKV Microneutralization Antibody (MN50) Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population

[Implementation note: If a baseline flavivirus subgroup includes fewer than 2 subjects, the % and 95% CI fields will be populated with 'N/A'.]

| L 1 | | | 8 | 1 | | J | , | | | 1 1 | | J | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Baseline Flavivirus<br>Immune Status | | 2.5 mc | g ZPIV | | | 5 mcg | ZPIV | | | Plac | cebo | |
| | | N* | n | % | 95% CI | N* | n | % | 95% CI | N* | n | % | 95% CI |
| | All Subjects | | | | | | | | | | | | |
| | Baseline ZIKV<br>Seropositive | | | | | | | | | | | | |
| | Baseline ZIKV<br>Seronegative | | | | | | | | | | | | |
| Day 29 | Baseline ZIKV<br>Seropositive and<br>DENV Seropositive | | | | | | | | | | | | |
| (Pre-Dose 2) | Baseline ZIKV<br>Seropositive and<br>DENV Seronegative | | | | | | | | | | | | |
| | Baseline ZIKV<br>Seronegative and<br>DENV Seropositive | | | | | | | | | | | | |
| | Baseline ZIKV<br>Seronegative and<br>DENV Seronegative | | | | | | | | | | | | |
| Repeat Day 29 for: | | | | | | | | | | | | | |
| Day 57 (28 Days<br>Post-Dose 2) | | | | | | | | | | | | | |
| Day 209 (180<br>Days Post-Dose<br>2) | | | | | | | | | | | | | |
| Day 750 (721<br>Days Post-Dose<br>2) | | | | | | | | | | | | | |
| Peak Post-<br>Baseline | | | | | | | | | | | | | |

# Table 26: ZIKV Microneutralization Antibody (MN50) Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status -- Immunogenicity Population (continued)

Seroconversion is defined as at least a 4-fold rise in ZIKV MN50 titers from baseline.

N\* = Number of subjects with results available at baseline and the specified time point

n = number of subjects seroconverting at the specified time point

95% CI = 95% confidence interval.

### Table with similar format:

Table 27: ZIKV Microneutralization Antibody (MN50) Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population

### **ZIKV ELISA Titers**

Tables with format similar to Table 20:

- Table 28: ZIKV ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status Immunogenicity Population
- Table 29: ZIKV ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status Per Protocol Population
- Table 30: ZIKV ELISA Geometric Mean Fold Rise (GMFR) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status Immunogenicity Population

[Implementation Note: Baseline results are not included in this table.]

Table 31: ZIKV ELISA Geometric Mean Fold Rise (GMFR) Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population

[Implementation Note: Baseline results are not included in this table.]

Tables with format similar to Table 24:

Table 32: ZIKV ELISA Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Immunogenicity Population

[Implementation note: seropositivity is defined as titers  $\geq 200$  and  $\geq 600$ .]

Table 33: ZIKV ELISA Seropositivity Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Per Protocol Population

[Implementation note: seropositivity is defined as titers  $\geq 200$  and  $\geq 600$ .]

Tables with format similar to Table 26:

- Table 34: ZIKV ELISA Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status Immunogenicity Population
- Table 35: ZIKV ELISA Seroconversion Results with 95% Confidence Intervals by Time Point, Treatment Group, and Baseline Flavivirus Immune Status Per Protocol Population

# 14.3 Safety Data

# 14.3.1 Displays of Adverse Events

# **Table 36:** Overall Summary of Adverse Events – All Subjects

| | | | eg ZPIV<br>(=X) | | g ZPIV<br>=X) | | cebo<br>=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| Event Category <sup>a</sup> | Subcategory | n (%) | 95% CI | n (%) | 95% CI | n (%) | 95% CI | n (%) | 95% CI |
| At least one local solicited adverse event b | | xx (xx) | xx.x, xx.x | xx (xx) | xx.x, xx.x | xx (xx) | xx.x, xx.x | xx (xx) | xx.x, xx.x |
| At least one systemic solicited adverse event <sup>b</sup> | | | | | | | | | |
| At least one unsolicited adverse event c | | | | | | | | | |
| | Any Severity | | | | | | | | |
| At least one related unsolicited adverse event c | Mild (Grade 1) | | | | | | | | |
| At least one related unsonched adverse event | Moderate (Grade 2) | | | | | | | | |
| | Severe (Grade 3) | | | | | | | | |
| | Any Severity | | | | | | | | |
| At least one related laboratory adverse event <sup>c</sup> | Mild (Grade 1) | | | | | | | | |
| At least one related laboratory adverse event | Moderate (Grade 2) | | | | | | | | |
| | Severe (Grade 3) | | | | | | | | |
| | Any Severity | | | | | | | | |
| | Mild (Grade 1) | | | | | | | | |
| At least one related unsolicited or laboratory adverse event <sup>c</sup> | Moderate (Grade 2) | | | | | | | | |
| | Severe (Grade 3) | | | | | | | | |
| | Any Relationship | | | | | | | | |
| At least one severe (Grade 3) unsolicited adverse event <sup>c</sup> | Related | | | | | | | | |
| | Unrelated | | | | | | | | |
| At least one serious adverse event <sup>d</sup> | | | | | | | | | |
| At least one related serious adverse event d | | | | | | | | | |
| At least one adverse event leading to early termination from the study <sup>d</sup> | | | | | | | | | |

# Table 36: Overall Summary of Adverse Events -- All Subjects (continued)

| | | | eg ZPIV<br>=X) | ٠ | g ZPIV<br>=X) | | cebo<br>=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| Event Category <sup>a</sup> | Subcategory | n (%) | 95% CI | n (%) | 95% CI | n (%) | 95% CI | n (%) | 95% CI |
| At least one adverse event leading to discontinuation of study product | | | | | | | | | |
| At least one adverse event of special interest (AESI) d | | | | | | | | | |
| At least one related AESI d | | | | | | | | | |
| At least one new onset chronic medical condition (NOCMC) d | | | | | | | | | |
| At least one related NOCMC d | | | | | | | | | |

N = Number of subjects in the safety population. CI = Exact (Clopper-Pearson) confidence interval.

n = Number of subjects experiencing the event.

<sup>&</sup>lt;sup>a</sup> Subjects are counted once for each category regardless of the number of events. <sup>b</sup> Solicited AEs are collected through Day 8 post each dose.

Non-serious unsolicited AEs within 28 days of either dose.

d At any time during the study.

Tables with similar format:

## Table 37: Overall Summary of Adverse Events – Baseline ZIKV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with specified baseline flavivirus immune status]

### **Table 38:** Overall Summary of Adverse Events – Baseline ZIKV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population with specified baseline flavivirus immune status]

## Table 39: Overall Summary of Adverse Events – Baseline ZIKV Seropositive and DENV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with specified baseline flavivirus immune status]

### Table 40: Overall Summary of Adverse Events – Baseline ZIKV Seropositive and DENV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population with specified baseline flavivirus immune status]

### Table 41: Overall Summary of Adverse Events – Baseline ZIKV Seronegative and DENV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with specified baseline flavivirus immune status]

### Table 42: Overall Summary of Adverse Events – Baseline ZIKV Seronegative and DENV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population with specified baseline flavivirus immune status]

## 14.3.1.1 Solicited Adverse Events

Table 43: Comparison of the Frequency, Type and Duration of Vaccine-Related Grade 3 Local, Systemic or Laboratory AEs and Grade 2 or Greater Local or Systemic Reactogenicity Through Day 8 Post Vaccination

| | | | 2.5 | mcg ZPIV | 5 m | cg ZPIV | Pla | icebo | p-va | lue |
|---|---|---|---|---|---|---|---|---|---|---|
| Post Dose Number | AE Type | Symptom/Lab<br>AE | n | Median<br>Duration<br>(Days) | n | Median<br>Duration<br>(Days) | n | Median<br>Duration<br>(Days) | <sup>a</sup> Frequency | <b>b</b> Duration |
| All Subjects | | | | | | | | | | |
| Post Dose 1 | Number of Subjects in the Safety<br>Received the Specified Dose | y Population Who | X | N/A | х | N/A | X | N/A | N/A | N/A |
| | Vaccine related Grade 3 local, | [Event 1] | x | X.X | х | x.x | x | x.x | X.XXX | x.xxx |
| | systemic or laboratory AE | [Event 2] | | | | | | | X.XXX | x.xxx |
| | | [Event 3] | | | | | | | X.XXX | x.xxx |
| | | Etc. | | | | | | | X.XXX | x.xxx |
| | *Grade 2 or greater local or | [Event 1] | | | | | | | x.xxx | x.xxx |
| | systemic reactogenicity | [Event 2] | | | | | | | X.XXX | x.xxx |
| | | [Event 3] | | | | | | | X.XXX | x.xxx |
| | | Etc. | | | | | | | X.XXX | x.xxx |
| Repeat Post Dose 1 for: | | | | | | | | | | |
| Baseline ZIKV Seropositive | | | | | | | | | | |
| Baseline ZIKV Seronegative | | | | | | | | | | |
| Baseline ZIKV Seropositive an | d DENV Seropositive | | | | | | | | | |
| Baseline ZIKV Seropositive an | d DENV Seronegative | | | | | | | | | |
| Baseline ZIKV Seronegative ar | nd DENV Seropositive | | | | | | | | | |
| Baseline ZIKV Seronegative ar | nd DENV Seronegative | | | | | | | | | |
| All Subjects | | | | | | | | | | |
| Post Dose 2 | Number of Subjects in the Safety<br>Received the Specified Dose | y Population Who | Х | N/A | х | N/A | X | N/A | N/A | N/A |
| | | [Event 1] | X | x.x | X | X.X | x | X.X | X.XXX | x.xxx |

Table 43: Comparison of the Frequency, Type and Duration of Vaccine-Related Grade 3 Local, Systemic or Laboratory AEs and Grade 2 or Greater Local or Systemic Reactogenicity Through Day 8 Post Vaccination (continued)

| | Vaccine related Grade 3 local, | [Event 2] | | | | | | | X.XXX | x.xxx |
|---|---|---|---|---|---|---|---|---|---|---|
| | systemic or laboratory AE | [Event 3] | | | | | | | X.XXX | x.xxx |
| | | Etc. | | | | | | | x.xxx | x.xxx |
| | *Grade 2 or greater local or | [Event 1] | | | | | | | X.XXX | x.xxx |
| | systemic reactogenicity | [Event 2] | | | | | | | X.XXX | x.xxx |
| | | [Event 3] | | | | | | | X.XXX | x.xxx |
| | | Etc. | | | | | | | X.XXX | x.xxx |
| Repeat Post Dose 2 for: | | | | | | | | | | |
| Baseline ZIKV Seropositive | | | | | | | | | | |
| Baseline ZIKV Seronegative | ; | | | | | | | | | |
| Baseline ZIKV Seropositive | and DENV Seropositive | | | | | | | | | |
| Baseline ZIKV Seropositive | and DENV Seronegative | | | | | | | | | |
| Baseline ZIKV Seronegative | and DENV Seropositive | | | | | | | | | |
| Baseline ZIKV Seronegative | and DENV Seronegative | | | | | | | | | |
| All Subjects | | | | | | | | | | |
| Post Any Dose | Number of Subjects in the | ne Safety Population | X | N/A | X | N/A | X | N/A | N/A | N/A |
| | Vaccine related Grade 3 local, | [Event 1] | X | X.X | х | X.X | x | x.x | X.XXX | x.xxx |
| | systemic or laboratory AE | [Event 2] | | | | | | | X.XXX | x.xxx |
| | | [Event 3] | | | | | | | X.XXX | x.xxx |
| | | Etc. | | | | | | | X.XXX | x.xxx |
| | *Grade 2 or greater local or | [Event 1] | | | | | | | X.XXX | x.xxx |
| | systemic reactogenicity | [Event 2] | | | | | | | X.XXX | x.xxx |
| | 1 | | | | | | | | X.XXX | V VVV |
| | | [Event 3] | | | | | | | Λ.ΛΛΛ | X.XXX |

# Table 43: Comparison of the Frequency, Type and Duration of Vaccine-Related Grade 3 Local, Systemic or Laboratory AEs and Grade 2 or Greater Local or Systemic Reactogenicity Through Day 8 Post Vaccination (continued)

Baseline ZIKV Seropositive

Baseline ZIKV Seronegative

Baseline ZIKV Seropositive and DENV Seropositive

Baseline ZIKV Seropositive and DENV Seronegative

Baseline ZIKV Seronegative and DENV Seropositive

Baseline ZIKV Seronegative and DENV Seronegative

n = Number of subjects

Only the frequency, not the duration of laboratory AEs will be compared.

<sup>\*</sup> Through Day 8 post vaccination

<sup>&</sup>lt;sup>a</sup> Frequencies of adverse events compared between ZPIV dosage groups using Fisher's Exact test.

<sup>&</sup>lt;sup>b</sup> Distribution of the duration of adverse events compared between ZPIV dosage groups using Wilcoxon 2-sample test.

Table 44: Number and Percentage of Subjects Experiencing Any Local or Systemic Solicited Events through Day 8 Post Vaccination by Dose, Baseline Flavivirus Immune Status, Severity and Treatment Group

| | | | g ZPIV | | g ZPIV | | cebo | All Su | |
|---|---|---|---|---|---|---|---|---|---|
| Baseline Flavivirus Immune | | (N=X) (N=X) | | (N=X) | | (N=X) | | | |
| Status | Severity | n | % | n | % | n | % | n | % |
| Post Dose 1 | | | T | T. | | T. | | | |
| | Number of Subjects | X | N/A | X | N/A | X | N/A | X | N/A |
| | None | XX | Xx | XX | XX | XX | XX | XX | XX |
| All Subjects | Mild | | | | | | | | |
| All Subjects | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Not Reported | | | | | | | | |
| | Number of Subjects | | | | | | | | |
| | None | | | | | | | | |
| D 1' THEN C '.' | Mild | | | | | | | | |
| Baseline ZIKV Seropositive | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Not Reported | | | | | | | | |
| | Number of Subjects | | | | | | | | |
| | None | | | | | | | | |
| D1: 7IVV C | Mild | | | | | | | | |
| Baseline ZIKV Seronegative | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Not Reported | | | | | | | | |
| | Number of Subjects | | | | | | | | |
| Baseline ZIKV Seropositive | None | | | | | | | | |
| and DENV Seropositive | Mild | | | | | | | | |
| | Moderate | | | | | | | | |

Table 44: Number and Percentage of Subjects Experiencing Any Local or Systemic Solicited Events through Day 8 Post Vaccination by Dose, Baseline Flavivirus Immune Status, Severity and Treatment Group (continued)

| | Severe |
|---|---|
| | Not Reported |
| | Number of Subjects |
| | None |
| Baseline DENV Seropositive | Mild |
| and DENV Seronegative | Moderate |
| | Severe |
| | Not Reported |
| Baseline DENV Seronegative | Number of Subjects |
| | None |
| | Mild |
| and DENV Seropositive | Moderate |
| | Severe |
| | Not Reported |
| Baseline DENV Seronegative and DENV Seronegative | Number of Subjects |
| | None |
| | Mild |
| | Moderate |
| | Severe |
| | Not Reported |
| Dancet for: | |

### Repeat for:

### Post Dose 2

### **Post Any Dose**

In this table, subjects who reported not having a symptom are listed as "None", while subjects who did not complete their Memory Aid or could not remember whether they had a symptom are listed as "Not Reported".

Severity is the maximum severity reported post dosing for each subject.

N=Number of subjects in the Safety population who received the specified dose.

# Table 44: Number and Percentage of Subjects Experiencing Any Local or Systemic Solicited Events through Day 8 Post Vaccination by Dose, Baseline Flavivirus Immune Status, Severity and Treatment Group (continued)

n = Number of subjects reporting an event

For subjects in Group 3 receiving vaccinations in both arms, the maximum severity in either arm is summarized

Table 45: Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – All Subjects

| Symptom | | 2.5 mcg ZPIV<br>(N=X) | 5 mcg ZPIV<br>(N=X) | Placebo<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| Post Dose 1 | | | | | |
| Any Local Reaction | n (%) | x (xx) | x (xx) | x (xx) | x (xx) |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Repeat for: | | | | | |
| Pain | | | | | |
| Erythema | | | | | |
| Induration (mm) | | | | | |
| Induration | | | | | |
| Pruritis | | | | | |
| Ecchymosis | | | | | |
| Tenderness | | | | | |
| Any Systemic Reaction | n (%) | x (xx) | x (xx) | x (xx) | x (xx) |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| Repeat for: | | | | | |
| Feverishness | | | | | |
| Fatigue | | | | | |
| Malaise | | | | | |
| Myalgia | | | | | |
| Arthralgia | | | | | |
| Headache | | | | | |
| Nausea | | | | | |
| Vomiting | | | | | |
| Diarrhea | | | | | |
| Abdominal Pain | | | | | |
| Rash | | | | | |
| Fever | | | | | |

Repeat for:

Post Dose 2

Post Any Dose

Each event is defined as any grade 1, 2 or 3 solicited reaction within 7 days following either dose.

N = Number of subjects in the safety population who received the specified dose; used as the denominator for percentages.

n = Number of subjects reporting an event

Tables with similar format:

Table 46: Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 47: Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 48: Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 49: Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 50: Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 51: Number, Percentage and 95% Confidence Interval of Subjects Experiencing Any Grade 1 or Greater Solicited Adverse Event, by Dose, Symptom and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

**Table 52:** Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity and Treatment Group - All Subjects

| | | | tions, Post Dos<br>Subjects | se 1 | | | |
|---|---|---|---|---|---|---|---|
| | | 2.5 mcg ZPIV<br>(N=X) | | 5 mcg ZPIV<br>(N=X) | | Placebo<br>(N=X) | |
| Reaction | Severity | n | % | n | % | n | % |
| | None | X | xx | X | XX | X | XX |
| | Mild | | | | | | |
| Any Local Reaction | Moderate | | | | | | |
| | Severe | | | | | | |
| | Not Reported | | | | | | |
| Repeat for: | | | | | | | |
| Pain | | | | | | | |
| Erythema | | | | | | | |
| Induration (mm) | | | | | | | |
| Induration | | | | | | | |
| Pruritis | | | | | | | |
| Ecchymosis | | | | | | | |
| Tenderness | | | | | | | |
| Repeat for: | | | | | | | |
| | | | tions, Post Dos<br>Subjects | se 2 | | | |
| | | | ons, Post Any | Dose | | | |
| | | | Subjects | | | | |

All Subjects

Subjects who reported not having a symptom are listed as "None", while subjects who did not complete their Memory Aid or could not remember whether they had a symptom are listed as "Not Reported".

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

N=Number of subjects in the Safety Population who received the specified dose.

n = Number of subjects reporting an event

For subjects receiving vaccinations in both arms, the maximum severity in either arm is summarized

Tables with similar format:

Table 53: Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 54: Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 55: Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 56: Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 57: Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.]

Table 58: Number and Percentage of Subjects Experiencing Solicited Local Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population with the specified flavivirus immune status at baseline.
Table 59: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – All Subjects

| | | 2.5 mc<br>(N | g ZPIV<br>=X) | | g ZPIV<br>=X) | | cebo<br>=X) |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % |
| | None | X | xx | X | XX | X | XX |
| | Mild | | | | | | |
| Any Systemic Symptom | Moderate | | | | | | |
| | Severe | | | | | | |
| | Not Reported | | | | | | |
| Repeat for: | | | 1 | | | | • |
| Feverishness | | | | | | | |
| Fatigue | | | | | | | |
| Malaise | | | | | | | |
| Myalgia | | | | | | | |
| Arthralgia | | | | | | | |
| Headache | | | | | | | |
| Nausea | | | | | | | |
| Vomiting | | | | | | | |
| Diarrhea | | | | | | | |
| Abdominal Pain | | | | | | | |
| Rash | | | | | | | |
| Fever | | | | | | | |
| Repeat for: | | | | | | | |
| Repeat for: | | | | | | | |

Subjects who reported not having a symptom are listed as "None", while subjects who did not complete their Memory Aid or could not remember whether they had a symptom are listed as "Not Reported".

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

N=Number of subjects in the Safety Population who received the specified dose.

n = Number of subjects reporting an event

For subjects receiving vaccinations in both arms, the maximum severity in either arm is summarized.

Tables with similar format:

Table 60: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population that were flavivirus seropositive at baseline.]

Table 61: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population that were flavivirus seronegative at baseline.]

Table 62: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population that were flavivirus seropositive at baseline.]

Table 63: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population that were flavivirus seropositive at baseline.]

Table 64: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects

[Implementation note: N = Number of subjects in the Safety population that were flavivirus seropositive at baseline.]

Table 65: Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose, Reaction, Severity, and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects

[Implementation note: N = Number of subjects in the Safety population that were flavivirus seropositive at baseline.]

Table 66: Number and Percentage of Subjects Experiencing Solicited Local or Systemic Events by Symptom, Severity, and Day Post Dosing – 2.5 mcg ZPIV – Post Dose 1

| | | | | 5 21 1 | | | | | 2.5 n | ncg ZP | IV, All | subject | S | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | ber = 1 | | | | | | | | | | | |
| Severity | Pre- | Dose | | mins<br>-Dose | Da | y 1 | Da | y 2 | Da | ıy 3 | Da | ny 4 | Da | ny 5 | Da | y 6 | Da | ny 7 | Day | <b>8</b> + | Any<br>Do | Post- |
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Reaction | | | | | | | | | | | | | | | | | | | | | | |
| None | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mild | | | | | | | | | | | | | | | | | | | | | | |
| Moderate | | | | | | | | | | | | | | | | | | | | | | |
| Severe | | | | | | | | | | | | | | | | | | | | | | |
| Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Repeat for: | | | | | | | | | | | | | | | | | | | | | | |
| Solicited Local | Events | | | | | | | | | | | | | | | | | | | | | |
| Any Local Read | ction | | | | | | | | | | | | | | | | | | | | | |
| Pain | | | | | | | | | | | | | | | | | | | | | | |
| Erythema | | | | | | | | | | | | | | | | | | | | | | |
| Induration (mn | 1) | | | | | | | | | | | | | | | | | | | | | |
| Induration | | | | | | | | | | | | | | | | | | | | | | |
| Pruritis | | | | | | | | | | | | | | | | | | | | | | |
| Ecchymosis | | | | | | | | | | | | | | | | | | | | | | |
| Tenderness | | | | | | | | | | | | | | | | | | | | | | |
| Solicited System | nic Even | its | | | | | | | | | | | | | | | | | | | | |
| Any Systemic F | Reaction | | | | | | | | | | | | | | | | | | | | | |
| Feverishness | | | | | | | | | | | | | | | | | | | | _ | | |
| Fatigue | | | | | | | | | | | | | | | | | | | | | | |
| Malaise | | | | | | | | | | | | | | | | | | | | | | |

Table 66: Number and Percentage of Subjects Experiencing Solicited Local or Systemic Events by Symptom, Severity, and Day Post Dosing – 2.5 mcg ZPIV – Post Dose 1

| | | | | | | | | | Dos | e Num | oer = 1 | (N=X) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Severity | Pre- | Dose | | nins<br>-Dose | Da | y 1 | Da | y 2 | Da | ny 3 | Da | y 4 | Da | y 5 | Da | y 6 | Da | ny 7 | Day | 8+ | | Post-<br>se* |
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Myalgia | | | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | | | | | | | | | | | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | | | | | | | | | | | |
| Nausea Vomiting Diarrhea | | | | | | | | | | | | | | | | | | | | | | |

# Rash Fever

In this table, subjects who reported not having a symptom are listed as "None".

Subjects who were not seen for assessment nor completed a memory aid, or subjects who could not remember whether they had a symptom are listed as "Not Reported".

N = Number of subjects in the Safety population and dosage group who received the specified dose.

n = Number of subjects reporting an event

Severity is the maximum severity reported post dosing for each subject for each day.

\* Maximum severity post dosing for each subject over all days.

Tables with similar format:

## 2.5 mcg ZPIV

Table 67: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 2.5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population and dosage group who received the specified dose.]

Table 68: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 2.5 mcg ZPIV – Post Any Dose

[Implementation note: N = Number of subjects in the Safety population and dosage group]

## 5 mcg ZPIV

Table 69: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety Population and dosage group.]

Table 70: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety Population and dosage group who received the specified dose.]

Table 71: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – 5 mcg ZPIV – Post Any Dose

[Implementation note: N = Number of subjects in the Safety Population and dosage group.]

## Placebo

Table 72: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Placebo – Post Dose 1

[Implementation note: N = Number of subjects in the Safety Population and dosage group.]

Table 73: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Placebo – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population and dosage group who received the specified dose.]

Table 74: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Placebo – Post Any Dose

[Implementation note: N = Number of subjects in the Safety Population and dosage group.]

## 2.5 mcg ZPIV

Table 75: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 76: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 77: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 2.5 mcg ZPIV – Post Any Dose

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status.]

## 5 mcg ZPIV

Table 78: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group and baseline flavivirus immune status who received the specified dose.]

Table 79: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 80: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – 5 mcg ZPIV – Post Any Dose

## Placebo

Table 81: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – Placebo – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 82: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – Placebo – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 83: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive Subjects – Placebo – Post Any Dose

## 2.5 mcg ZPIV

Table 84: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety Population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 85: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety Population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 86: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom,
Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 2.5 mcg ZPIV –
Post Any Dose

[Implementation note: N = Number of subjects in the Safety Population, dosage group, and baseline flavivirus immune status.]

## 5 mcg ZPIV

Table 87: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety Population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 88: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety Population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 89: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – 5 mcg ZPIV – Post Any Dose

## Placebo

Table 90: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – Placebo – Post Dose 1

[Implementation note: N = Number of subjects in the Safety Population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 91: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – Placebo – Post Dose 2

[Implementation note: N = Number of subjects in the Safety Population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 92: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative Subjects – Placebo – Post Any Dose

## 2.5 mcg ZPIV

Table 93: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 94: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 95: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Any Dose

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status.]

## 5 mcg ZPIV

Table 96: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group and baseline flavivirus immune status who received the specified dose.]

Table 97: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 98: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – 5 mcg ZPIV – Post Any Dose

## Placebo

Table 99: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Placebo – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 100: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Placebo – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 101: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Placebo – Post Any Dose

## 2.5 mcg ZPIV

Table 102: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 103: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 104: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Any Dose

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status.]

## 5 mcg ZPIV

Table 105: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group and baseline flavivirus immune status who received the specified dose.]

Table 106: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 107: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – 5 mcg ZPIV – Post Any Dose

## Placebo

Table 108: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – Placebo – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 109: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – Placebo – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 110: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seropositive DENV Seronegative Subjects – Placebo – Post Any Dose

## 2.5 mcg ZPIV

Table 111: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 112: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 113: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 2.5 mcg ZPIV – Post Any Dose

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status.]

## 5 mcg ZPIV

Table 114: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group and baseline flavivirus immune status who received the specified dose.]

Table 115: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 116: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – 5 mcg ZPIV – Post Any Dose

## Placebo

Table 117: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – Placebo – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 118: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – Placebo – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 119: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seropositive Subjects – Placebo – Post Any Dose

## 2.5 mcg ZPIV

Table 120: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 121: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 122: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 2.5 mcg ZPIV – Post Any Dose

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status.]

## 5 mcg ZPIV

Table 123: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 5 mcg ZPIV – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group and baseline flavivirus immune status who received the specified dose.]

Table 124: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 5 mcg ZPIV – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 125: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – 5 mcg ZPIV – Post Any Dose

## Placebo

Table 126: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – Placebo – Post Dose 1

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 127: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – Placebo – Post Dose 2

[Implementation note: N = Number of subjects in the Safety population, dosage group, and baseline flavivirus immune status who received the specified dose.]

Table 128: Number and Percentage of Subjects Experiencing Solicited Local Events by Symptom, Severity, and Day Post Dosing – Baseline ZIKV Seronegative DENV Seronegative Subjects – Placebo – Post Any Dose

## 14.3.1.2 Unsolicited Adverse Events

Table 129: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship to Study Treatment, and Baseline Flavivirus Immune Status – 2.5 mcg ZPIV

| | | | | | | | ibjects<br>=X) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Any | | | | | | Severit | y | | | | | Relati | ionship | to Trea | tment | |
| MedDRA System Organ | | ] | Inciden | ee | | Mild | | 1 | Modera | te | | Severe | | N | ot Relat | ted | | Related | 1 |
| Class | MedDRA Preferred Term | n | % | m | n | % | m | n | % | m | n | % | m | n | % | m | n | % | m |
| Any SOC | Any PT | х | XX | X | х | XX | Х | X | XX | Х | X | XX | х | X | XX | X | X | XX | X |
| [SOC 1] | Any PT | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | |

#### Repeat For:

Baseline ZIKV Seropositive

Baseline ZIKV Seronegative

Baseline ZIKV Seropositive and DENV Seropositive

Baseline ZIKV Seropositive and DENV Seronegative

Baseline ZIKV Seronegative and DENV Seropositive

Baseline ZIKV Seronegative and DENV Seronegative

 $N^* = Number of subjects in the Safety population with the specified baseline flavivirus immune status. used as denominator for percentages; n=Number of subjects reporting the event; m= Number of events.$ 

Table includes all events reported per subject from first administration of study vaccine through 28 days after the last vaccination.

## Tables with similar format:

- Table 130: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship to Study Treatment, and Baseline Flavivirus Immune Status 5 mcg ZPIV
- Table 131: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship to Study Treatment, and Baseline Flavivirus Immune Status Placebo

Table 132: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class, Preferred Term, Severity, Dose, and Baseline Flavivirus Immune Status – 2.5 mcg ZPIV

| Baseline<br>Flavivirus | MedDRA<br>System | Preferred<br>Term | Severity | | | Dose 1 = X) | | | | Dose 2<br>= X) | | | Post-A<br>(N | ny Dose<br>= X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Immune Status | Organ<br>Class | | | n | % | 95%<br>CI | m | n | % | 95%<br>CI | m | n | % | 95%<br>CI | m |
| All Subjects<br>(N*=X) | Any SOC | Any PT | Any<br>Severity | xx | xx | xx.x,<br>xx.x | xx | xx | xx | XX.X,<br>XX.X | xx | xx | xx | XX.X,<br>XX.X | xx |
| | | | Mild | | | | | | | | | | | | |
| | | | Moderate | | | | | | | | | | | | |
| | | | Severe | | | | | | | | | | | | |
| | [SOC 1] | Any PT | Any<br>Severity | | | | | | | | | | | | |
| | | | Mild | | | | | | | | | | | | |
| | | | Moderate | | | | | | | | | | | | |
| | | | Severe | | | | | | | | | | | | |
| | | [PT 1] | Any<br>Severity | | | | | | | | | | | | |
| | | | Mild | | | | | | | | | | | | |
| | | | Moderate | | | | | | | | | | | | |
| | | | Severe | | | | | | | | | | | | |
| Repeat for: | | | | 1 | T | T | | 1 | 1 | 1 | | 1 | | 1 | 1 |
| Baseline ZIKV<br>Seropositive<br>(N* = X) | | | | | | | | | | | | | | | |
| Baseline ZIKV<br>Seronegative<br>(N* = X) | | | | | | | | | | | | | | | |
| Baseline ZIKV<br>Seropositive and<br>DENV<br>Seropositive | | | | | | | | | | | | | | | |

Table 132: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class, Preferred Term, Severity, Dose, and Baseline Flavivirus Immune Status – 2.5 mcg ZPIV (continued)

| Baseline<br>Flavivirus | MedDRA<br>System | Preferred<br>Term | Severity | | | Dose 1<br>= X) | | | Post-I<br>(N = | Oose 2 = X) | | | Post-A | ny Dose<br>= X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Immune Status | Organ<br>Class | | | n | % | 95%<br>CI | m | n | % | 95%<br>CI | m | n | % | 95%<br>CI | m |
| $(\mathbf{N}^* = \mathbf{X})$ | | | | | | | | | | | | | | | |
| Baseline ZIKV Seropositive and DENV Seronegative (N* = X) | | | | | | | | | | | | | | | |
| Baseline ZIKV Seronegative and DENV Seropositive (N* = X) | | | | | | | | | | | | | | | |
| Baseline ZIKV<br>Seronegative and<br>DENV<br>Seronegative<br>(N* = X) | | | | | | | | | | | | | | | |

N = Number of subjects in the Safety Population who received the specified dose; N\* = Number of subjects in the Safety population with the specified baseline flavivirus immune status. used as denominator for percentages; n=Number of subjects reporting an event under the SOC and PT combination; m = Number of events under the SOC and PT combination.

Post dose columns include events reported within 28 days following the dose; Post-Any Dose column includes events reported within 28 days following either dose. 95% CI = 95% exact Clopper-Pearson confidence interval

## Tables with similar format:

- Table 133: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class, Preferred Term, Severity, Dose, and Baseline Flavivirus Immune Status 5 mcg ZPIV
- Table 134: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class, Preferred Term, Severity, Dose, and Baseline Flavivirus Immune Status Placebo

Table 135: Number and Percentage of Subjects Reporting NOCMCs by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status

| | | | | 2.5 mc;<br>(N= | g ZPIV<br>=X) | | | 5 mcg<br>(N= | ZPIV<br>=X) | | | | cebo<br>=X) | | | | bjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baseline<br>Flavivirus<br>Immune<br>Status | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term | n | % | 95 %<br>CI | m | n | % | 95 %<br>CI | m | n | % | 95 %<br>CI | m | n | % | 95 %<br>CI | m |
| | Any SOC | Any PT | x | XX | xx.x,<br>xx.x | Х | X | XX | XX.X,<br>XX.X | X | X | XX | XX.X,<br>XX.X | х | X | xx | XX.X,<br>XX.X | х |
| | [SOC 1] | Any PT | | | | | | | | | | | | | | | | |
| All Subjects | | [PT 1] | | | | | | | | | | | | | | | | |
| $(\mathbf{N}^* = \mathbf{X})$ | | [PT 2] | | | | | | | | | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | | | | | |

Repeat for:

**Baseline ZIKV Seropositive** 

 $(N^* = X)$ 

**Baseline ZIKV Seronegative** 

 $(N^* = X)$ 

Baseline ZIKV Seropositive and DENV Seropositive

 $(\mathbf{N}^* = \mathbf{X})$ 

Baseline ZIKV Seropositive and DENV Seronegative

 $(\mathbf{N}^* = \mathbf{X})$ 

**Baseline ZIKV Seronegative and DENV Seropositive** 

(N\* = X)

Baseline ZIKV Seronegative and DENV Seronegative

(N\* = X

N = Number of subjects in the Safety population; N\* = Number of subjects in the Safety population with the specified baseline flavivirus immune status used as the denominator for percentages; n = Number of subjects reporting an event under the SOC and PT combination; m = Number of events under the SOC and PT combination.

Table includes events reported from time of first administration of study vaccine through 28 days after the last vaccination.

Table with similar format:

Table 136: Number and Percentage of Subjects Reporting AESIs Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status

Table 137: Duration (Days) of AESIs Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status

| Baseline Flavivirus<br>Immune Status | MedDRA System<br>Organ Class | MedDRA Preferred Term | Statistic | 2.5 mcg ZPIV<br>(N=X) | 5 mcg ZPIV<br>(N=X) | Placebo<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|
| | | | n | х | х | х | х |
| | | A my DT | Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | | Any PT | Median | x.x | x.x | x.x | x.x |
| | Any SOC | | Min, Max | x, x | x, x | X, X | X, X |
| | Ally SOC | | n | | | | |
| | | [PT 1] | Mean (SD) | | | | |
| | | | Median | | | | |
| | | | Min, Max | | | | |
| | | | n | | | | |
| | | Any PT | Mean (SD) | | | | |
| | | Any P1 | Median | | | | |
| All Subjects | [SOC 1] | | Min, Max | | | | |
| (N*=X) | | | n | | | | |
| | | [PT 1] | Mean (SD) | | | | |
| | | | Median | | | | |
| | | | Min, Max | | | | |
| | | | n | | | | |
| | | Any PT | Mean (SD) | | | | |
| | | Any P1 | Median | | | | |
| | [800.3] | | Min, Max | | | | |
| | [SOC 2] | | n | | | | |
| | | [DT 1] | Mean (SD) | | | | |
| | | [PT 1] | Median | | | | |
| | | | Min, Max | | | | |

Table 137: Duration (Days) of AESIs Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status (continued)

| Baseline Flavivirus<br>Immune Status | MedDRA System<br>Organ Class | MedDRA Preferred Term | Statistic | 2.5 mcg ZPIV<br>(N=X) | 5 mcg ZPIV<br>(N=X) | Placebo<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|
| Repeat for: | | | | | | | • |
| Baseline ZIKV Seroj<br>(N* = X) | positive | | | | | | |
| Baseline ZIKV Seron (N* = X) | negative | | | | | | |
| Baseline ZIKV Seroj<br>(N* = X) | positive and DENV Ser | opositive | | | | | |
| Baseline ZIKV Seroj<br>(N* = X) | positive and DENV Ser | onegative | | | | | |
| Baseline ZIKV Seron (N* = X) | negative and DENV Se | ropositive | | | | | |
| Baseline ZIKV Seron (N* = X) | negative and DENV Se | ronegative | | | | | |
| • | , , , , , , | oulation; N* = Number of su<br>elated to study treatment | bjects in the Sa | afety population with the s | pecified flavivirus status | used as the denominat | or for percentages; n = |

Table with similar format to Table 110:

Table 138: Number and Percentage of Subjects Reporting Serious Adverse Events Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status

Table with similar format to Table 111:

Table 139: Duration (Days) of Serious Adverse Events Related to Study Treatment by MedDRA System Organ Class, Preferred Term, Treatment Group, and Baseline Flavivirus Immune Status

Table 140: Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – All Subjects

[Implementation note: This table can include any subjects who did not have a baseline flavivirus status observed.]

| | | 2.5 mcg<br>(N= | | | | 5 mcg /<br>(N= | | | | Place<br>(N= | | | | All Sub<br>(N=) | • | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Infection Confirmation<br>Status | Number<br>of<br>Events | of | % of Subjects | 95% CI | Number<br>of<br>Events | Number<br>of<br>Subjects | % of Subjects | 95% CI | Number<br>of Events | Number<br>of<br>Subjects | % of<br>Subjects | 95% CI | Number<br>of Events | Number<br>of<br>Subjects | % of Subjects | 95%<br>CI |
| All Events | X | X | XX | x.x, x.x | X | X | XX | x.x, x.x | х | x | xx | x.x, x.x | х | х | XX | x.x, x.x |
| Events Requiring<br>Concomitant Medication | | | | | | | | | | | | | | | | |
| Events Requiring Medical<br>Treatment <sup>a</sup> | | | | | | | | | | | | | | | | |

N = Number of subjects in the Safety population

## Tables with similar format:

# Table 141: Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seropositive Subjects

[Implementation note: If no subjects are flavivirus positive at baseline, replace this table with the following note: 'Table not generated since no positive arbovirus results were reported for ZIKV or DENV.']

- Table 142: Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative Subjects
- Table 143: Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects
- Table 144: Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects
- Table 145: Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects

<sup>%=</sup>percentage of subjects reporting at least one AFI/ARI event out of total number of subjects in the Safety population in the group

<sup>95%</sup> CI is calculated using the Clopper-Pearson methodology for a binomial distribution.

This table includes subjects who only received dose 1.

<sup>&</sup>lt;sup>c</sup>Includes hospitalization or other medical care

Table 146: Summary of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects

# Table 147: Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method – All Subjects

[Implementation note: This table can include any subjects who did not have a baseline flavivirus status observed.]

| | | 2.5 mcg<br>(N= | | | | 5 mcg /<br>(N=) | | | | Place<br>(N=) | | | | All Sub<br>(N=) | J | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Infection Confirmation<br>Status | Number<br>of<br>Events | of | % of<br>Subjects | 95% CI | Number<br>of Events | Number<br>of<br>Subjects | % of | 95% CI | Number<br>of Events | Number<br>of<br>Subjects | % of Subjects | 95% CI | Number<br>of Events | Number<br>of<br>Subjects | % of<br>Subjects | 95%<br>CI |
| Positive by PCR <sup>a</sup> | X | X | XX | x.x, x.x | X | Х | XX | x.x, x.x | Х | X | XX | x.x, x.x | х | X | XX | x.x, x.x |
| Positive by 4-Fold Titer Rise <sup>b</sup> | | | | | | | | | | | | | | | | |
| Any Positive Confirmation <sup>a,b</sup> | | | | | | | | | | | | | | | | |
| Negative Lab Confirmation | | | · | | | | | | | | | | | | | |

N = Number of subjects in the Safety Population

<sup>%=</sup>percentage of subjects reporting at least one AFI/ARI event/total number of subjects in the Safety population in the group

<sup>95%</sup> CI is calculated using the Clopper-Pearson methodology for a binomial distribution.

This table includes subjects who only received dose 1.

<sup>&</sup>lt;sup>a</sup> PCR confirmation includes a positive PCR result for at least one of ZIKV (blood or urine) or DENV.

<sup>&</sup>lt;sup>b</sup> 4-fold rise in either ZIKV or DENV neutralization titers after the ARI/AFI illness visit compared to before the illness visit.

<sup>&</sup>lt;sup>c</sup>Includes hospitalization or other medical care

## Tables with similar format:

- Table 148: Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method Baseline ZIKV Seropositive Subjects
- Table 149: Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method Baseline ZIKV Seronegative Subjects
- Table 150: Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method Baseline ZIKV Seropositive and DENV Seropositive Subjects
- Table 151: Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method Baseline ZIKV Seropositive and DENV Seronegative Subjects
- Table 152: Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method Baseline ZIKV Seronegative and DENV Seropositive Subjects
- Table 153: Number of Laboratory Confirmed ZIKV or DENV Infections Overall and by Confirmation Method Baseline ZIKV Seronegative and DENV Seronegative Subjects

Table 154: Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method – All Subjects

[Implementation note: This table can include any subjects who did not have a baseline flavivirus status observed.]

| | | 2.5 mcg<br>(N*= | | | | 5 mcg !<br>(N*= | | | | Place<br>(N*= | | | | All Sub<br>(N*= | jects<br>X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Infection Confirmation<br>Status | Number<br>of<br>Subjects | Number<br>of<br>Events | % of<br>Events | 95% CI | Number<br>of<br>Subjects | Number<br>of<br>Events | % of<br>Events | 95% CI | Number<br>of<br>Subjects | Number<br>of<br>Events | % of<br>Events | 95% CI | Number<br>of<br>Subjects | Number<br>of<br>Events | % of<br>Events | 95%<br>CI |
| | | | | | | | All Events | | | | | | | | | |
| Positive by PCR <sup>a</sup> | X | X | XX | x.x, x.x | X | x | XX | x.x, x.x | х | X | XX | x.x, x.x | х | х | XX | x.x, x.x |
| Positive by 4-Fold Titer Rise <sup>b</sup> | | | | | | | | | | | | | | | | |
| Any Positive Confirmation <sup>a,b</sup> | | | | | | | | | | | | | | | | |
| Negative Lab Confirmation | | | | | | | | | | | | | | | | |
| | | | | | Even | nts Requirin | g Concom | itant Medi | cation | | | | | | | |
| Positive by PCR <sup>a</sup> | | | | | | | | | | | | | | | | |
| Positive by 4-Fold Titer Rise <sup>b</sup> | | | | | | | | | | | | | | | | |
| Any Positive Confirmation <sup>a,b</sup> | | | | | | | | | | | | | | | | |
| Negative Lab Confirmation | | | | | | | | | | | | | | | | |
| | | | | | Ev | vents Requi | ring Medic | al Treatme | ent <sup>c</sup> | | | | | | | |
| Positive by PCR <sup>a</sup> | | | | | | | | | | | | | | | | |
| Positive by 4-Fold Titer Rise <sup>b</sup> | | | | | | | | | | | | | | | | |
| Any Positive Confirmation <sup>a,b</sup> | | | | | | | | | | | | | | | | |
| Negative Lab Confirmation | | | | | | | | | | | | | | | | |
| $N^* = Total number of AFI/ARI$ | events | | • | • | • | • | • | • | | • | | • | | | | • |

 $N^* = \text{Total number of AFI/ARI events}$ 

<sup>%=</sup> number of AFI/ARI events / total number of AFI/ARI events (N\*)

<sup>95%</sup> CI is calculated using the Clopper-Pearson methodology for a binomial distribution.

This table includes subjects who only received dose 1.

<sup>&</sup>lt;sup>a</sup> PCR confirmation includes a positive PCR result for at least one of ZIKV (blood or urine) or DENV.

<sup>&</sup>lt;sup>b</sup> 4-fold rise in either ZIKV or DENV neutralization titers after the ARI/AFI illness visit compared to before the illness visit.

<sup>&</sup>lt;sup>c</sup>Includes hospitalization or other medical care

## Tables with similar format:

- Table 155: Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method Baseline ZIKV Seropositive Subjects
- Table 156: Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method Baseline ZIKV Seronegative Subjects
- Table 157: Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method Baseline ZIKV Seropositive and DENV Seropositive Subjects
- Table 158: Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method Baseline ZIKV Seropositive and DENV Seronegative Subjects
- Table 159: Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method Baseline ZIKV Seronegative and DENV Seropositive Subjects
- Table 160: Summary of ARI/AFI Events Occurring Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Status and Confirmation Method Baseline ZIKV Seronegative and DENV Seronegative Subjects

Table 161: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – All Subjects

[Implementation Note: If 100% of subject in all groups are counted in the "None" rows, then suppress the "Mild", "Moderate", and "Severe" columns. This table can include any subjects who did not have a baseline flavivirus status observed.]

| | | ncg ZPIV<br>(N=X) | | | | cg ZPIV<br>(N=X) | | | | lacebo<br>(N=X) | | All Subjects<br>(N=X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe |
| Symptom | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Any Symptom | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Fever | | | | | | | | | | | | | | | | |
| Feverishness | | | | | | | | | | | | | | | | |
| Lethargy | | | | | | | | | | | | | | | | |
| Restlessness | | | | | | | | | | | | | | | | |
| Rash not at injection site | | | | | | | | | | | | | | | | |
| Nonpurulent conjunctivitis | | | | | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | | | | | |
| Respiratory distress | | | | | | | | | | | | | | | | |
| Retro-orbital pain | | | | | | | | | | | | | | | | |
| Myalgia/Muscle pain | | | | | | | | | | | | | | | | |
| Arthralgia/Joint pain | | | | | | | | | | | | | | | | |
| Arthritis | | | | | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | | | | | |
| Abdominal pain | | | | | | | | | | | | | | | | |
| Vomiting* | | | | | | | | | | | | | | | | |
| Persistent vomiting* | | | | | | | | | | | | | | | | |
| Bleeding* | | | | | | | | | | | | | | | | |

Table 161: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – All Subjects

| | 2.5 mcg ZPIV<br>(N=X) | | | | | | icg ZPIV<br>(N=X) | | | | lacebo<br>(N=X) | | All Subjects<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe |
| Symptom | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

N = number of subjects reporting at least one AFI/ARI

n=number of subjects reporting the symptom

%=percentage of subjects reporting the symptom out of the total number of subjects reporting at least one AFI/ARI

If multiple AFI/ARI are reported for a subject, then the maximum severity is considered for each symptom.

This table includes subjects who only received dose 1.

\* Reported as None/Any

#### Tables with similar format:

- Table 162: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive Subjects
- Table 163: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative Subjects
- Table 164: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects
- Table 165: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects
- Table 166: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects
- Table 167: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative and DENV Seronegative Subjects

# Table 168: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – All Subjects

[Implementation Note: If 100% of AFI/ARI events in all columns are counted in the "None" rows, then suppress the "Mild", "Moderate", and "Severe" columns. This table can include any subjects who did not have a baseline flavivirus status observed.]

| Infection Confirmation Status | | cg ZPIV<br>N=X) | | | eg ZPIV<br>N=X) | | | | acebo<br>N=X) | | All Subjects (N=X) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Any Symptom | | | | | | | | | | | | | | | | |
| Positive by PCR <sup>a</sup> (N*=X) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Positive by 4-Fold Titer Rise <sup>b</sup> (N*=X) | | | | | | | | | | | | | | | | |
| Any Positive Confirmation <sup>a,b</sup> (N*=X) | | | | | | | | | | | | | | | | |
| Negative Lab Confirmation (N*=X) | | | | | | | | | | | | | | | | |
| Repeat for: | | | | | | | | | | | | | | | | |
| Fever | | | | | | | | | | | | | | | | |
| Feverishness | | | | | | | | | | | | | | | | |
| Lethargy | | | | | | | | | | | | | | | | |
| Restlessness | | | | | | | | | | | | | | | | |
| Rash not at injection site | | | | | | | | | | | | | | | | |
| Nonpurulent conjunctivitis | | | | | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | | | | | |
| Respiratory distress | | | | | | | | | | | | | | | | |
| Retro-orbital pain | | | | | | | | | | | | | | | | |
| Myalgia/Muscle pain | | | | | | | | | | | | | | | | |
| Arthralgia/Joint pain | | | | | | | | | | | | | | | | |
| Arthritis | | | | | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | | | | | |
| Abdominal pain | | | | | | | | | | | | | | | | |
| Vomiting* | | | | | | | | | | | | | | | | |
| Persistent vomiting* | | | | | | | | | | | | | | | | |

Table 168: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group – All Subjects (continued)

| | 2.5 mcg ZPIV<br>(N=X) | | | | 5 mcg ZPIV<br>(N=X) | | | | | | acebo<br>N=X) | | All Subjects<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Infection Confirmation Status | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

#### Bleeding\*

N = number of subjects reporting at least one AFI/ARI

N\* = Number of subjects with ARI/AFI and specified confirmation results n = number of subjects reporting the symptom

%=number of subjects reporting the symptom out of N\*

If multiple AFI/ARI are reported for a subject, then the maximum severity is considered for each symptom. "4-Fold Rise" refers to at least a 4-fold rise in ZIKV or DENV MN50 titers after the AFI/ARI illness visit compared to before the illness visit.

This table includes subjects who only received dose 1.

\* Reported as None/Any

#### Tables with similar format:

- Table 169: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group Baseline ZIKV Seropositive Subjects
- Table 170: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group Baseline ZIKV Seronegative Subjects
- Table 171: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects
- Table 172: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects
- Table 173: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects
- Table 174: Maximum Severity of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by ZIKV or DENV Infection Confirmation Status and Treatment Group Baseline ZIKV Seronegative and DENV Seronegative Subjects
Table 175: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – All Subjects

[Implementation note: This table can include any subjects who did not have a baseline flavivirus status observed.]

| Symptom | | 2.5 mc;<br>(N= | g ZPIV<br>=X) | | | 5 mcg<br>(N= | ZPIV<br>=X) | | | | cebo<br>=X) | | | | bjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max |
| Any Symptom | х | x.x (x.x) | x.x | x, x | Х | x.x (x.x) | x.x | x, x | X | x.x (x.x) | x.x | x, x | X | x.x (x.x) | x.x | x, x |
| Repeat for: | | | | | | | | | | | | | | | | |
| Fever | | | | | | | | | | | | | | | | |
| Feverishness | | | | | | | | | | | | | | | | |
| Lethargy | | | | | | | | | | | | | | | | |
| Restlessness | | | | | | | | | | | | | | | | |
| Rash not at injection site | | | | | | | | | | | | | | | | |
| Nonpurulent conjunctivitis | | | | | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | | | | | |
| Respiratory distress | | | | | | | | | | | | | | | | |
| Retro-orbital pain | | | | | | | | | | | | | | | | |
| Myalgia/Muscle pain | | | | | | | | | | | | | | | | |
| Arthralgia/Joint pain | | | | | | | | | | | | | | | | |
| Arthritis | | | | | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | | | | | |
| Abdominal pain | | | | | | | | | | | | | | | | |
| Vomiting* | | | | | | | | | | | | | | | | |
| Persistent vomiting* | | | | | | | | | | | | | | | | |
| Bleeding* | | | | | | | | | | | | | | | | |

Table 175: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group – All Subjects (continued)

| Symptom 2.5 mcg ZPIV (N=X) 5 mcg ZPIV (N=X) Placebo (N=X) | All Subjects<br>(N=X) |
|---|---|
|---|---|

N = number of subjects reporting at least one AFI/ARI

n = number of subjects reporting the symptom

If multiple AFI/ARI are reported for a subject, then the maximum severity is considered for each symptom; if multiple AFI/ARI are reported for a subject, then the maximum duration is considered for each symptom

This table includes subjects who only received dose 1.

\* Reported as None/Any

#### Tables with similar format:

- Table 176: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive Subjects
- Table 177: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative Subjects
- Table 178: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects
- Table 179: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects
- Table 180: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects
- Table 181: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group Baseline ZIKV Seronegative and DENV Seronegative Subjects

Table 182: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status – All Subjects

[Implementation note: This table can include any subjects who did not have a baseline flavivirus status observed.]

| | | | 2.5 mc<br>(N* | g ZPIV<br>=X) | | | 5 mcg<br>(N* | ZPIV<br>=X) | | | | cebo<br>==X) | | | All Su<br>(N* | ibjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Infection<br>Confirmation Status | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max |
| | Positive by PCR <sup>a</sup> | X | x.x<br>(x.x) | x.x | x, x | X | x.x<br>(x.x) | x.x | x, x | X | x.x<br>(x.x) | x.x | x, x | X | x.x<br>(x.x) | x.x | x, x |
| | Positive by 4-Fold<br>Titer Rise <sup>b</sup> | | | | | | | | | | | | | | | | |
| Any Symptom | Any Positive<br>Confirmation <sup>a,b</sup> | | | | | | | | | | | | | | | | |
| | Negative Lab<br>Confirmation | | | | | | | | | | | | | | | | |
| Fever | | | | | | | | | | | | | | | | | |
| Feverishness | | | | | | | | | | | | | | | | | |
| Lethargy | | | | | | | | | | | | | | | | | |
| Restlessness | | | | | | | | | | | | | | | | | |
| Rash not at injection site | | | | | | | | | | | | | | | | | |
| Nonpurulent conjunctivitis | | | | | | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | | | | | | |
| Respiratory distress | | | | | | | | | | | | | | | | | |
| Retro-orbital pain | | | | | | | | | | | | | | | | | |
| Myalgia/Muscle pain | | | | | | | | | | | | | | | | | |
| Arthralgia/Joint pain | | | | | | | | | | | | | | | | | |
| Arthritis | | | | | | | | | | | | | | | | | |

Table 182: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status – All Subjects (continued)

| | | | 2.5 mc<br>(N* | g ZPIV<br>=X) | | | | ZPIV<br>=X) | | | | cebo<br>=X) | | | All Su<br>(N* | ıbjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Infection<br>Confirmation Status | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max | n | Mean<br>(SD) | Median | Min,<br>Max |
| Nausea | | | | | | | | | | | | | | | | | |
| Abdominal pain | | | | | | | | | | | | | | | | | |
| Vomiting* | | | | | | | | | | | | | | | | | |
| Persistent vomiting* | | | | | | | | | | | | | | | | | |
| Bleeding* | | | | | | | | | | | | | | | | | |

N\* = number of subjects reporting at least one AFI/ARI

If multiple AFI/ARI are reported for a subject, then the maximum severity is considered for each symptom; if multiple AFI/ARI are reported for a subject, then the maximum duration is considered for each symptom.

This table includes subjects who only received dose 1.

n = number of subjects reporting the symptom

<sup>&</sup>lt;sup>a</sup> PCR confirmation includes a positive PCR result for at least one of ZIKV (blood or urine) or DENV.

<sup>&</sup>lt;sup>b</sup> 4-fold rise in either ZIKV or DENV neutralization titers after the ARI/AFI illness visit compared to before the illness visit.

<sup>\*</sup> Reported as None/Any

#### Table with similar format:

- Table 183: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status Baseline ZIKV Seropositive Subjects
- Table 184: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status Baseline ZIKV Seronegative Subjects
- Table 185: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status Baseline ZIKV Seropositive and DENV Seropositive Subjects
- Table 186: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status Baseline ZIKV Seropositive and DENV Seronegative Subjects
- Table 187: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status Baseline ZIKV Seronegative and DENV Seropositive Subjects
- Table 188: Duration (Days) of Symptoms of AFI/ARI Events Reported Through 12 Months Post Final Vaccination by Treatment Group and ZIKV or DENV Infection Confirmation Status Baseline ZIKV Seronegative and DENV Seronegative Subjects

# 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

### **Table 189:** Listing of Serious Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | No. of Days<br>Post Dose<br>the Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | D: , Treatment ( | Group: , Baseline | Flavivirus Imn | nune Status:, A | E Number | : | | | | | | |
| Comments | s: | | | | | | | | | | | |
| Subject ID | D: , Treatment ( | Group: , Baseline | Flavivirus Imn | nune Status:, A | E Number | : | | | | | | |
| Comments | s: | | • | | | | | | | • | | |
| Listing inc | cludes serious a | dverse events rep | oorted at any tin | ne during the | study. | | | | | | | |

### Table 190: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days<br>Post<br>Associated<br>Dose<br>(Duration) | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Tr | reatment Group: , | Baseline Flavivir | us Immune Status | s:, AE Number: | | | | | | |
| <b>Comments:</b> | | | | | | | | | | |
| Subject ID: , Tr | reatment Group: , | Baseline Flavivir | us Immune Status | s:, AE Number: | | | | | | |
| Comments: | | | | | | | | | | |

### **Table 191: Listing of AESIs and NOCMCs**

[Implementation Note: sort order is Subject ID, Number of Doses Received at Time of Event, and Date of Product Administration.]

| Adverse Event | Number of<br>Doses Received<br>at Time of<br>Event | No. of Days<br>Post Associated<br>Dose | Duration of<br>Event | Severity | MedDRA<br>System Organ<br>Class | AESI? | NOCMC? | Relationship | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Trea | ntment Group: , Ba | seline Flavivirus Im | mune Status:, AE | Number: | | | | | |
| Comments: | | | | | | | | | |
| Subject ID: , Trea | ntment Group: , Ba | seline Flavivirus Im | mune Status:, AE I | Number: | | | | | |
| Comments: | | , | | | , | | | | |

### 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

[Placeholder for the CSR]

### 14.3.4 Abnormal Laboratory Value Listings (by Subject)

### **Table 192:** Listing of Abnormal Laboratory Results – Chemistry

| Subject<br>ID | Treatment<br>Group | Baseline<br>Flavivirus<br>Immune<br>Status | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Tables with similar format:

**Table 193:** Listing of Abnormal Laboratory Results – Hematology

**Table 194:** Listing of Abnormal Laboratory Results – Urinalysis

#### 14.3.5 Displays of Laboratory Results

### 14.3.5.1 Chemistry Results

Table 195: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Chemistry Parameter

| | | | N | one | | ild/<br>de 1 | Mode<br>Gra | | | | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Time Point</b> | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| All Subjects | | | | | | | | | | | | |
| | 2.5 mcg ZPIV | х | х | XX | x | xx | х | xx | x | xx | х | XX |
| D 1' | 5 mcg ZPIV | | | | | | | | | | | |
| Baseline | Placebo | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |
| Repeat for: | | | | | | | | | | | | |
| Day 8 | | | | | | | | | | | | |
| Day 15 | | | | | | | | | | | | |
| Day 36 | | | | | | | | | | | | |
| Day 43 | | | | | | | | | | | | |
| Max Severity Post Baseline | | | | | | | | | | | | |
| Danast for | 1 | | | 1 | | 1 | ı | ı | 1 | 1 | 1 | 1 |

Repeat for:

**Baseline ZIKV Seropositive** 

**Baseline ZIKV Seronegative** 

**Baseline ZIKV Seropositive and DENV Seropositive** 

**Baseline ZIKV Seropositive and DENV Seronegative** 

**Baseline ZIKV Seronegative and DENV Seropositive** 

**Baseline ZIKV Seronegative and DENV Seronegative** 

N=Number of subjects in the Safety population who completed the specified visit.

The "Max Severity Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

#### Tables with similar format:

- Table 196: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status ALT
- Table 197: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status AST
- Table 198: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status Total
  - **Bilirubin**
- Table 199: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status BUN
- Table 200: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status Creatinine

Table 201: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Chemistry Parameter

| | | | Mi<br>Gra | | | erate/<br>ide 2 | Sev<br>Gra | |
|---|---|---|---|---|---|---|---|---|
| <b>Time Point</b> | Treatment Group | N | n | % | n | % | n | % |
| All Subjects | · | | | | | | | |
| | 2.5 mcg ZPIV | X | x | xx | х | xx | x | XX |
| <b>D</b> | 5 mcg ZPIV | | | | | | | |
| Day 8 | Placebo | | | | | | | |
| | All Subjects | | | | | | | |
| Repeat for: | | | | | | | | |
| Day 15 | | | | | | | | |
| Day 36 | | | | | | | | |
| Day 43 | | | | | | | | |
| Max Severity Post<br>Baseline | | | | | | | | |
| Reneat for: | | | • | | • | • | • | |

Repeat for:

**Baseline ZIKV Seropositive** 

**Baseline ZIKV Seronegative** 

**Baseline ZIKV Seropositive and DENV Seropositive** 

**Baseline ZIKV Seropositive and DENV Seronegative** 

**Baseline ZIKV Seronegative and DENV Seropositive** 

**Baseline ZIKV Seronegative and DENV Seronegative** 

N=Number of subjects in the safety population who completed the specified visit and results are available.

The "Max Severity Post Baseline" rows indicate the maximum severity of abnormal laboratory results related to study treatment experienced by each subject at any time point post baseline, including unscheduled assessments.

#### Tables with similar format:

- Table 202: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status ALT
- Table 203: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status AST
- Table 204: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status Total Bilirubin
- Table 205: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status BUN
- Table 206: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status Creatinine

**Table 207:** Laboratory Summary Statistics by Time Point and Treatment Group – ALT

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| All Subjects | · | | | | | |
| | 2.5 mcg ZPIV | xx | XX.X | xx.x | xx | xx, xx |
| t | 5 mcg ZPIV | | | | | |
| Baseline | Placebo | | | | | |
| | All Subjects | | | | | |
| Repeat for: | | | | | | |
| Day 8 | | | | | | |
| Day 8, Change from Baseline | | | | | | |
| Day 15 | | | | | | |
| Day 15, Change from Baseline | | | | | | |
| Day 36 | | | | | | |
| Day 36, Change from Baseline | | | | | | |
| Day 43 | | | | | | |
| Day 43, Change from Baseline | | | | | | |
| Repeat for: | | | | | | |
| Baseline ZIKV Seropositive | | | | | | |
| Baseline ZIKV Seronegative | | | | | | |
| Baseline ZIKV Seropositive and DENV<br>Seropositive | | | | | | |
| Baseline ZIKV Seropositive and DENV<br>Seronegative | | | | | | |
| Baseline ZIKV Seronegative and DENV<br>Seropositive | | | | | | |
| Baseline ZIKV Seronegative and DENV<br>Seronegative | | | | | | |
| N=Number of subjects in the Safety population w | ho completed the specified visit and r | esults are availab | le. | - | | |

#### Tables with similar format:

Table 208: Laboratory Summary Statistics by Time Point and Treatment Group – AST

Table 209: Laboratory Summary Statistics by Time Point and Treatment Group – Total Bilirubin

Table 210: Laboratory Summary Statistics by Time Point and Treatment Group – BUN

Table 211: Laboratory Summary Statistics by Time Point and Treatment Group – Creatinine

### 14.3.5.2 Hematology Results

Table with format similar to Table 195:

Table 212: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Hematology Parameter

Table 213: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – WBC

| Time Point | Transferrent | | No | one | Gra | ild/<br>ide 1<br>ow) | Gra | ild/<br>de 1<br>igh) | Gra | erate/<br>de 2<br>ow) | Gra | erate/<br>de 2<br>gh) | Gra | rere/<br>ide 3<br>ow) | Gra | vere/<br>ade 3<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment<br>Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| All Subjects | | | • | • | • | • | • | • | | • | • | | | • | • | • | • | |
| | 2.5 mcg ZPIV | x | х | xx | X | xx | X | XX | X | xx | X | XX | X | xx | х | XX | х | XX |
| | 5 mcg ZPIV | | | | | | | | | | | | | | | | | |
| Baseline | Placebo | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |
| Repeat for: | | | | | | | | | | | | | | | | | | |
| Day 8 | | | | | | | | | | | | | | | | | | |
| Day 15 | | | | | | | | | | | | | | | | | | |
| Day 36 | | | | | | | | | | | | | | | | | | |
| Day 43 | | | | | | | | | | | | | | | | | | |
| Max Severity<br>Post Baseline | | | | | | | | | | | | | | | | | | |

Repeat for:

**Baseline ZIKV Seropositive** 

**Baseline ZIKV Seronegative** 

**Baseline ZIKV Seropositive and DENV Seropositive** 

**Baseline ZIKV Seropositive and DENV Seronegative** 

**Baseline ZIKV Seronegative and DENV Seropositive** 

**Baseline ZIKV Seronegative and DENV Seronegative** 

N=Number of subjects in the Safety population who completed the specified visit.

The "Max Severity Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

Table with format similar to Table 195:

Table 214: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status—Hemoglobin

Table with format similar to Table 213:

Table 215: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status–Hematocrit

Table with format similar to Table 195:

Table 216: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status—Platelet Count

Table with format similar to Table 201:

Table 217: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any Hematology Parameter

Table 218: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status—WBC

| | | | Gra | ild/<br>nde 1<br>ow) | Gra | ild/<br>de 1<br>gh) | Gra | erate/<br>nde 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | ere/<br>de 3<br>ow) | Gra | vere/<br>ade 3<br>igh) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| All Subjects | | | | • | | | | • | | | • | | | |
| | 2.5 mcg ZPIV | X | Х | XX | х | XX | Х | xx | Х | XX | x | XX | Х | XX |
| D 0 | 5 mcg ZPIV | | | | | | | | | | | | | |
| Day 8 | Placebo | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | |
| Repeat for: | | | | | | | | | | | | | | |
| Day 15 | | | | | | | | | | | | | | |
| Day 36 | | | | | | | | | | | | | | |
| Day 43 | | | | | | | | | | | | | | |
| Max Severity Post Baseline | | | | | | | | | | | | | | |
| Repeat for: | | | | | | | | | | | | | | |
| Baseline ZIKV Seropositive | | | | | | | | | | | | | | |
| Baseline ZIKV Seronegative | | | | | | | | | | | | | | |
| Baseline ZIKV Seropositive and DENV Seropositive | | | | | | | | | | | | | | |
| Baseline ZIKV Seropositive and DENV Seronegative | | | | | | | | | | | | | | |
| Baseline ZIKV Seronegative and DENV Seropositive | | | | | | | | | | | | | | |
| Baseline ZIKV Seronegative and DENV Seronegative | | | | | | | | | | | | | | |

N=Number of subjects in the safety population who completed the specified visit and results are available.

The "Max Severity Post Baseline" rows indicate the maximum severity of abnormal laboratory results related to study treatment experienced by each subject at any time point post baseline, including unscheduled assessments.

Table with format similar to Table 201:

Table 219: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Hemoglobin

Table with format similar to Table 218:

Table 220: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Hematocrit

Table with format similar to Table 201:

Table 221: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Platelet Count

#### Tables with format similar to Table 207:

- Table 222: Laboratory Summary Statistics by Time Point and Treatment Group WBC
- Table 223: Laboratory Summary Statistics by Time Point and Treatment Group Hemoglobin
- Table 224: Laboratory Summary Statistics by Time Point and Treatment Group Hematocrit
- Table 225: Laboratory Summary Statistics by Time Point and Treatment Group Platelet Count

#### 14.3.5.3 Urinalysis Results

Tables with format similar to Table 195:

Table 226: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and

**Baseline Flavivirus Immune Status – Any Urinalysis Parameter** 

Table 227: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and

**Baseline Flavivirus Immune Status – Urine Protein** 

Table 228: Laboratory Results by Maximum Severity, Time Point, Treatment Group, and

**Baseline Flavivirus Immune Status- Urine Glucose** 

Tables with format similar to Table 201:

Table 229: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity,

Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Any

**Urinalysis Parameter** 

Table 230: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity,

Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Urine

**Protein** 

Table 231: Abnormal Laboratory Results Related to Study Treatment by Maximum Severity,

Time Point, Treatment Group, and Baseline Flavivirus Immune Status – Urine

Glucose

### 14.3.6 Displays of Vital Signs

Table 232: Vital Signs by Maximum Severity, Time Point and Treatment Group – Any Assessment

| | | | N | one | | ild/<br>ade 1 | | lerate/<br>ade 2 | | vere/<br>ade 3 | Any S | everity |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Time Point</b> | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | 2.5 mcg ZPIV | XX | xx | xx | XX | xx | xx | XX | xx | xx | xx | XX |
| Danilia. | 5 mcg ZPIV | | | | | | | | | | | |
| Baseline | Placebo | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |
| Repeat for: | | | | | | | | | | | | |
| Day 1 | | | | | | | | | | | | |
| Day 2 | | | | | | | | | | | | |
| Day 8 | | | | | | | | | | | | |
| Day 15 | | | | | | | | | | | | |
| Day 29 | | | | | | | | | | | | |
| Day 30 | | | | | | | | | | | | |
| Day 36 | | | | | | | | | | | | |
| Day 43 | | | | | | | | | | | | |
| Day 57 | | | | | | | | | | | | |
| Max Severity Post Baseline | | | | | | | | | | | | |

N=Number of subjects in the Safety population who completed the specified visit and have any vital signs data available from the visit.

The "Max Severity Post Baseline" rows indicates the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

#### Tables with similar format:

- Table 233: Vital Signs by Maximum Severity, Time Point and Treatment Group Oral Temperature
- Table 234: Vital Signs by Maximum Severity, Time Point and Treatment Group Pulse
- Table 235: Vital Signs by Maximum Severity, Time Point and Treatment Group Systolic Blood Pressure
- Table 236: Vital Signs by Maximum Severity, Time Point and Treatment Group Diastolic Blood Pressure

### 14.4 Summary of Concomitant Medications

Table 237: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group

| | | | 2.5 mcg ZPIV<br>(N=X) | | 5 mcg ZPIV<br>(N=X) | | Placebo<br>(N=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|
| WHO Drug Code<br>Level 1, Anatomic Group | WHO Drug Code<br>Level 2, Therapeutic Subgroup | n | % | n | % | n | % | n | % |
| Any Level 1 Code | Any Level 2 Code | x | XX | х | xx | X | xx | х | xx |
| | [Any Level 1, Code 1] | | | | | | | | |
| n - 11 C 1 11 | [Level 2, Code 1] | | | | | | | | |
| [Level 1, Code 1] | [Level 2, Code 2] | | | | | | | | |
| | [Etc.] | | | | | | | | |
| | [Any Level 1, Code 2] | | | | | | | | |
| FI - 11 C 1 21 | [Level 2, Code 1] | | | | | | | | |
| [Level 1, Code 2] | [Level 2, Code 2] | | | | | | | | |
| | [Etc.] | | | | | | | | |
| | Any | | | | | | | | |
| | [Level 2, Code 1] | | | | | | | | |
| [Etc.] | [Level 2, Code 2] | | | | | | | | |
| | [Etc.] | | | | | | | | |

N = Number of subjects in the Safety population

n = Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

## APPENDIX 2. FIGURE MOCK-UPS

## LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 170 |
|---|---|---|
| Figure 2: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – All Subjects – Immunogenicity Population | 171 |
| Figure 3: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – All Subjects – Per Protocol Population | 172 |
| Figure 4: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seropositive Subjects – Immunogenicity Population | 172 |
| Figure 5: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seropositive Subjects – Per Protocol Population | 172 |
| Figure 6: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seronegative Subjects – Immunogenicity Population | 172 |
| Figure 7: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seronegative Subjects, – Per Protocol Population | |
| Figure 8: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Immunogenicity Population. | 172 |
| Figure 9: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Per Protocol Population | 172 |
| Figure 10: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects – Immunogenicity Population | 172 |
| Figure 11: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects – Per Protocol Population | |
| Figure 12: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects – Immunogenicity Population | 172 |
| Figure 13: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects – Per Protocol Population | |

| Figure 14: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects – Immunogenicity Population |
|---|---|
| Figure 15: | Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects – Per Protocol Population172 |
| Figure 16: | Geometric Mean ZIKV Microneutralization (MN50) Titer (GMT), by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population |
| Figure 17: | Geometric Mean ZIKV Microneutralization (MN50) Titer (GMT), by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population |
| Figure 18: | Percent of Subjects Seropositive at Threshold of ≥10 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population |
| Figure 19: | Percent of Subjects Seropositive at Threshold of ≥10 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population |
| Figure 20: | Percent of Subjects Seropositive at Threshold of ≥100 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population176 |
| Figure 21: | Percent of Subjects Seropositive at Threshold of ≥100 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population |
| Figure 22: | Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population |
| Figure 23: | Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV<br>Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status,<br>Time Point, and Treatment Group – Per Protocol Population |
| Figure 24: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – All Subjects – Immunogenicity Population |
| Figure 25: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – All Subjects – Per Protocol Population |
| Figure 26: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seropositive Subjects – Immunogenicity Population |

| Figure 27: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seropositive Subjects – Per Protocol Population | 177 |
|---|---|---|
| Figure 28 | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seronegative Subjects – Immunogenicity Population | 177 |
| Figure 29: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seronegative Subjects – Per Protocol Population | 177 |
| Figure 30: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Immunogenicity Population | 177 |
| Figure 31: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seropositive Subjects – Per Protocol Population | 177 |
| Figure 32: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects – Immunogenicity Population | 177 |
| Figure 33: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seropositive and DENV Seronegative Subjects – Per Protocol Population | 177 |
| Figure 34 | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects – Immunogenicity Population | 177 |
| Figure 35: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seropositive Subjects – Per Protocol Population | 177 |
| Figure 36 | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects – Immunogenicity Population | |
| Figure 37: | Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group – Baseline ZIKV Seronegative and DENV Seronegative Subjects – Per Protocol Population | 177 |
| Figure 38: | Geometric Mean ZIKV ELISA Titer (GMT) by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population | 178 |
| Figure 39: | Geometric Mean ZIKV ELISA Titer (GMT) by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population | 178 |
| Figure 40: | Percent of Subjects Seropositive at Threshold of ≥200 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population | 178 |

| Figure 41: | Percent of Subjects Seropositive at Threshold of ≥200 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population | 178 |
|---|---|---|
| Figure 42: | Percent of Subjects Seropositive at Threshold of ≥600 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population | 178 |
| Figure 43: | Percent of Subjects Seropositive at Threshold of ≥600 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population | 178 |
| Figure 44: | Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population | 178 |
| Figure 45: | Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population | 178 |
| Figure 46: | Maximum Severity of Solicited Local Adverse Events by Symptom and Treatment Group – Post Any Dose | 179 |
| Figure 47: | Maximum Severity of Solicited Local Adverse Events by Symptom and Treatment Group – Post Dose 1 | 180 |
| Figure 48: | Maximum Severity of Solicited Local Adverse Events by Symptom and Treatment Group – Post Dose 2 | 180 |
| Figure 49: | Maximum Severity of Solicited Systemic Adverse Events by Symptom and Treatment Group – Post Any Dose | 181 |
| Figure 50: | Maximum Severity of Solicited Systemic Adverse Events by Symptom and Treatment Group – Post Dose 1 | 182 |
| Figure 51: | Maximum Severity of Solicited Systemic Adverse Events by Symptom and Treatment Group – Post Dose 2 | 182 |
| Figure 52: | Maximum Severity of Solicited Local Symptoms by Days Post Treatment and Treatment Group – Post Any Dose | 183 |
| Figure 53: | Maximum Severity of Solicited Local Symptoms by Days Post Treatment and Treatment Group – Post Dose 1 | 184 |
| Figure 54: | Maximum Severity of Solicited Local Symptoms by Days Post Treatment and Treatment Group – Post Dose 2 | 184 |
| Figure 55: | Maximum Severity of Solicited Systemic Symptoms by Days Post Treatment and Treatment Group – Post Any Dose | 185 |
| Figure 56: | Maximum Severity of Solicited Systemic Symptoms by Days Post Treatment and Treatment Group – Post Dose 1 | 186 |
| Figure 57: | Maximum Severity of Solicited Systemic Symptoms by Days Post Treatment and Treatment Group – Post Dose 2 | |

| Figure 58: | Frequency of Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity – Post-Any Dose | 187 |
|---|---|---|
| Figure 59: | Frequency of Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity – Post-Dose 1 | 188 |
| Figure 60: | Frequency of Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity – Post- Dose 2 | 188 |
| Figure 61: | Frequency of Related Adverse Events by MedDRA System Organ Class,<br>Treatment Group, and Severity – Post-Any Dose | 188 |
| Figure 62: | Frequency of Related Adverse Events by MedDRA System Organ Class,<br>Treatment Group, and Severity – Post-Dose 1 | 188 |
| Figure 63: | Frequency of Related Adverse Events by MedDRA System Organ Class,<br>Treatment Group, and Severity – Post- Dose 2 | 188 |
| Figure 64: | Clinical Laboratory Results by Maximum Severity and Treatment Group – Chemistry | 189 |
| Figure 65: | Clinical Laboratory Results by Maximum Severity and Treatment Group – Hematology | 190 |
| Figure 66: | Clinical Laboratory Results by Maximum Severity and Treatment Group – Urinalysis | 191 |
| Figure 67: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – ALT | 192 |
| Figure 68: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – AST | 193 |
| Figure 69: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – Total Bilirubin | 193 |
| Figure 70: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – BUN | 193 |
| Figure 71: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – Creatinine | 193 |
| Figure 72: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – WBC | 193 |
| Figure 73: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – Hemoglobin | 193 |
| Figure 74: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – Hematocrit | 193 |
| Figure 75: | Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – Platelet Count | |

#### 10.1 Disposition of Subjects

Figure 1: CONSORT Flow Diagram


### 14.2.2 Immunogenicity Response Figures by Measure, Treatment Group, and Time Point

Figure 2: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group – All Subjects – Immunogenicity Population



Figures with format similar to Figure 2:

- Figure 3: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group All Subjects Per Protocol Population
- Figure 4: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seropositive Subjects Immunogenicity Population
- Figure 5: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seropositive Subjects Per Protocol Population
- Figure 6: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seronegative Subjects Immunogenicity Population
- Figure 7: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seronegative Subjects, Per Protocol Population
- Figure 8: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects Immunogenicity Population
- Figure 9: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects Per Protocol Population
- Figure 10: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects Immunogenicity Population
- Figure 11: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects Per Protocol Population
- Figure 12: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects Immunogenicity Population
- Figure 13: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects Per Protocol Population
- Figure 14: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seronegative Subjects Immunogenicity Population
- Figure 15: Reverse Cumulative Distribution of ZIKV Microneutralization Assay (MN50) Titer by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seronegative Subjects Per Protocol Population

Figure 16: Geometric Mean ZIKV Microneutralization (MN50) Titer (GMT), by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population



Note: The bars represent the upper and lower limits of the 95% confidence interval for GMT.

Figure with similar format:

Figure 17: Geometric Mean ZIKV Microneutralization (MN50) Titer (GMT), by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Per Protocol Population

Figure 18: Percent of Subjects Seropositive at Threshold of ≥10 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group – Immunogenicity Population



Note: The bars represent the upper and lower limits of the 95% confidence interval for the percent of subjects seropositive.

#### Figures with similar format:

- Figure 19: Percent of Subjects Seropositive at Threshold of ≥10 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Per Protocol Population
- Figure 20: Percent of Subjects Seropositive at Threshold of ≥100 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Immunogenicity Population
- Figure 21: Percent of Subjects Seropositive at Threshold of ≥100 of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Per Protocol Population
- Figure 22: Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Immunogenicity Population
- Figure 23: Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV Microneutralization (MN50) Assay, by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Per Protocol Population

Same formats as Figure 2 to Figure 23:

#### RCD Curves

- Figure 24: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group All Subjects Immunogenicity Population
- Figure 25: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group All Subjects Per Protocol Population
- Figure 26: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seropositive Subjects Immunogenicity Population
- Figure 27: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seropositive Subjects Per Protocol Population
- Figure 28 Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seronegative Subjects Immunogenicity Population
- Figure 29: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seronegative Subjects Per Protocol Population
- Figure 30: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects Immunogenicity Population
- Figure 31: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seropositive Subjects Per Protocol Population
- Figure 32: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects Immunogenicity Population
- Figure 33: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seropositive and DENV Seronegative Subjects Per Protocol Population
- Figure 34 Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects Immunogenicity Population
- Figure 35: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seropositive Subjects Per Protocol Population
- Figure 36 Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seronegative Subjects Immunogenicity Population
- Figure 37: Reverse Cumulative Distribution of ZIKV ELISA by Time Point and Treatment Group Baseline ZIKV Seronegative and DENV Seronegative Subjects Per Protocol Population

#### **GMT**

- Figure 38: Geometric Mean ZIKV ELISA Titer (GMT) by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Immunogenicity Population
- Figure 39: Geometric Mean ZIKV ELISA Titer (GMT) by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Per Protocol Population

#### Seropositivity, Threshold ≥200

- Figure 40: Percent of Subjects Seropositive at Threshold of ≥200 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Immunogenicity Population
- Figure 41: Percent of Subjects Seropositive at Threshold of ≥200 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Per Protocol Population

#### Seropositivity, Threshold ≥600

- Figure 42: Percent of Subjects Seropositive at Threshold of ≥600 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Immunogenicity Population
- Figure 43: Percent of Subjects Seropositive at Threshold of ≥600 of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Per Protocol Population

#### Seroconversion

- Figure 44: Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Immunogenicity Population
- Figure 45: Percent Seroconversion (≥4-Fold Rise from Baseline) of ZIKV ELISA Assay by Baseline Flavivirus Immune Status, Time Point, and Treatment Group Per Protocol Population

#### 14.3.1.1 Solicited Adverse Events

Figure 46: Maximum Severity of Solicited Local Adverse Events by Symptom and Treatment Group – Post Any Dose



Figures with format similar to Figure 46:

- Figure 47: Maximum Severity of Solicited Local Adverse Events by Symptom and Treatment Group Post Dose 1
- Figure 48: Maximum Severity of Solicited Local Adverse Events by Symptom and Treatment Group Post Dose 2

Figure 49: Maximum Severity of Solicited Systemic Adverse Events by Symptom and Treatment Group – Post Any Dose



Figures with format similar to Figure 49:

Figure 50: Maximum Severity of Solicited Systemic Adverse Events by Symptom and Treatment

**Group – Post Dose 1** 

Figure 51: Maximum Severity of Solicited Systemic Adverse Events by Symptom and Treatment

**Group – Post Dose 2** 

Figure 52: Maximum Severity of Solicited Local Symptoms by Days Post Treatment and Treatment Group – Post Any Dose



Figures with format similar to Figure 52:

- Figure 53: Maximum Severity of Solicited Local Symptoms by Days Post Treatment and Treatment Group Post Dose 1
- Figure 54: Maximum Severity of Solicited Local Symptoms by Days Post Treatment and Treatment Group Post Dose 2

Figure 55: Maximum Severity of Solicited Systemic Symptoms by Days Post Treatment and Treatment Group – Post Any Dose



Figures with format similar to Figure 55:

- Figure 56: Maximum Severity of Solicited Systemic Symptoms by Days Post Treatment and Treatment Group Post Dose 1
- Figure 57: Maximum Severity of Solicited Systemic Symptoms by Days Post Treatment and Treatment Group Post Dose 2

#### 14.3.1.2 Unsolicited Adverse Events

Figure 58: Frequency of Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity – Post-Any Dose



### Figures with similar format:

- Figure 59: Frequency of Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity Post-Dose 1
- Figure 60: Frequency of Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity Post- Dose 2
- Figure 61: Frequency of Related Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity Post-Any Dose
- Figure 62: Frequency of Related Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity Post-Dose 1
- Figure 63: Frequency of Related Adverse Events by MedDRA System Organ Class, Treatment Group, and Severity Post- Dose 2

### 14.3.5 Displays of Laboratory Results

#### 14.3.5.1 Chemistry Results

Figure 64: Clinical Laboratory Results by Maximum Severity and Treatment Group – Chemistry



### 14.3.5.2 Hematology Results

Figure 65: Clinical Laboratory Results by Maximum Severity and Treatment Group – Hematology



### 14.3.5.3 Urinalysis Results

Figure 66: Clinical Laboratory Results by Maximum Severity and Treatment Group – Urinalysis



#### 14.3.5 Displays of Laboratory Results

### Figure 67: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group – ALT

[Implementation note: the figure below is just an example. There will a single panel and individual curves for 2.5 mcg ZPIV, 5 mcg ZPIV and Placebo groups. The x-axis will have Day 8, Day 15, Day 36, and Day 43. Separate panels for male and female subjects will be generated for parameters graded separately by sex.]



The bars represent the upper and lower limits of the 95% confidence interval for mean change from baseline.

#### Figures with similar format:

- Figure 68: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group AST
- Figure 69: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group Total Bilirubin
- Figure 70: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group BUN
- Figure 71: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group Creatinine
- Figure 72: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group WBC
- Figure 73: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group Hemoglobin
- Figure 74: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group Hematocrit
- Figure 75: Laboratory Results by Time Point: Mean Changes from Baseline by Treatment Group Platelet Count

# APPENDIX 3. LISTINGS MOCK-UPS

# LISTINGS

| Listing 1: | Listing of Subjects Receiving Investigational Product | 196 |
|---|---|---|
| Listing 2: | Early Terminations or Discontinued Subjects | 197 |
| Listing 3: | Subject-Specific Protocol Deviations | 198 |
| Listing 4: | Non-Subject-Specific Protocol Deviations | 199 |
| Listing 5: | Subjects Excluded from Analysis Populations | 200 |
| Listing 6: | Demographic Data | 201 |
| Listing 7: | Pre-Existing and Concurrent Medical Conditions | 202 |
| Listing 8: | Individual Immunogenicity Response Data | 203 |
| Listing 9: | Solicited Events – Systemic Symptoms | 204 |
| Listing 10: | Solicited Events – Local Symptoms | 205 |
| Listing 11: | Unsolicited Adverse Events. | 206 |
| Listing 12: | Listing of Subject Information for Subjects Reporting ARI or AFI | 207 |
| Listing 13: | Listing of Medical Treatment Sought for Subjects Reporting ARI or AFI | 208 |
| Listing 14: | Listing of AFI/ARI Symptoms Reported in Subjects Experiencing ARI or AFI | 209 |
| Listing 15: | Listing of Vital Signs in Subjects Reporting ARI or AFI | |
| Listing 16: | Listing of Laboratory Results in Subjects Reporting ARI or AFI | 211 |
| Listing 17: | Clinical Laboratory Results – Chemistry | 212 |
| Listing 18: | Clinical Laboratory Results – Hematology | 213 |
| Listing 19: | Clinical Laboratory Results – Urinalysis | 214 |
| Listing 20: | Vital Signs | 215 |
| Listing 21: | Physical Exam Findings | 216 |
| Listing 22: | Concomitant Medications | 217 |
| Listing 23: | Pregnancy Reports – Maternal Information | 218 |
| Listing 24: | Pregnancy Reports – Gravida and Para | 218 |
| Listing 25: | Pregnancy Reports – Live Birth Outcomes | 219 |
| Listing 26: | Pregnancy Reports – Still Birth Outcomes | 219 |
| Listing 27: | Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion | 210 |

# **Listing 1:** Listing of Subjects Receiving Investigational Product

[Placeholder for the CSR]

# 16.2 Database Listings by Subject

# **16.2.1 Discontinued Subjects**

# **Listing 2:** Early Terminations or Discontinued Subjects

[Implementation note: Listing will be sorted by Treatment Group, Subject ID, alphabetically by Category.]

| Treatment Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

#### **16.2.2 Protocol Deviations**

# **Listing 3:** Subject-Specific Protocol Deviations

[Implementation note: Listing will be sorted by Treatment Group, Subject ID, DV number.]

| Treatment<br>Group | Subject<br>ID | Deviation<br>Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted<br>in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

# **Listing 4:** Non-Subject-Specific Protocol Deviations

[Implementation note: Listing will be sorted by DV number.]

| Deviation<br>Number | Deviation<br>Category | Start Date | End Date | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

### 16.2.3 Subjects Excluded from the Immunogenicity Analysis

# **Listing 5:** Subjects Excluded from Analysis Populations

[Implementation note: Listing will be sorted by Treatment Group, Subject ID]

| Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|
| | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |
| | Subject ID | Subject ID Subject is Included | Subject ID Subject is Included Subject is Excluded | Subject ID Subject is Included Subject is Excluded Results Available? |

<sup>&</sup>quot;Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

### 16.2.4 Demographic Data

### **Listing 6:** Demographic Data

[Implementation note: If a subject is multi-racial, in "Race" column, note "Multiple: (list races, separated by a comma)." The 'Seropositive Flaviviruses at Baseline' will list all flaviviruses that the subject was seropositive to at baseline, or 'None' if none. Listing will be sorted by Treatment Group then Subject ID.]

| Treatment Group | Subject ID | Age at Enrollment (years) | BMI at Screening (kg/m²) | Sex | Ethnicity | Race | Seropositive Flaviviruses at Baseline |
|---|---|---|---|---|---|---|---|

# **Listing 7:** Pre-Existing and Concurrent Medical Conditions

[Implementation note: Listing will be sorted by Treatment Group, Subject ID, MH number.]

| Treatment<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

### 16.2.6 Individual Immunogenicity Response Data

### **Listing 8:** Individual Immunogenicity Response Data

[Implementation note: Listing will be sorted by Treatment Group, Subject ID, Planned Time Point. The 'Seropositive Flaviviruses at Baseline' will list all flaviviruses that the subject was seropositive to at baseline, or 'None' if none.]

| Treatment Group | Subject ID | Seropositive<br>Flaviviruses at<br>Baseline | Planned Time Point | Actual Study Day | ZIKV MN50 Titer | ZIKV ELISA Titer | DENV MN50 Titer |
|---|---|---|---|---|---|---|---|

#### 16.2.7 Adverse Events

#### 16.2.7.1 Solicited Events

### **Listing 9:** Solicited Events – Systemic Symptoms

[Implementation note: Listing will be sorted by Treatment Group, Subject ID, Dose Number, Post Dose Day, Symptom.]

| Treatment<br>Group | Subject ID | Dose Number | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

### **Listing 10:** Solicited Events – Local Symptoms

[Implementation note: Listing will be sorted by Treatment Group, Subject ID, Dose Number, Post Dose Day, Symptom.]

| Treatment Group | Subject ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity |
|---|---|---|---|---|---|---|
| | | | | MA | | |
| | | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

#### 16.2.7.2 Unsolicited Events

### **Listing 11: Unsolicited Adverse Events**

[Implementation note: This listing includes all unsolicited adverse events. If the event is ongoing, indicate "ongoing" in the Duration column. Listing will be sorted by Treatment Group, Subject ID, Associated with Dose No., No. of Days Post Associated Dose.]

| Adverse<br>Event | Associated<br>with Dose<br>No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | | | I | l | | I | I | | | | |
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | <u>I</u> | | <u> </u> | <u>I</u> | | <u> </u> | <u> </u> | <u>I</u> | | 1 | |
| For addition | nal details about | SAEs, see the | table titled 'List | ting of Serious | Adverse Events | , . | | | | | |
# Listing 12: Listing of Subject Information for Subjects Reporting ARI or AFI

[Implementation note: Columns indicating a 4-fold rise in neutralization titers will be either 'No' or 'Yes; [Day X, Day Y]']

| Adverse Event Treatment Group: , 5 | Illness<br>Start Date<br>(Study<br>Day)<br>Subject ID: , A | Associated<br>with Dose #<br>E Number: | # of Days<br>Post<br>Associated<br>Dose | Blood<br>ZIKV qT-<br>PCR<br>Result | Urine<br>ZIKV qT-<br>PCR<br>Result | Blood<br>DENV qT-<br>PCR<br>Result | Blood<br>CHIKV<br>qT-PCR<br>Result | Last Immunogenicity Visit Prior to the Illness Visit (Study Day) | First<br>Immunogenicity<br>Visit Following<br>the Illness Visit<br>(Study Day) | 4-fold rise<br>in Blood<br>ZIKV<br>Titers<br>After<br>Illness<br>Visit? | 4-fold rise<br>in Blood<br>DENV<br>Titers<br>After<br>Illness<br>Visit? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Comments: | | | | | | | | | | | |

## Listing 13: Listing of Medical Treatment Sought for Subjects Reporting ARI or AFI

[Implementation note: "ZIKV or DENV Infection Confirmation Results" will have a format such as 'No/Yes; PCR positive (Day X)/Yes; 4-fold rise in [DENV/ZIKV] titers (Day Y to Day Z)/Yes; PCR positive (Day X), 4-fold rise in [ZIKV/DENV] titers (Day Y, Day Z)]

| Treatment<br>Group | Subject ID | Illness<br>Number | Study Day | ZIKV or DENV Infection<br>Confirmation | Medical Facility | Date Treatment<br>Sought | Outcome |
|---|---|---|---|---|---|---|---|

### Listing 14: Listing of AFI/ARI Symptoms Reported in Subjects Experiencing ARI or AFI

[Implementation Note: Listing will be sorted by Treatment Group, Subject ID, and Illness Number.

"ZIKV or DENV Infection Confirmation" will have a format such as 'No/Yes; PCR positive (Day X)/Yes; 4-fold rise in [DENV/ZIKV] titers (Day Y, Day Z)/Yes; PCR positive (Day X), 4-fold rise in [ZIKV/DENV] titers (Day Y to Day Z)]

| Treatment<br>Group | Subject<br>ID | Illness<br>Number | Study Day | ZIKV or DENV Infection<br>Confirmation | Symptom | Severity | Start Day | Duration (Days) | Required<br>Concomitant<br>Medication? |
|---|---|---|---|---|---|---|---|---|---|

## Listing 15: Listing of Vital Signs in Subjects Reporting ARI or AFI

[Implementation Note: Listing will be sorted by Treatment Group, Subject ID, and Illness Number.

"ZIKV or DENV Infection Confirmation" will have a format such as 'No/Yes; PCR positive (Day X)/Yes; 4-fold rise in [DENV/ZIKV] titers (Day Y, Day Z)/Yes; PCR positive (Day X), 4-fold rise in [ZIKV/DENV] titers (Day Y to Day Z)]

| Treatment<br>Group | Subject<br>ID | Illness<br>Number | Study<br>Day | ZIKV or DENV<br>Infection<br>Confirmation | Temperature<br>(C) | Systolic Blood<br>Pressure (mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate (beats/min) | Weight<br>(kg) | Height (cm) | BMI (kg/m²) |
|---|---|---|---|---|---|---|---|---|---|---|---|

## Listing 16: Listing of Laboratory Results in Subjects Reporting ARI or AFI

[Implementation Note: Listing will be sorted by Treatment Group, Subject ID, and Illness Number.

"ZIKV or DENV Infection Confirmation" will have a format such as 'No/Yes; PCR positive (Day X)/Yes; 4-fold rise in [DENV/ZIKV] titers (Day Y, Day Z)/Yes; PCR positive (Day X), 4-fold rise in [ZIKV/DENV] titers (Day Y to Day Z)]

| Treatment<br>Group | Subject<br>ID | Sex | Age | Illness<br>Number | Study<br>Day | ZIKV or DENV<br>Infection<br>Confirmation<br>Results | Lab Test | Laboratory<br>Parameter<br>(Units) | Relationship<br>to Treatment | If Not<br>Related,<br>Alternate<br>Etiology | Action<br>Taken<br>with Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

### 16.2.8 Individual Laboratory Measurements

## **Listing 17:** Clinical Laboratory Results – Chemistry

[Implementation Note: Listing will be sorted by Treatment Group, Subject ID, and Planned Time Point]

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study Day | Sex | Age (years) | Laboratory Parameter (Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

## **Listing 18:** Clinical Laboratory Results – Hematology

[Implementation Note: Listing will be sorted by Treatment Group, Subject ID, and Planned Time Point]

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study<br>Day | Sex | Age<br>(years) | Laboratory Parameter<br>(Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

## **Listing 19:** Clinical Laboratory Results – Urinalysis

[Implementation Note: Listing will be sorted by Treatment Group, Subject ID, and Planned Time Point]

| Treatment Group | Subject ID | Planned Time Point | Actual Study<br>Day | Sex | Age (years) | Laboratory Parameter (Units) | Result (Severity Grade) |
|---|---|---|---|---|---|---|---|

### 16.2.9 Vital Signs and Physical Exam Findings

# **Listing 20:** Vital Signs

[Implementation Note: This listing includes all vital sign assessments, scheduled and unscheduled. The severity should be included in parentheses after the result for abnormal assessments. The listing will be sorted by Treatment Group, Subject ID, and Planned Time Point]

| Treatment<br>Group | Subject ID | Planned<br>Time Point | Actual<br>Study Day | Temperature (°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate<br>(beats/min) | Respiratory Rate (breaths/min) | Weight (kg) | Height (cm) | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|---|---|---|

### **Listing 21:** Physical Exam Findings

[Implementation Note: This listing includes all physical exam findings, scheduled and unscheduled. If a subject does not have any findings upon examination, they will not be included in this listing. If reported as an AE, display "Yes" with the AE Number in parentheses, e.g., "Yes (7)". The listing will be sorted by Treatment Group, Subject ID, Planned Time Point.]

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|

#### **Listing 22:** Concomitant Medications

[Implementation Note: If ongoing, display "Ongoing" in the "Medication End Day" column. If taken for an AE or MH, display "Yes" with the AE or MH Number in parentheses, e.g., "Yes (7)". The listing will be sorted by Treatment Group, Subject ID, and CM Number.]

| Treatment<br>Group | Subject<br>ID | CM<br>Number | Medication | Medication<br>Start Day | Medication End<br>Day | Indication | Taken for<br>ARI/AFI? | Taken for<br>ZIKV or<br>DENV<br>Infection? | Taken for an AE? (AE Description; Number) | Taken for a<br>condition on<br>Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### 16.2.8.6 Pregnancy Reports

#### **Listing 23:** Pregnancy Reports – Maternal Information

[Implementation Note: Only include the "Pregnancy Number" column if a subject has more than 1 pregnancy. Date of Conception will be calculated based on estimated delivery date. BMI will be calculated based on pre-pregnancy height and weight. Mother's weight gain will be calculated based on pre-pregnancy weight and end of pregnancy weight. If a major congenital anomaly with previous pregnancy, display "Yes" and the text from the "specify" field, separated by a colon. If any substance use is reported, include a listing of substance use. If autopsy revealed an alternate etiology, display "Yes" and the text from the "specify" field, separated by a colon. If abnormality in product of conception, display "Yes" and the text from the "specify" field, separated by a colon. Sort order: Treatment Group, Subject ID, Pregnancy Number.]

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 24: Pregnancy Reports – Gravida and Para

| | | | Live Births | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>a</sup> | Late<br>TB <sup>a</sup> | Post<br>TB <sup>a</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>a</sup> Term Birth

### **Listing 25:** Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Congenital Anomalies are included in the Adverse Event listing.

#### **Listing 26:** Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress<br>During<br>Labor and<br>Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

### **Listing 27:** Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|